## Johnson & Johnson Vision Care, Inc.

## Clinical Study Protocol

Comparison of Two Silicone Hydrogel Multifocal Contact Lenses

Protocol CR-6344

Version: 1.0

Date: 19 July 2019

Investigational Products: Dailies Total  $1^{\circledR}$  multifocal contact lenses manufactured in

delefilcon A

Air Optix® multifocal contact lenses Plus HydraGlyde® manufactured in lotrafilcon B

Key Words: Presbyopia, Multifocal, Delefilcon A, Lotrafilcon B, Daily Wear, Reusable, Daily Disposable, Dispensing, Randomized

### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, ISO 14155,<sup>1</sup> the International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP),<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> and all applicable regulatory requirements.

#### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

# **TABLE OF CONTENTS**

| PROTO | OCOL TITLE, NUMBER, VERSION | 6 |
|---|---|---|
| | OR NAME AND ADDRESS | |
| | CAL MONITOR | |
| | ORIZED SIGNATURES | |
| | GE HISTORY | |
| | PSIS | |
| | ONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS | |
| | TRODUCTION AND BACKGROUND | |
| 1.1. | Name and Descriptions of Investigational Products | |
| 1.2. | Intended Use of Investigational Products | |
| 1.3. | Summary of Findings from Nonclinical Studies | |
| 1.4. | Summary of Known Risks and Benefits to Human Subjects | |
| 1.5.<br>Clini | Relevant Literature References and Prior Clinical Data Relevant to a cal Study | Proposed |
| 2. ST | TUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES | 17 |
| 2.1. | Objectives | 17 |
| 2.2. | Endpoints | 17 |
| 2.3. | Hypotheses | 17 |
| 3. TA | ARGETED STUDY POPULATION | 17 |
| 3.1. | General Characteristics | 17 |
| 3.2. | Inclusion Criteria | 18 |
| 3.3. | Exclusion Criteria. | 18 |
| 3.4. | Enrollment Strategy | 19 |
| 4. ST | UDY DESIGN AND RATIONALE | 19 |
| 4.1. | Description of Study Design | 19 |
| 4.2. | Study Design Rationale | 19 |
| 4.3. | Enrollment Target and Study Duration | 19 |
| 5. TE | ST ARTICLE ALLOCATION AND MASKING | 20 |
| 5.1. | Test Article Allocation | 20 |
| 5.2. | Masking | 20 |
| 5.3. | Procedures for Maintaining and Breaking the Masking | 20 |
| 6 ST | TIDY INTERVENTION | 21 |

| 6.1. | Identity of Test Articles | 21 |
|--------|--------------------------------------------------|----|
| 6.2. | Ancillary Supplies/Products | 22 |
| 6.3. | Administration of Test Articles | 22 |
| 6.4. | Packaging and Labeling | 22 |
| 6.5. | Storage Conditions | 22 |
| 6.6. | Collection and Storage of Samples | 23 |
| 6.7. | Accountability of Test Articles | 23 |
| 7. STU | UDY EVALUATIONS | 24 |
| 7.1. | Time and Event Schedule | 24 |
| 7.2. | Detailed Study Procedures | 28 |
| VIS | SIT 1 | 28 |
| VIS | SIT 2 | 34 |
| VIS | SIT 3 | 39 |
| VIS | SIT 4 | 42 |
| VIS | SIT 5 | 47 |
| VIS | SIT 6 | 51 |
| FIN | IAL EVALUATION | 54 |
| 7.3. | Unscheduled Visits | 54 |
| 7.4. | Laboratory Procedures | 56 |
| 8. SU | BJECTS COMPLETION/WITHDRAWAL | |
| 8.1. | Completion Criteria | 57 |
| 8.2. | Withdrawal/Discontinuation from the Study | 57 |
| 9. PR | E-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | 58 |
| 10. D | EVIATIONS FROM THE PROTOCOL | 58 |
| 11. S' | TUDY TERMINATION | 58 |
| 12. P | ROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | 59 |
| 13. A | DVERSE EVENTS | 60 |
| 13.1. | Definitions and Classifications | 60 |
| 13.2. | Assessing Adverse Events | 62 |
| 13.2.1 | . Causality Assessment | 63 |
| 13.2.2 | . Severity Assessment | 63 |
| 13.3. | Documentation and Follow-Up of Adverse Events | 63 |
| 13.4. | Reporting Adverse Events | 65 |
| 13.4.1 | Reporting Adverse Events to Sponsor | 65 |

| 13.4.2. | Reporting Adverse Events to the Responsible IEC/IRB and Health Authoritie | s. 66 |
|---|---|---|
| 13.4.3. | Event of Special Interest. | 66 |
| 13.5. | Reporting of Pregnancy | 66 |
| 14. ST | ATISTICAL METHODS | 66 |
| 14.1. | General Considerations. | 66 |
| 14.2. | Sample Size Justification. | 67 |
| 14.3. | Analysis Populations | 67 |
| 14.4. | Level of Statistical Significance | 67 |
| 14.5. | Primary Analysis | 68 |
| 14.6. | Secondary Analysis | 68 |
| 14.7. | Other Exploratory Analyses | 69 |
| 14.8. | Interim Analysis | 69 |
| 14.9. | Procedure for Handling Missing Data and Drop-Outs | 69 |
| 14.10. | Procedure for Reporting Deviations from Statistical Plan | 69 |
| 15. DA | TA HANDLING AND RECORD KEEPING/ARCHIVING | 69 |
| 15.1. | Electronic Case Report Form/Data Collection | 69 |
| 15.2. | Subject Record. | 70 |
| 16. DA | TA MANAGEMENT | 70 |
| 16.1. | Access to Source Data/Document | 70 |
| 16.2. | Confidentiality of Information | 71 |
| 16.3. | Data Quality Assurance | 71 |
| 17. MC | ONITORING | 71 |
| 18. ET | HICAL AND REGULATORY ASPECTS | 72 |
| 18.1. | Study-Specific Design Considerations | 72 |
| 18.2. | Investigator Responsibility | |
| 18.3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 72 |
| 18.4. | Informed Consent | 73 |
| 18.5. | Privacy of Personal Data | 74 |
| 19. ST | UDY RECORD RETENTION | 75 |
| 20. FIN | VANCIAL CONSIDERATIONS | 75 |
| | BLICATION | |
| | FERENCES | |
| | X A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES) | 77 |
| <b>A DDENIDI</b> | X B. PATIENT INSTRUCTION GUIDE | 100 |

| APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT) | 110 |
|----------------------------------------------------------------|---------|
| APPENDIX D: BINOCULAR OVER REFRACTION | 116 |
| APPENDIX E: PRESBYOPIC SYMPTOMS QUESTIONNAIRE | 117 |
| APPENDIX F: OCULAR DOMINANCE | 118 |
| APPENDIX G: ALCON DAILIES TOTAL 1 MULTIFOCAL CONTACT LEN GUIDE | |
| APPENDIX H: ALCON AIR OPTIX MULTIFOCAL CONTACT LENS PLUS | |
| HYDRAGLYDE FITTING GUIDE | |
| APPENDIX I: | |
| , LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS | 196 |
| EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING | 204 |
| DETERMINATION OF NEAR ADD | 209 |
| NEAR logMAR VISUAL ACUITY MEASUREMENT PROCEDURE | E 217 |
| LENS FITTING CHARACTERISTICS | 220 |
| SUBJECT REPORTED OCULAR SYMPTOMS | 227 |
| DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFI | |
| BIOMICROSCOPY SCALE | 236 |
| KERATOMETRY | 242 |
| DISTANCE AND NEAR VISUAL ACUITY EVALUATION | 244 |
| ETDRS DISTANCE VISUAL ACUITY MEASURMENT PROCEDU | VRE 249 |
| VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMING. | |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | 259 |
| TABLE OF CONTENTS Figure 1: Study Flowchart | 13 |
| TABLE OF CONTENTS | |
| Table 1: Test Articles | |
| Table 2: Ancillary Supplies | |
| Table 3: Time and Events | 24 |

#### PROTOCOL TITLE, NUMBER, VERSION

Title: Comparison of Two Silicone Hydrogel Multifocal Contact Lenses

Protocol Number: CR-6344

Version: 1.0 Date: 19 July 2019

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

#### **MEDICAL MONITOR**

Name: Thomas R. Karkkainen, OD, MS, FAAO

Title: Sr. Principal Research Optometrist

Address: 7500 Centurion Parkway, Jacksonville, Florida 32256

Email: TKarkkai@its.jnj.com

The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

#### **AUTHORIZED SIGNATURES**

The signature below constitutes the approval of this protocol and the attachments, and provides the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations,<sup>4</sup> ICH guidelines,<sup>2</sup> ISO 14155,<sup>1</sup> and the Declaration of Helsinki.<sup>3</sup>

| Author | See Electronic Signature Report Thomas R. Karkkainen, OD, MS, FAAO Sr. Principal Research Optometrist, Clinical Sciences | DATE |
|---|---|---|
| Clinical Operations<br>Manager | See Electronic Signature Report Clinical Operations Manager, Clinical Operations | DATE |
| Biostatistician | See Electronic Signature Report Biostatistician IV, Clinical Sciences | DATE |
| Data Management | See Electronic Signature Report Clinical Project Manager-Data and Systems, Clinical Operations | DATE |
| Reviewer | See Electronic Signature Report Clinical Research Fellow, Clinical Sciences | DATE |
| Approver | See Electronic Signature Report Presbyopia Platform Sr. Manager, Clinical Operations | DATE |

## **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section<br>Number(s) Affected | Date |
|---|---|---|---|
| 1.0 | Tom Karkkainen | Original Protocol | 19-July-2019 |

## **SYNOPSIS**

| Protocol Title | Comparison of Two Silicone Hydrogel Multifocal Contact |
|---|---|
| | Lenses IIVC 7500 Centurion Parkway Jacksonville FL 32256 |
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Development Phase 2 |
| Trial Registration | This study will be registered on ClinicalTrials.gov. |
| Test Article(s) | Investigational Products: Dailies Total 1® multifocal contact |
| | lenses manufactured in delefilcon A material. |
| | Air Optix <sup>®</sup> multifocal contact lenses Plus HydraGlyde <sup>®</sup> |
| | manufactured in lotrafilcon B material. |
| Wear and Replacement | Wear Schedule: The Test lenses are used as daily wear. One |
| Schedules | of the Test lenses will be reusable, cleaned and stored each |
| | night and the other will be daily disposable with a new lens |
| | worn each day. |
| | Replacement Schedule: The Test and/or Control lenses that is |
| | fit at Visit 1 will be replaced at Visit 2 optimization visit and |
| | then worn as daily reusable modality without further planned |
| | replacement for 7±1 day. There will be a 7±3 day wash-out |
| | period before the remaining lens is fit, and the procedures are |
| | repeated. The test lenses will also be replaced when lost or |
| | damaged. |
| Objectives | This study is an evaluation of the lens fit and handling |
| | response of both the Air Optix® multifocal contact lenses Plus |
| | HydraGlyde and the Dailies Total 1 <sup>®</sup> multifocal contact lens. |
| Study Endpoints | Primary endpoints: Lens centration and lens movement |
| _ | Secondary endpoints: Lens handling Other observations: |
| | number of lenses needed to fit (optimize) the subject, visual |
| | acuity and subjective responses. |
| Study Design | This is a single-masked, randomized-controlled, dispensing |
| | clinical trial. A total of approximately 40 eligible hyperopic |
| | and myopic subjects will be targeted to complete the study. |
| | The subjects will be fit in the first study lens based on the |
| | randomization scheme and wear the lens for 3±1 day then |
| | undergo optimization, if applicable, and wear the optimized |
| | pair with a follow-up in 7±1 day. The remaining lens will be |
| | fit according to the random scheme at Visit 4 following a 7±3 |
| | day wash-out period. The procedures will be repeated for the |
| | 2 <sup>nd</sup> lens. |
| | The primary endpoints will be lens centration and lens |
| | movement. |
| Sample Size | A total of approximately 40 subjects will be targeted to |
| _ | complete. |
| Study Duration | The study will last approximately 2-4 months. |

| Anticipated Study | Healthy male and female volunteers with presbyopia will be |
|---|---|
| Population | invited to participate in the study. Subjects will be adapted |
| | soft contact lens wearers in both eyes. Additional information |
| | regarding the eligibility of the population can be found in the |
| | inclusion/exclusion criteria outlined below. |
| Eligibility Criteria | Potential subjects must satisfy all the following criteria to be |
| | enrolled in the study |
| | 1. The subject must read, understand, and sign the |
| | STATEMENT OF INFORMED CONSENT and |
| | receive a fully executed copy of the form. |
| | 2. The subject must appear able and willing to adhere to |
| | the instructions set forth in this clinical protocol. |
| | 3. The subject must be between 40 and 70 years of age (inclusive). |
| | 4. The subject's distance spherical equivalent refraction |
| | must be in the range of +1.25 D to +3.75 D or -1.25 D |
| | to -4.00 D in each eye. |
| | 5. The subject's refractive cylinder must be ≤0.75 D in each eye. |
| | 6. The subject's ADD power must be in the range of |
| | +0.75 D to +2.50 D. |
| | 7. The subject must have best corrected visual acuity of |
| | 20/20 <sup>-3</sup> or better in each eye. |
| | 8. Subjects must own a wearable pair of spectacles if |
| | required for their distance vision. |
| | 9. The subject must be an adapted soft contact lens |
| | wearer in both eyes (i.e. worn lenses a minimum of |
| | 2 days per week for at least 8 hours per wear day, for |
| | 1 month of more duration). |
| | 10. The subject must either already be wearing a |
| | presbyopic contact lens correction (e.g., reading |
| | spectacles over contact lenses, multifocal or |
| | monovision contact lenses, etc.) or if not respond |
| | positively to at least one symptom on the "Presbyopic |
| | Symptoms Questionnaire". |
| | Potential subjects who meet any of the following criteria will |
| | be excluded from participating in the study: |
| | 1. Currently pregnant or lactating. |
| | 2. Any active or ongoing ocular or systemic allergies that |
| | may interfere with contact lens wear. |
| | 3. Any active or ongoing systemic disease, autoimmune |
| | disease, or use of medication, which may interfere with |
| | contact lens wear. This may include, but not be limited |
| | to, diabetes, hyperthyroidism, Sjögren's syndrome, |
| | xerophthalmia, acne rosacea, Stevens-Johnson |

| | syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis). 4. Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear. 5. Entropion, ectropion, extrusions, chalazia, recurrent styes, dry eye, glaucoma, history of recurrent corneal erosions. 6. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, dacryocystorhinostomy, cataract surgery, retinal surgery, etc.). 7. A history of amblyopia, strabismus or binocular vision abnormality. 8. Any current ocular infection or inflammation. 9. Any current ocular abnormality that may interfere with contact lens wear. 10. Use of any of the following oral medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral antihistamines (e.g., Chlor-Trimeton, and Benadryl), systemic steroids. 11. Use of any ocular medication, with the exception of rewetting drops. 12. History of herpetic keratitis. 13. Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment. 14. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician). 15. Any known hypersensitivity or allergic reaction to OPTI-FREE® Puremoist® multi-purpose care solution, sodium fluorescein or single-use preservative free rewetting drops solution. |
|---|---|
| | Coordinator, Technician). 15. Any known hypersensitivity or allergic reaction to OPTI-FREE® Puremoist® multi-purpose care solution, |
| Disallowed | Use of any prescription or over-the-counter (OTC) |
| Medications/Interventions | medications that may affect contact lens wear. |
| Measurements and | logMAR Visual acuity and Subjective responses for vision |
| Procedures | using the CLUE questionnaire. |
| Microbiology or Other | None |
| Laboratory Testing | |

| Study Termination | The occurrence of one or more Unanticipated Adverse Device |
|---|---|
| | Effect (UADE), or any SAE where relationship to study agent |
| | cannot be ruled out, will result in stopping further dispensing |
| | investigational product. In the event of a UADE or SAE, the |
| | Sponsor Medical Monitor may unmask the treatment regimen |
| | of subject(s) and may discuss this with the Principal |
| | Investigator before any further subjects are enrolled. |
| Ancillary Supplies/ Study- | Rewetting drops, lens cases, glass vials, saline, ETDRS light |
| Specific Materials | cabinet, logMAR charts, and Near logMAR charts. OPTI- |
| | FREE® Puremoist® Contact Solution. |
| Principal Investigator(s) | A full list of Principal Investigators, clinical sites, and |
| and Study | institutions is kept separately from the Study Protocol and is |
| Institution(s)/Site(s) | included in the study Trial Master File. |

Figure 1: Study Flowchart



#### COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS

ADD Plus Power Required for Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience
BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience

COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonization

IDE Investigational Device Exemption
IEC Independent Ethics Committee
IRB Institutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LC Limbus Center

LogMAR Logarithm of Minimal Angle of Resolution MedDRA<sup>©</sup> Medical Dictionary for Regulatory Activities

MOP Manual of Procedures

NIH National Institutes of Health

OD Right Eye

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

OS Left Eye
OU Both Eyes

PD Protocol Deviation

PHI Protected Health Information

PI Principal Investigator
PIG Patient Instruction Guide

PQC Product Quality Complaint PRO Patient Reported Outcome

QA Quality Assurance QC Quality Control

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation

SOP Standard Operating Procedure

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

Competitors have launched multifocal lenses that have the same optical design but are manufactured in different silicone hydrogel materials. The optical designs are center near aspheric. For aspheric designs the mechanical fit of the lens, centration in particular, can have a significant impact on the optical performance of the lens. The purpose of this study is to evaluate two such designs, Air Optix® multifocal contact lenses Plus HydraGlyde® manufactured in lotrafilcon B and Dailies Total 1® manufactured in delefilcon-A, and compare their mechanical fitting characteristics.

#### 1.1. Name and Descriptions of Investigational Products

Test Lenses: J Dailies Total 1® multifocal contact lenses manufactured in delefilcon A. Air Optix® multifocal contact lenses Plus HydraGlyde® manufactured in lotrafilcon B

#### 1.2. Intended Use of Investigational Products

All lenses are intended to correct spherical refractive error and presbyopia. For this study one of the lenses is intended to be used as a daily wear, reusable lens. These lenses will be cleaned, disinfected and stored in multipurpose lens solutions. The second test lens will be worn as a daily disposable lens, with the lenses being discarded after a day of wear. The Lens systems will be fit in a randomized fashion. After fitting, each subject will return for an optimization visit and then a follow-up. The sequence will then be repeated with the additional study lens type. Each study lens type will be worn for a total of approximately 8-12 days.

#### 1.3. Summary of Findings from Nonclinical Studies

Not Applicable

#### 1.4. Summary of Known Risks and Benefits to Human Subjects

Anticipated risks and adverse reactions with this lens are similar to those with other soft daily wear contact lenses used to correct presbyopia. A listing of examples of adverse reactions is found in the Section 13 of this protocol. The investigator should follow normal clinical guidelines regarding examination and care of subjects who participate in this trial. Refer to study lens package insert for additional details. The study multifocal contact lens is designed for the correction of refractive spherical ametropia and presbyopia. one study contact lenses is manufactured in lotrafilcon B and will be worn in a daily wear, reusable modality. The other study contact lens is manufactured in delefilcon A and will be worn in a daily wear, disposable modality. These lens is not intended for extended wear in this study.

# 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

Information about both the Air Optix® Plus HydraGlyde® Multifocal Contact Lenses and Dailies Total 1® Multifocal Contact Lenses may be found in the package inserts.

#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

#### 2.1. Objectives

This study is an evaluation of the lens fit and handling response of both the Air Optix<sup>®</sup> multifocal contact lenses Plus HydraGlyde and the Dailies Total 1<sup>®</sup> multifocal contact lens.

#### 2.2. Endpoints

Primary endpoints: lens centration and lens movement

Secondary endpoints: Subjective lens handling

Other observations: number of lenses needed to fit (optimize) the subject, visual acuity and subjective responses.

#### 2.3. Hypotheses

The following hypotheses will be tested throughout this investigation.

#### **Primary Hypotheses:**

- 1. After 6-8 days of wear in the optimized lenses, the proportion of lenses graded as being centered for the test lens will be non-inferior compared to the control lens. A non-inferiority margin of 0.67 odds ratio will be used.
- 2. After 6-8 days of wear in the optimized lenses, the proportion of lenses graded as having optimal lens movement in primary gaze for the test lens will be non-inferior compared to the control lens. A non-inferiority margin of 0.67 odds ratio will be used.

#### Secondary Hypothesis:

1. After 6-8 days of wear in the optimized lenses, the overall lens handling of the test lens system will be non-inferior compared to that of the control lens system. A non-inferiority margin of -5 CLUE points will be used.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

Healthy male and female subjects who are habitual soft contact lens wearers will be recruited. Subjects will be at least 40 years of age and not older than 70 years of age. They will be hyperopic or myopic and have presbyopia.

#### 3.2. Inclusion Criteria

Potential subjects must satisfy all the following criteria to be enrolled in the study:

- 1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. The subject must appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. The subject must be between 40 and 70 years of age (inclusive).
- 4. The subject's distance spherical equivalent refraction must be in the range of +1.25 D to +3.75 D or -1.25 D to -4.00 D in each eye.
- 5. The subject's refractive cylinder must be  $\leq 0.75$  D in each eye.
- 6. The subject's ADD power must be in the range of +0.75 D to +2.50 D.
- 7. The subject must have best corrected visual acuity of  $20/20^{-3}$  or better in each eye.
- 8. Subjects must own a wearable pair of spectacles if required for their distance vision.
- 9. The subject must be an adapted soft contact lens wearer in both eyes (i.e. worn lenses a minimum of 2 days per week for at least 8 hours per wear day, for 1 month of more duration).
- 10. The subject must either already be wearing a presbyopic contact lens correction (e.g., reading spectacles over contact lenses, multifocal or monovision contact lenses, etc.) or if not respond positively to at least one symptom on the "Presbyopic Symptoms Questionnaire".

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

- 1. Currently pregnant or lactating.
- 2. Any active or ongoing ocular or systemic allergies that may interfere with contact lens wear.
- 3. Any active or ongoing systemic disease, autoimmune disease, or use of medication, which may interfere with contact lens wear. This may include, but not be limited to, diabetes, hyperthyroidism, Sjögren's syndrome, xerophthalmia, acne rosacea, Stevens-Johnson syndrome, and immunosuppressive diseases or any infectious diseases (e.g. hepatitis, tuberculosis).
- 4. Clinically significant (Grade 3 or 4) corneal edema, corneal vascularization, corneal staining, tarsal abnormalities or bulbar injection, or any other corneal or ocular abnormalities which would contraindicate contact lens wear.
- 5. Entropion, ectropion, extrusions, chalazia, recurrent styes, dry eye, glaucoma, history of recurrent corneal erosions.
- 6. Any previous, or planned, ocular or intraocular surgery (e.g. radial keratotomy, PRK, LASIK, lid procedures, dacryocystorhinostomy, cataract surgery, retinal surgery, etc.).
- 7. A history of amblyopia, strabismus or binocular vision abnormality.
- 8. Any current ocular infection or inflammation.
- 9. Any current ocular abnormality that may interfere with contact lens wear.
- 10. Use of any of the following oral medications within 1 week prior to enrollment: oral retinoid isotretinoin (e.g. Accutane), oral tetracyclines, topical scopolamine, oral antihistamines (e.g., Chlor-Trimeton, and Benadryl), systemic steroids.

- 11. Use of any ocular medication, with the exception of rewetting drops.
- 12. History of herpetic keratitis.
- 13. Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
- 14. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician).
- 15. Any known hypersensitivity or allergic reaction to OPTI-FREE® Puremoist® multipurpose care solution, sodium fluorescein or single-use preservative free rewetting drop solution.

#### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.

#### 4. STUDY DESIGN AND RATIONALE

#### 4.1. Description of Study Design

The clinical study is a randomized-controlled, single-masked, crossover clinical trial. There are two study treatments. A total of approximately 50 subjects will be enrolled with 40 (20 myopic and 20 hyperopic) eligible subjects targeted to complete the study. The first Test article will be dispensed for  $3\pm1$  day and an optimization visit will occur. The final lens pair will be dispensed for  $7\pm1$  day and the at the follow-up the final lens measurements will occur. Subjects will complete a  $7\pm3$  days washout between each fitting. The second study lens will then be fit and follow the same sequence as the first lens.

#### 4.2. Study Design Rationale

The study is intended to compare two study lens types and the initial performance, in terms of the mechanical lens fit and handling after a period of lens dispensing. The lenses are dispensed to determine the handling responses and the comparison is made after a total of 8-12 days of wear.

The crossover study design was chosen to control for variables that may impact the lens performance between subjects. A washout period between Period 1 and Period 2 of wear is used to minimize the chance of carryover effect in the study data.

#### 4.3. Enrollment Target and Study Duration

A total of approximately 50 eligible subjects will be enrolled with 40 targeted to complete the study. The study will last approximately 2-4 months.

#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

The study lenses will be worn in a bilateral and random fashion using a  $2\times2$  crossover design with 2 lens types and 2 periods. Using a computer-generated randomization scheme provided by the study biostatistician, each subject will randomly be assigned to one of two unique sequences (Test/Control or Control/Test). Randomization will be stratified by site.

Permuted block randomization will be used to avoid bias in the assignment of subjects to treatment, and to enhance the validity of statistical comparisons across treatment groups. Each block will contain two different lens trial sequences.

The order of lens wear will be based on the randomization scheme assigned to the study site. The study site will follow the randomization scheme provided and will complete enrollment according to the randomization list and will not pre-select or assign subjects.

#### 5.2. Masking

This is a single-masked study with the subjects being masked. The masking will be partial as the subjects will have different wear modalities however the brand name of the lenses will not be revealed to the subject.

Under normal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the subject. In such cases, the Investigator may, in an emergency, contact the medical monitor. In the event the mask is broken, the Sponsor must be informed as soon as possible. The date, time, and reason for the unmasking must be documented in the subject record. The Investigator is also advised not to reveal the study treatment assignment to the clinical site or Sponsor personnel.

Subjects who have had their treatment assignment unmasked are expected to return for all remaining scheduled evaluations. Subjects who are discontinued may be replaced.

#### 5.3. Procedures for Maintaining and Breaking the Masking

The test articles mask shall not be broken unless information concerning the lens type is necessary for the urgent medical treatment of a subject. The Sponsor must be notified before the mask is broken.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- 1. Investigator or designee (documented on the Delegation Log) will consult the lens fitting schedule/randomization scheme to obtain the test article assignment for that subject prior to dispensing
- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme if applicable

3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section

#### 6. STUDY INTERVENTION

### 6.1. Identity of Test Articles

The following contact lenses will be used in this study:

Table 1: Test Articles

| | Test | Control |
|---|---|---|
| Name | Dailies Total 1® Multifocal | Air Optix® Multifocal Contact |
| | Contact Lenses | Lenses Plus HydraGlyde® |
| Manufacturer | Alcon | Alcon |
| Lens Material | delefilcon A | Lotrafilcon B |
| Nominal Base Curve @ 22°C | 8.5 mm | 8.6 |
| Nominal Diameter @ 22°C | 14.1 mm | 14.2 mm |
| Nominal Distance | +0.75 D to +4.00 D and -0.75 | +0.75 D to +4.00 D and -0.75 D |
| Powers (D) | D to -4.00 D in 0.25 D steps | to -4.00 D in 0.25 D steps |
| Nominal Cylinder | None | None |
| Powers (D) and Axes | | |
| Nominal ADD Powers (D) | LO, MED, HI | LO, MED, HI |
| Water Content | 33% | 33% |
| Center Thickness | 0.09 mm | 0.08 mm @ -3.00 D |
| | (-1.00 D) | 9-2 |
| Oxygen Permeability | 156 | 110 |
| (Dk) | | |
| Wear Schedule in<br>Current Study | Daily Wear | Daily Wear |
| Replacement Frequency | Daily | 2 weeks |
| Packaging Form (vial, blister, etc.) | Blister | Blister |

#### 6.2. Ancillary Supplies/Products

The following solutions will be used in this study:

Table 2: Ancillary Supplies

| | Single-Use Preservative-Free Rewetting Solutions (any one of these three rewetting | | | Multipurpose Solution |
|---|---|---|---|---|
| | | ons may be sup | | |
| | Eye-Cept® | ScleralFil® | LacriPure | OPTI_FREE® |
| Solution | Rewetting | Preservative | Saline | Puremoist® |
| Name/Description | Drops | Free Saline | Solution | multipurpose contact |
| | | Solution | 11154 PLA 9004 PLA | lens solution |
| Manufacturer | Optics | B&L | Menicon | Alcon |
| Manufacturei | Laboratory | | | The section of the se |
| | Non- | Non- | Non- | Polyquanternium-1 |
| | Preserved | preserved | preserved | 0.001% and |
| Preservative | | | - | myristamidopropyl |
| | | | | dimethylamine |
| | | | | 0.0006% |

#### 6.3. Administration of Test Articles

Test articles will be dispensed to subject meeting all eligibility requirements, including any dispensing requirements set forth in this clinical protocol. Subjects will be dispensed an adequate supply of test articles to complete the study. Lost or damaged test articles may be replaced at the discretion of the Investigator and/or the Sponsor.

#### 6.4. Packaging and Labeling

The test articles will be packaged in blisters, as the primary packaging. The test article will be over-labeled to mask the subject to the identity of the lens. The test articles will be in investigational cartons sealed with a tamper evident seal, commercial cartons, or in plastic bags as the secondary packaging form. The sample study label is shown below:



#### 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions.

#### 6.6. Collection and Storage of Samples

When possible, any lens or test article associated with an Adverse Events and/or a Product Quality Complaint must be retained and stored in a glass vial with moderate solution pending directions from the sponsor for potential return back to JJVC.

#### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test article must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed for the subject for trial fitting, to wear out of the office, or issued for the subject to replace appropriately between visits
- 2. What was returned to the Investigator unused
- 3. The number and reason for unplanned replacements

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will return all unused test articles the Sponsor.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor <u>immediately.</u>

## 7. STUDY EVALUATIONS

## 7.1. Time and Event Schedule

Table 3: Time and Events

| Visit Information | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit |
|---|---|---|---|---|---|
| VISIT IIIOIIIIIIII | Screening, | Treatment 1 | Treatment 1 | Baseline | Treatme |
| | Baseline, | Follow-up 1 | Follow-up 2 | Treatment 2 | Follow-u |
| | Treatment 1 | Optimization | Tollow up 2 | Treatment 2 | Optimiza |
| Time Point | Day 0 | Day 3±1 | Day 7±1 | Day 7±3 | Day 3= |
| Time Tom | Day | from V1 | from V2 | from V3 | from V |
| | | Hom v i | Hom v2 | Day 0 | Hom . |
| | | | Complete | Day | |
| | | | 7±3 days | | |
| | | | washout before | | |
| | | | V4 | | |
| Estimated Visit Duration | 2.5 hours | 1.0 hour | 1.5 hour | 1.5 hour | 1.0 ho |
| Statement of Informed | 2.3 Hours | 1.0 11001 | 1.3 11041 | 1.5 11001 | 1.0 110 |
| A Contract at the contract of the contract of the profession of the contract o | | | 1 | 1 | |
| Consent | X | + | <del> </del> | <del> </del> | - |
| Demographics | X | 1 2 | <u> </u> | <u> </u> | |
| Medical | [ | | 1 | 1 | |
| History/Concomitant | | | 1 | 1 | |
| Medications | X | | <b></b> ' | <u> </u> | |
| Adverse Events and | [ | | 1 | 1 | |
| Concomitant Medications | [ | | <u>'</u> | 1 | |
| Review | <u> </u> | X | x | X | X |
| Compliance | | X | X | | X |
| Habitual Contact Lens | [ | | 1 | 1 | |
| Information | X | | <u></u> | <u> </u> | |

| Visit Information | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit |
|---|---|---|---|---|---|
| | Screening, | Treatment 1 | Treatment 1 | Baseline | Treatme |
| | Baseline, | Follow-up 1 | Follow-up 2 | Treatment 2 | Follow-u |
| | Treatment 1 | Optimization | _ | | Optimiza |
| Time Point | Day 0 | Day 3±1 | Day 7±1 | Day 7±3 | Day 3 |
| | | from V1 | from V2 | from V3 | from V |
| | | | | Day 0 | |
| | | | Complete | | |
| | | | 7±3 days | | |
| | | | washout before | | |
| | | | V4 | | |
| Estimated Visit Duration | 2.5 hours | 1.0 hour | 1.5 hour | 1.5 hour | 1.0 ho |
| Contact Lens History | X | | | | |
| Wear Time and | | | | | |
| Comfortable Wear Time | | | | | |
| with Habitual lenses | X | | | | |
| Wear Time and | | | | | |
| Comfortable Wear Time | | | | | |
| with Study lenses | ( | X | X | | X |
| Screening | | | | | |
| Inclusion/Exclusion | | | | | |
| Criteria | X | | | | |
| Subject Reported Ocular | | | | | |
| Symptoms | X | X | X | X | X |
| | X | | | | |
| | X | 8 | X | | |
| Distance and Near | | | | | |
| Entrance Visual Acuity | X | X | X | X | X |
| Lens Removal | X | X | X | X | X |
| Keratometry | X | | | | |
| Subjective Refraction and | X | | | | |

| Visit Information | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit |
|---|---|---|---|---|---|
| | Screening, | Treatment 1 | Treatment 1 | Baseline | Treatme |
| | Baseline, | Follow-up 1 | Follow-up 2 | Treatment 2 | Follow-u |
| | Treatment 1 | Optimization | | | Optimiza |
| Time Point | Day 0 | Day 3±1 | Day 7±1 | Day 7±3 | Day 3= |
| | | from V1 | from V2 | from V3 | from V |
| | | | | Day 0 | |
| | | | Complete | | |
| | | | 7±3 days | | |
| | | | washout before | | |
| | | | V4 | | |
| Estimated Visit Duration | 2.5 hours | 1.0 hour | 1.5 hour | 1.5 hour | 1.0 ho |
| Distance Visual Acuity | | | | | |
| Near ADD Determination | X | | <u> </u> | | |
| Ocular Dominance | X | | ' | | |
| ADD Refinement | X | | | | |
| Near Visual Acuity | X | | | | |
| Biomicroscopy | X | X | X | X | X |
| Baseline Inclusion/ | | | ! | | |
| Exclusion Criteria | X | | | | |
| Continuance | | | ! | X | |
| Lens Selection | X | x (If modified) | | X | x (If modi |
| Lens Insertion | X | X | | X | X |
| 10 Minute Settling | | | 1 | | |
| | X | X | | X | X |
| Visual Satisfaction / | | | ! | | |
| Subjective Acceptance | X | X | X | X | X |
| Study Lens Distance and | | | ! | | |
| Near Visual Acuity | X | X | X | X | X |
| Distance Over Refraction | | | ! | | |
| and Visual Acuity | X | X | | X | X |

| Visit Information | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit |
|---|---|---|---|---|---|
| | Screening, | Treatment 1 | Treatment 1 | Baseline | Treatme |
| | Baseline, | Follow-up 1 | Follow-up 2 | Treatment 2 | Follow-u |
| | Treatment 1 | Optimization | | | Optimiza |
| Time Point | Day 0 | Day 3±1 | Day 7±1 | Day 7±3 | Day 3 |
| | | from V1 | from V2 | from V3 | from V |
| | | | | Day 0 | |
| | | | Complete | | |
| | | | 7±3 days | | |
| | | | washout before | | |
| | | | V4 | | |
| Estimated Visit Duration | 2.5 hours | 1.0 hour | 1.5 hour | 1.5 hour | 1.0 ho |
| Subjective Lens Fit | | | | | |
| Assessment | X | X | X | X | X |
| Binocular Over Refraction | | 8 | X | | |
| Compliance | | X | X | | X |
| | | X | X | | X |
| Visual Performance | | | X | | |
| Modifications | X | X | | X | X |
| | X | X | | X | X |
| Distance and Near Exit | | | | | |
| Visual Acuity | X | X | X | X | X |
| Dispensing Criteria | X | X | | X | X |
| Instructions | X | X | X | X | X |
| Schedule Follow-up | X | X | X | X | X |
| Final Evaluation | | | | | |

## 7.2. Detailed Study Procedures

#### VISIT 1

Subjects must report to the visit wearing their habitual contact lenses to accurately assess baseline PRO (CLUE and MRD) performance. If the subject is not wearing their lenses they must be rescheduled.

| | Visit 1: Screening | |
|---|---|---|
| Step | Procedure | Details |
| 1.1 | Statement of<br>Informed Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. NOTE: The subject must be provided a signed copy of this document. |
| 1.2 | Demographics | Record the subject's age, gender, race and ethnicity. |
| 1.3 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subjects' medical history and concomitant medications. |
| 1.4 | Habitual Lenses | Questions regarding the subject's habitual lens type and parameters. |
| 1.5 | Contact Lens History | Record the subject's correction type (i.e. monovision, multifocal, sphere with readers, etc.). |
| 1.6 | Wear time and<br>Comfortable Wear<br>time with Habitual<br>lenses | Record the subjects wear time and comfortable wear time with their habitual contact lenses. |
| 1.7 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. |

| | Visit 1: Baseline | |
|------|-------------------|---------|
| Step | Procedure | Details |
| 1.8 | | |
| | 85 SS | |

| 1.9 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
|---|---|---|
| 1.10 | Entrance Visual<br>Acuity | Distance and near Snellen visual acuity will be measured for each eye with the subject's habitual contact lenses in place. |
| | | For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| 1.11 | Lens Removal | Have the subject remove their habitual lenses and store in an approved storage solution. |
| 1.12 | Keratometry | Keratometry will be performed OD and OS and the steep and flat dioptric power and corresponding meridians recorded. |
| 1.13 | Subjective Refraction<br>and Distance Visual<br>Acuity | An optimal, binocular balanced distance sphero-cylindrical refraction will be performed. Record the refraction and distance visual acuity to the nearest letter. |
| | | NOTE: Best distance visual acuity with sphero-cylindrical refraction must be at least 20/20-3 in each eye for the subject to be eligible in the study. |
| 1.14 | Near ADD Determination | The near reading addition will be determined using the binocular crossed cylinder technique (BCC) at 40 cm followed by optimization in a trial frame in step 1.16 below. |
| 1.15 | Ocular Dominance | Determine the distance ocular dominance with the best distance correction in place using a +1.00-blur test. If the results are equivocal use the sighting dominance test to determine the dominant eye used for the study. |
| 1.16 | ADD Refinement | Place the BCC result in the trial frame and refine the near prescription with trial lenses (or flippers) under binocular conditions. |
| 1.17 | Near Visual Acuity | Using the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm. Record the near visual acuity OD, OS and OU at 40 cm. |
| 1.18 | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. |
| | | For the conjunctival redness 0.5 unit increments will be used in the grading. Corneal Staining Assessment will be graded in 1.0 increments. |

| | | If any of these slit lamp findings are Grade 3 or higher, the subject will be discontinued. If discontinued a final examination must be completed. |
|---|---|---|
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| 1.19 | Eligibility after<br>Baseline | All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. If so, proceed to lens fitting. If not, complete the final evaluation and discharge the subject. |

| | | Visit 1: Treatment 1 Lens Fitting | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.20 | Randomization | Record the randomization ID. | 200 |
| 1.21 | Lens Selection | Select the lens pair and power based on the randomization scheme, spherical equivalent refraction and fitting guide for each eye. | |
| ji. | | Record the Test lens parameters (power and lot number). | |
| 1.22 | Lens Insertion | Subjects will insert the lenses themselves. If the lens is uncomfortable, inspect for damage and remove, reinsert or replace as necessary. Damaged lenses will be stored in labeled vial with sterile saline, and clearly differentiated | |
| | | from the other worn lenses that will be shipped back to the Sponsor. Complete the Quality Product Complaint form. | |
| 1.23 | Lens Settling | Allow the study lenses to settle for a minimum of 10 minutes. | a. |
| 1.24 | Determine Visual<br>Satisfaction | Determine if the subject's vision is acceptable with the lenses. Allow the subject to look down a hallway or out of a window for distance vision assessments, and for them to read a book, magazine or similar for near vision. | |
| 1.25 | Study Lens Distance<br>and Near Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. | |

| | [a | | No. |
|---|---|---|---|
| | | NOTE: Use the ETDRS 2000 Series Chart 1 | |
| | | or 2 near card placed at 40 cm to measure | |
| 101 | B | the Near visual acuity | |
| 1.26 | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. | |
| 1.27 | Subjective Lens Fit<br>Assessment | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). | |
| | | <ul> <li>The subject should not proceed to wear the lenses if any of the following is observed:</li> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up).</li> <li>If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation</li> </ul> | |
| 1.28 | Modifications | If the subject reports unsatisfactory vision or is unable to obtain 20/30 distance visual acuity OU with the lenses, then a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required, however at the Investigator's discretion and based upon their findings on the measured visual acuity and/or over- refraction the investigator may make a modification. Up to two attempts at modification are permitted if necessary, in order to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. | |

| 1.29 | | Follow the fitting guide allowing for at least 10 minutes of settling time between each lens modification attempted. If modifications are required steps 1.21-1.27 will be repeated for each modification. |
|---|---|---|
| 1.30 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. NOTE: The distance visual acuity must be at least 20/30 OU for the lenses to be dispensed. |
| 1.31 | Dispensing Criteria | <ul> <li>The lenses will be dispensed for 2-4 days.</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable general lens fit.</li> </ul> |
| 1.32 | Patient Instructions<br>(Daily Reusable<br>Lenses) | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear reusable basis.</li> <li>No additional lenses will be dispensed.</li> <li>OPTI-FREE® PureMoist® disinfecting solutions will be used to rub, rinse and store the lenses each day.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> </ul> |

## Subjects will be instructed to wear their glasses when not wearing the study lenses. A patient instruction booklet will be provided. **NOTE:** In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the **Product Quality Complaint Form. The lens** will be stored in labeled vial with sterile saline and returned to the Sponsor. 1.33 **Patient Instructions** Instruct the Subject the following: (Daily Disposable The lenses will be worn on a daily wear Lenses) Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed. A new lens will be opened and worn each day. Instruct the subject to bring back all unworn study lenses. Instruct the subject no cleaning or disinfecting solutions will be used for this lens type. If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness. Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study. Subjects will be instructed to wear their glasses when not wearing the study lenses. A patient instruction booklet will be provided.

| | | NOTE: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline and returned to the Sponsor. |
|---|---|---|
| 1.34 | Schedule<br>Follow-up | The subject will be scheduled to return for their follow-up appointment in 3±1 day. NOTE: To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

### VISIT 2

The subjects must present to Visit 2 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| Visit 2: Treatment 1 Follow-up 1 | | | |
|---|---|---|---|
| Step | Procedure | Details | CTP |
| 2.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. | |
| 2.2 | Wear time and<br>Comfortable Wear<br>time with Study<br>lenses | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. | |
| 2.3 | Compliance | Record the subject's compliance with wearing the study lenses. NOTE: Subjects must have worn lenses for at least 6 hours per day To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. | |
| 2.4 | | | |
| 2.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. | |

| 2.6 | Subjective | Record whether the subject's distance and near | |
|---|---|---|---|
| | Acceptance | vision with the lenses is acceptable. | |
| 2.7 | Distance and Near | Measure the distance and near visual acuity | 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |
| | Entrance Visual | OD, OS and OU. Record the results. | The state of the s |
| | Acuity | | |
| | | NOTE: Use the ETDRS 2000 Series Chart 1 | |
| | | or 2 near card placed at 40 cm to measure | |
| | | the Near visual acuity | <u> </u> |
| 2.8 | Distance Over- | Perform a distance over-refraction OD and OS | |
| | Refraction and | using loose lenses outside of the phoropter | |
| | Distance Visual | under ambient room illumination. The | |
| | Acuity | distance over-refraction may also be refined | |
| | | under binocular conditions. Record the results | |
| | | and distance visual acuity OD and OS. | |
| | | The results of the distance over-refraction may | |
| | | also be checked for the impact on near vision | |
| | | under monocular and/or binocular conditions. | |
| 2.9 | Determination of | If the subject reports unsatisfactory vision or is | |
| | Lens Optimization | unable to obtain 20/30 distance visual acuity | |
| | | OU with the lenses, then a modification must | |
| | | be attempted. | |
| | | If the subject reports satisfactory vision with | |
| | | the lenses a modification is not required, | |
| | | however at the Investigator's discretion and | |
| | | based upon their findings on the measured | |
| | | visual acuity and/or over- refraction the | |
| | | investigator may make a modification. | |
| | | Up to two attempts at modification are | |
| | | permitted if necessary, in order to achieve an | |
| | | acceptable distance and near binocular | |
| | | performance for the subject, and to enable | |
| | | them to wear that particular lens type. | |
| | | Follow the fitting guide and steps 1.21-1.27 in | |
| | | Visit 1 Fitting allowing for at least 10 minutes | |
| | | of settling time between each lens | |
| P. | | modification. | 41- |
| 2.10 | Lens Fit Assessment: | Evaluate and grade lens centration, primary | |
| | | gaze movement, upgaze movement and | 3.2 |
| | | tightness (push-up test). | |
| | | The subject should not proceed to wear the | |
| | | lenses if any of the following is observed: | |
| | | presence of limbal exposure (appearance of | |
| | | clear cornea) in any gaze | |
| | | presence of edge lift | |
| | · c | | |

| | | presence of unacceptable movement (excessive or insufficient) in <u>all three</u> movement categories (primary gaze, upgaze, and push-up). If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. | |
|---|---|---|--|
| 2.11 | Collection of unworn<br>lenses (if applicable) | If the subject was fit in the daily disposable lenses at visit 1 collect unworn lenses returned by the subject when lens power has been optimized. If lens power was not changed allow the subject to use the unworn lenses dispensed at | |
| 2.12 | Lens Removal | Visit 1 and dispense enough lenses of the same power to last the subject until their next visit. The study lenses will be removed and | |
| | (Service of Service (Service ) | discarded. | |
| 2.13 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit Lamp Classification Scales will be used to grade the findings. For the conjunctival redness | |
| 2.14 | Insertion of Study<br>Lenses | Dispense the subject a new pair of lenses that match the distance and ADD power of the lenses that were removed in Step 2.12 above. | |
| 2.15 | | | |
| 2.16 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. | |
| 2.17 | Dispensing Criteria | NOTE: The distance visual acuity must be at least 20/30 OU for the lenses to be dispensed. The lenses will be dispensed for 7±1 day. • Distance Snellen acuity equal to or better than 20/30 OU • Subject must indicate that the vision is acceptable. • Subject must indicate that the comfort of the lenses is acceptable. • Lenses must have an acceptable general lens fit. |
|---|---|---|
| 2.18 | Patient Instructions (Reusable Lenses) | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear reusable basis.</li> <li>No additional lenses will be dispensed.</li> <li>OPTI-FREE® PureMoist® disinfecting solutions will be used to rub, rinse and store the lenses each day.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>Subjects will be instructed to bring their habitual contacts or spectacles to the next visit.</li> <li>NOTE: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline and returned to the Sponsor.</li> </ul> |

| 2.20 | Schedule Follow-up | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed.</li> <li>A new lens will be opened and worn each day.</li> <li>Instruct the subject to bring back all unworn study lenses.</li> <li>Instruct the subject no cleaning or disinfecting solutions will be used for this lens type.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>Subjects will be instructed to bring their habitual contacts or spectacles to the next visit.</li> <li>NOTE: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline and returned to the Sponsor.</li> <li>The subject will be scheduled to return for their follow-up appointment in 7±1 day.</li> </ul> |
|---|---|---|

| NOTE: To count the follow-up visit as a day |
|----------------------------------------------|
| of wear the Subject must have worn the |
| study lenses for 6 hours prior to the visit. |

The subjects must present to Visit 3 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 3: Treatment 1 Follow-up 2 | |
|---|---|---|
| Step | Procedure | Details |
| 3.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 3.2 | Wear time and<br>Comfortable Wear<br>time with Study<br>lenses | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |
| 3.3 | Compliance | Record the subject's compliance with wearing the study lenses. NOTE: Subjects must have worn lenses for at least 6 hours per day To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. |
| 3.4 | PRO (CLUE and<br>MRD) and CLDEQ-8<br>Questionnaires | The subject will evaluate the vision characteristics, comfort characteristics, handling characteristics, and visual symptoms of the study lenses using the PRO (CLUE and MRD) questionnaires. |
| 3.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire |
| 3.6 | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. |
| 3.7 | Distance and Near<br>Entrance Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| 3.8 | Visual Performance<br>Distance (4 M)<br>Intermediate (64 cm)<br>Near (40 cm) | Visual performance will be recorded OD, OS, and OU for the following: Distance, Bright Illuminance |

| | | , | |
|---|---|---|---|
| | | High and Low Contrast ETDRS Charts 4 M- HC#1, HC#2, HC#3 and LC#1, LC#2, LC#3 Near, Bright Illuminance Reduced Guillon-Poling Charts Intermediate (64 cm) High Contrast and Low Contrast Near (40 cm) High Contrast and Low Contrast | |
| | | Distance, Dim Illuminance (with <u>Distance</u> goggles) High Contrast ETDRS Charts 4 M-HC#4, HC#5, HC#6 Near, Dim Illuminance (with <u>Near</u> goggles) Reduced Guillon-Poling charts High Contrast Intermediate (64 cm) and Near (40 cm). | |
| | | <ul> <li>NOTE:</li> <li>The room illuminance must be between 7.3 and 7.9 EV (394-597 lux).</li> <li>Distance, HC-1 Chart luminance Acceptable Range 10.5-10.7 EV</li> </ul> | |
| | | <ul> <li>(181-208 cd/m2).</li> <li>Guillon-Poling, Near Chart Luminance Acceptable Range 10.8- 11.1 EV (223-274 cd/m2).</li> <li>Do not use the Mesopic filter for Dim luminance (Dim luminance will be</li> </ul> | |
| 3.9 | Binocular Distance<br>Over-refraction and<br>Distance Visual<br>Acuity | simulated by using the goggles) Perform a binocular over-refraction and record the OD and OS results and distance visual acuity. Note: No lens changes are allowed based on the over-refraction. | Appendix<br>D |
| 3.10 | Lens Fit Assessment: | <ul> <li>Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test).</li> <li>The subject should not proceed to wear the lenses if any of the following is observed:</li> </ul> | |
| | | <ul> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement</li> </ul> | |

| | | (excessive or insufficient) in <u>all three</u> movement categories (primary gaze, upgaze, and push-up). |
|---|---|---|
| | | If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. |
| 3.11 | Collection of unworn lenses (if applicable) | If the first lens type fit on the subject was the daily disposable lenses collect unworn lenses returned by the subject. |
| 3.12 | Lens Removal | Have the subject remove the study lenses and store in saline in a labeled glass vial. Note: Lenses do not need to be stored in a refrigerator. |
| 3.13 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit Lamp Classification Scales will be used to grade the findings. For the conjunctival redness unit increments will be used in the grading. Corneal Staining Assessment will be graded in 1.0 increments. |
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
| 3.14 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the subject's habitual correction in place. |
| | | For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| 3.15 | Schedule<br>Follow-up | The subject will be scheduled to return for their next appointment in 7±3 days. |
| | | NOTE: Subject may wear their habitual spectacles or contact lenses during the washout period. |

The subjects may present to Visit 4 wearing their habitual spectacles or contact lenses, if required for their distance vision.

| | Visit 4: Baseline Treatment 2 | |
|---|---|---|
| Step | Procedure | Details |
| 4.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 4.2 | Subject Reported<br>Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 4.3 | Distance and Near<br>Entrance Visual<br>Acuity | Distance and near Snellen visual acuity will be measured for each eye with the subject's habitual correction in place. |
| | | For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| 4.4 | Lens Removal (if applicable) | Have the subject remove their habitual lenses and store in an approved storage solution. |
| 4.5 | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. For the conjunctival redness (100 to 100 to |
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| 4.6 | Continuance | Determine whether the subject is eligible to continue in the study based on the examination findings. |

| | Visit 4: Treatment 2 Lens Fitting | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 4.7 | Lens Selection | Select the lens pair and power based on the randomization scheme, spherical equivalent refraction and fitting guide for each eye. | Appendix<br>G or H<br>(Fitting<br>Guides) |

| | | Record the Test lens parameters (power and lot number). |
|---|---|---|
| 4.8 | Lens Insertion | Subjects will insert the lenses themselves. If the lens is uncomfortable, inspect for damage and remove, reinsert or replace as necessary. |
| | | Damaged lenses will be stored in labeled vial with sterile saline, and clearly differentiated from the other worn lenses that will be shipped back to the Sponsor. Complete the Quality Product Complaint form. |
| 4.9 | Lens Settling | Allow the study lenses to settle for a minimum of 10 minutes. |
| 4.10 | Determine Visual<br>Satisfaction | Determine if the subject's vision is acceptable with the lenses. Allow the subject to look down a hallway or out of a window for distance vision assessments, and for them to read a book, magazine or similar for near vision. |
| 4.11 | Distance and Near<br>Entrance Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the |
| | | nearest letter OD, OS and OU. |
| 4.12 | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. |
| 4.13 | Subjective Lens Fit<br>Assessment | Evaluate overall lens fit acceptance (acceptable or unacceptable) based on centration, movement and other fitting characteristics. An unacceptable fit is deemed by one of the following criteria: Iimbal exposure at primary gaze or with extreme eye movement; edge lift; excessive movement in primary and up gaze; or |

| | | insufficient movement in all three of the following conditions: primary gaze, up gaze, and Josephson push up. If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. | |
|---|---|---|---|
| 4.14 | Modifications | If the subject reports unsatisfactory vision or is unable to obtain 20/30 distance visual acuity OU with the lenses, then a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required, however at the Investigator's discretion and based upon their findings on the measured visual acuity and/or over- refraction the investigator may make a modification. Up to two attempts at modification are permitted if necessary, in order to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. Follow the fitting guide allowing for at least 10 minutes of settling time between each lens modification attempted. If modifications are required steps 4.7-4.13 will be repeated for each modification. | Appendix<br>G or H<br>(Fitting<br>Guides) |
| 4.15 | | | |
| 4.16 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. NOTE: The distance visual acuity must be at least 20/30 OU for the lenses to be dispensed. | |
| 4.17 | Dispensing Criteria | <ul> <li>The lenses will be dispensed for 3±1 day.</li> <li>Distance Snellen acuity equal to or better than 20/30 OU.</li> </ul> | |

| 4.18 | Patient Instructions (Daily Reusable Lenses) | <ul> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable general lens fit.</li> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear reusable basis.</li> <li>No additional lenses will be dispensed.</li> <li>OPTI-FREE® PureMoist® disinfecting solutions will be used to rub, rinse and store the lenses each day.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for</li> </ul> |
|---|---|---|
| | | <ul> <li>dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>Subjects will be instructed to bring their habitual contacts or spectacles to the next visit.</li> <li>A patient instruction booklet will be provided.</li> </ul> |
| | | NOTE: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline and returned to the Sponsor. |
| 4.19 | Patient Instructions (Daily Disposable Lenses) | <ul><li>Instruct the Subject the following:</li><li>The lenses will be worn on a daily wear basis.</li></ul> |

| | | <ul> <li>Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed.</li> <li>A new lens will be opened and worn each day.</li> <li>Instruct the subject to bring back all unworn study lenses.</li> <li>Instruct the subject no cleaning or disinfecting solutions will be used for this lens type.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses</li> </ul> |
|---|---|---|
| | | <ul> <li>for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>A patient instruction booklet will be provided.</li> <li>NOTE: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site</li> </ul> |
| | | and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline and returned to the Sponsor. |
| 4.20 | Schedule<br>Follow-up | The subject will be scheduled to return for their follow-up appointment in 3±1 day. NOTE: To count the follow-up visit as a day |
| | | of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

The subjects must present to Visit 5 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 5: Treatment 2 Follow-up 1 | |
|---|---|---|
| Step | Procedure | Details |
| 5.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. Record any adverse events or medical history changes from the previous study visit. |
| 5.2 | Wear time and<br>Comfortable Wear<br>time with Study<br>lenses Wear Time | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. |
| 5.3 | Compliance | Record the subject's compliance with wearing the study lenses. NOTE: Subjects must have worn lenses for at least 6 hours per day To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. |
| 5.4 | | |
| 5.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 5.6 | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. |
| 5.7 | Distance and Near<br>Entrance Visual<br>Acuity | Measure the distance and near visual acuity OD, OS and OU. Record the results. NOTE: Use the ETDRS 2000 Series Chart 1 or 2 near card placed at 40 cm to measure the Near visual acuity |
| 5.8 | Distance Over-<br>Refraction and<br>Distance Visual<br>Acuity | Perform a distance over-refraction OD and OS using loose lenses outside of the phoropter under ambient room illumination. The distance over-refraction may also be refined under binocular conditions. Record the results and distance visual acuity OD and OS. The results of the distance over-refraction may also be checked for the impact on near vision under monocular and/or binocular conditions. |

| 5.9 | Determination of Lens Optimization | If the subject reports unsatisfactory vision or is unable to obtain 20/30 distance visual acuity OU with the lenses, then a modification must be attempted. If the subject reports satisfactory vision with the lenses a modification is not required, however at the Investigator's discretion and based upon their findings on the measured visual acuity and/or over- refraction the investigator may make a modification. Up to two attempts at modification are permitted if necessary, in order to achieve an acceptable distance and near binocular performance for the subject, and to enable them to wear that particular lens type. Follow the fitting guide and steps 4.7-4.13 in Visit 4 Fitting allowing for at least 10 minutes of settling time between each lens modification. | Appendix G or H (Fitting Guides) |
|---|---|---|---|
| 5.10 | Lens Fit Assessment: | <ul> <li>Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test).</li> <li>The subject should not proceed to wear the lenses if any of the following is observed:</li> <li>presence of limbal exposure (appearance of clear cornea) in any gaze</li> <li>presence of edge lift</li> <li>presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up).</li> <li>If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form.</li> </ul> | |
| 5.11 | Collection of unworn lenses (if applicable) | If the subject was fit in the daily disposable lenses at visit 4 collect unworn lenses returned by the subject when lens power has been optimized. | |

| 5.12 | Lens Removal | If lens power was not changed allow the subject to use the unworn lenses dispensed at Visit 4 and dispense enough lenses of the same power to last the subject until their next visit. The study lenses will be removed and |
|---|---|---|
| 3.12 | Lens Kemovai | discarded. |
| 5.13 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit Lamp Classification Scales will be used to grade the findings. For the conjunctival redness unit increments will be used in the grading. Corneal Staining Assessment will be graded in 1.0 increments. |
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |
| 5.14 | Insertion of Study<br>Lenses | Dispense the subject a new pair of lenses that match the distance and ADD power of the lenses that were removed in Step 5.12 above. |
| 5.15 | | |
| 5.16 | Distance and Near<br>Exit Visual Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| g | | NOTE: The distance visual acuity must be at least 20/30 OU for the lenses to be dispensed. |
| 5.17 | Dispensing Criteria | <ul> <li>The lenses will be dispensed for 7±1 day.</li> <li>Distance Snellen acuity equal to or better than 20/30 OU</li> </ul> |
| | | <ul> <li>Subject must indicate that the vision is acceptable.</li> <li>Subject must indicate that the comfort of the lenses is acceptable.</li> <li>Lenses must have an acceptable general lens fit.</li> </ul> |

| 5.18 | Patient Instructions (Reusable Lenses) | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear reusable basis.</li> <li>No additional lenses will be dispensed.</li> <li>OPTI-FREE® PureMoist® disinfecting solutions will be used to rub, rinse and store the lenses each day.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>Subjects will be instructed to bring their habitual contacts or spectacles to the next visit.</li> <li>NOTE: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline and returned to the Sponsor.</li> </ul> |
|---|---|---|
| 5.19 | Patient Instructions (Daily Disposable Lenses) | <ul> <li>Instruct the Subject the following:</li> <li>The lenses will be worn on a daily wear basis.</li> <li>Only enough lenses will be dispensed to the subject to wear for the required number of days until their follow-up visit. No additional lenses will be dispensed.</li> <li>A new lens will be opened and worn each day.</li> <li>Instruct the subject to bring back all unworn study lenses.</li> </ul> |

| | | <ul> <li>Instruct the subject no cleaning or disinfecting solutions will be used for this lens type.</li> <li>If determined necessary by the Investigator sterile non-preserved rewetting drops may be dispensed to be used as needed for dryness.</li> <li>Subjects will be instructed to wear lenses for a minimum of 6 hours a day, every day during the study.</li> <li>Subjects will be instructed to wear their glasses when not wearing the study lenses.</li> <li>Subjects will be instructed to bring their habitual contacts or spectacles to the next visit.</li> </ul> |
|---|---|---|
| | | NOTE: In the event a lens is lost or damaged, the subject will return to the investigator site for replacement. As much as reasonably possible, a damaged lens should be returned to the investigational site and then returned to the Sponsor. If lens damage is present, complete the Product Quality Complaint Form. The lens will be stored in labeled vial with sterile saline and returned to the Sponsor. |
| 5.20 | Schedule<br>Follow-up | The subject will be scheduled to return for their follow-up appointment in 7±1 day. NOTE: To count the follow-up visit as a day of wear the Subject must have worn the study lenses for 6 hours prior to the visit. |

The subjects must present to Visit 6 wearing the study lenses. To be counted as a day of wear the lenses need to have been worn for at least six (6) hours prior to the visit.

| | Visit 6: Treatment 2 Follow-up 2 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 6.1 | Adverse Events and<br>Concomitant<br>Medications Review | Review the subject's concomitant medications and record any changes from the previous study visit. | So a |

| | T | D 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | 5 |
|---|---|---|---|
| | | Record any adverse events or medical history changes from the previous study visit. | |
| 6.2 | Wear time and<br>Comfortable Wear<br>time with Study<br>lenses | Record the hours the subject has worn the study lenses and the comfortable wear time on the day of follow-up. | |
| 6.3 | Compliance | Record the subject's compliance with wearing the study lenses. NOTE: Subjects must have worn lenses for at least 6 hours per day To be counted as a day of wear at this visit the Subject must have worn the study lenses for 6 hours prior to the visit. | |
| 6.4 | | | |
| 6.5 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire | |
| 6.6 | Subjective<br>Acceptance | Record whether the subject's distance and near vision with the lenses is acceptable. | |
| 6.7 | Distance and Near<br>Entrance Visual<br>Acuity | Distance and near Snellen visual acuity will be measured for each eye with the study contact lenses in place. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. | |
| 6.8 | Visual Performance<br>Distance (4 M)<br>Intermediate (64 cm)<br>Near (40 cm) | Visual performance will be recorded OD, OS, and OU for the following: Distance, Bright Illuminance High and Low Contrast ETDRS Charts 4 M- HC#1, HC#2, HC#3 and LC#1, LC#2, LC#3 Near, Bright Illuminance Reduced Guillon-Poling Charts Intermediate (64 cm) High Contrast and Low Contrast Near (40 cm) High Contrast and Low Contrast Distance, Dim Illuminance (with Distance goggles) High Contrast ETDRS Charts 4 M-HC#4, HC#5, HC#6 | |

| | | Near, Dim Illuminance (with Near goggles) Reduced Guillon-Poling charts High Contrast Intermediate (64 cm) and Near (40 cm). NOTE: • The room illuminance must be between 7.3 and 7.9 EV (394-597 lux). • Distance, HC-1 Chart luminance Acceptable Range 10.5-10.7 EV (181-208 cd/m2). • Guillon-Poling, Near Chart Luminance Acceptable Range 10.8-11.1 EV (223-274 cd/m2). • Do not use the Mesopic filter for Dim luminance (Dim luminance will be simulated by using the goggles) | |
|---|---|---|---|
| 6.9 | Binocular Distance<br>Over-refraction and<br>Distance Visual<br>Acuity | Perform a binocular over-refraction and record the OD and OS results and distance visual acuity. Note: No lens changes are allowed based on the over-refraction. | Appendix<br>D |
| 6.10 | Lens Fit Assessment: | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). The subject should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift • presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up). If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. | |

| 6.11 | Collection of unworn lenses (if applicable) | If the second lens type fit on the subject was<br>the daily disposable lenses collect unworn<br>lenses returned by the subject. |
|---|---|---|
| 6.12 | Lens Removal | Have the subject remove the study lenses and store in saline in a labeled glass vial. NOTE: Lenses do not need to be stored in a refrigerator. |
| 6.13 | Biomicroscopy | Perform biomicroscopy OD and OS. Slit Lamp Classification Scales will be used to grade the findings. For the conjunctival redness 0.5 unit increments will be used in the grading. Corneal Staining Assessment will be graded in 1.0 increments. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. |

### FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| | Final Evaluation | | |
|---|---|---|---|
| Step | Procedure | Details | CTP |
| F.1 | Final Exam Form | Indicate if the subject completed the study successfully. If subject discontinued from the study, indicate the reason. | |
| F.2 | Subjective<br>spherocylindrical<br>Refraction | Perform bare-eye subjective spherocylindrical refraction with a phoropter and record the best corrected <u>distance</u> visual acuity to the nearest letter (OD, OS, and OU). | |
| F.3 | Exit Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. | |

# 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected at a minimum:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate
- Date and time of the visit and all procedures completed at the unscheduled visit
- Review of adverse event and concomitant medications
- Documentation of any test article dispensed or collected from the subject, if applicable
- Slit lamp findings (using the Slit Lamp Classification Scale)

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pretreatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information will be collected during an unscheduled visit.

| | Unscheduled Visit | |
|---|---|---|
| Step | Procedure | Details |
| U.1 | Chief Complaints | Record the subject's chief complaints for reasons for the unscheduled visit |
| U.2 | Adverse Events and<br>Concomitant Medications<br>Review | Review the subject's concomitant medications and record any changes from the previous study visit. |
| U.3 | Subject Reported Ocular<br>Symptoms | Subjects will respond to a verbal open-<br>ended symptoms questionnaire. |
| U.4 | Entrance VA | Record the entrance distance and near visual acuity (OD, OS and OU) to the nearest letter. For near measures use the ETDRS 2000 Series Chart 1 or 2. The acuity will be recorded to the nearest letter OD, OS and OU. |
| U.5 | Subjective Sphero-<br>cylindrical Refraction | An optimal, binocular balanced distance sphero-cylindrical refraction will be performed. Record the refraction and distance visual acuity to the nearest letter. |
| U.6 | Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. |

| | Unscheduled Visit | |
|---|---|---|
| | | For the conjunctival redness 0.5 unit increments will be used in the grading. Corneal Staining Assessment will be graded in 1.0 increments. |
| U.7 | Lens Dispensing | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops may be instilled. Additional study lenses may be dispensed |
| | Zem Dispensing | when required. |
| U.8 | Lens Fit Assessment: | Evaluate and grade lens centration, primary gaze movement, upgaze movement and tightness (push-up test). |
| | | The subject should not proceed to wear the lenses if any of the following is observed: • presence of limbal exposure (appearance of clear cornea) in any gaze • presence of edge lift • presence of unacceptable movement (excessive or insufficient) in all three movement categories (primary gaze, upgaze, and push-up). |
| | | If either lens is deemed unacceptable, the subject will be discontinued from the study. Remove the lenses, perform a slit-lamp evaluation, and complete the Final Evaluation form. |
| U.9 | Exit Visual Acuity | Record the subject's exit distance and near visual acuity (OD, OS and OU) to the nearest letter. |
| | | For near measures use the ETDRS 2000<br>Series Chart 1 or 2. The acuity will be<br>recorded to the nearest letter OD, OS and<br>OU. |

# 7.4. Laboratory Procedures

Not Applicable

#### 8. SUBJECTS COMPLETION/WITHDRAWAL

# 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- provided informed consent
- they are eligible
- completed all study visits

# 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject death during the study period
- Subject withdrawal of consent
- Subject not compliant to protocol
- Subject lost to follow-up
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant)
- Subject develops significant or serious adverse events causing discontinuation of study lens wear
- Subjects who have experienced a Corneal Infiltrative Event (CIE)
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment)
- Subject missed two consecutive study visits
- Subject not compliant with study lens wear schedule
- Subject not successfully dispensed due to lack of efficacy and safety including poor vision, poor comfort or unacceptable fit

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled)
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study
- Record the spherocylindrical refraction with best corrected distance visual acuity
- Collect used test article(s) (worn or brought to the visit) from the subject and discard them, unless otherwise stated in Section 6.7
- Collect all unused test article(s) from the subject

An additional subject may be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

#### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications and therapies are medications or therapies that contraindicate contact lens wear. See the Exclusion criteria for specific details.

### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Major protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked, and corrective actions implemented as appropriate.

If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

#### 11. STUDY TERMINATION

If more than 2 subjects in the investigational soft contact lens group develop serious expected (e.g., definite or probable MK) or unexpected device related adverse events, the study will be suspended. Upon review and consultation with IRB, DMC, and JJV safety review committee, the study may be terminated. This potential stopping rule is established based on our trial involving approximately 200 subjects wearing the investigational soft contact lens for up to 3 years with an assumed MK rate that is below 0.2% per patient-year. The rate of 0.2% per patient year is the established rate for extended wear lenses in adults, which was requested by the FDA as a criterion for evaluating a contact lens for pediatric use in an FDA response to a pre-IDE submission. To be conservative, 200 independent patient years were used in the calculation. The probability of observing 2 cases or more incidents of MK is 0.061, and 3 cases or more incidents of MK is 0.007 (given a MK rate of 0.2% per patient year).

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to

specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated, as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

# 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)"
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site
- Lens replacements that occur due to drops/fall-outs
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency (i.e. tears, rips, etc.), only in situations where there is no deficiency alleged by the subject

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness)
- Who received the complaint
- Study number
- Clinical site information (contact name, site ID, telephone number)
- Lot number(s)
- Unique Subject Identifier(s)
- Indication of who first observed complaint (site personnel or subject)

- OD/OS indication, along with whether the lens was inserted
- Any related AE number if applicable
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.)
- Eye Care Provider objective (slit lamp) findings if applicable
- Confirmation of product availability for return (and tracking information, if available), or rationale if product is not available for return

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device. **NOTES:** 

*Note 1* to entry: This definition includes events related to the investigational medical device or the comparator.

*Note 2* to entry: This definition includes events related to the procedures involved. *Note 3* to entry: For users or other persons, this definition is restricted to events related to investigational medical devices."<sup>1</sup>

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study
- 2. Was present prior to the study but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states
- 3. Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event

Serious Adverse Event (SAE) – An SAE is any untoward medical occurrence that:

- Results in death
- Is life threatening
- Requires in-patient hospitalization or prolongation of existing hospitalization

- Results in persistent or significant disability/incapacity (e.g., a sight threatening event, a significant persistent or permanent change, impairment, damage, or disruption to the subject's body)
- Is a congenital anomaly/birth defect, or
- Requires intervention to prevent permanent damage (the use of the test article resulting in a condition which requires medical or surgical intervention to preclude permanent impairment of the body structure or a body function). Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered an SAE when, based upon appropriate medical judgment, they may jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the outcomes listed in the above definition

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – Those events that are usually symptomatic and warrant discontinuation (temporary or permanent) of the test article (excluding Serious Adverse Events).

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of > 2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation > 2 weeks

**Non-Significant Adverse Events** — Those conditions that are usually asymptomatic and usually do not warrant discontinuation (temporary or permanent) of the test article. However, the Investigator may choose to treat as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis
- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device.

#### **NOTES:**

*Note 1* to entry: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

*Note 2* to entry: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device."

Unanticipated Adverse Device Effect (UADE) – Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

# 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in Section 13.1)
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related; unlikely related; possibly related; related see definition in Section 13.2.1)
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild; moderate; severe for all events see definition in Section 0)
- Outcome not recovered or not resolved; recovering or resolving; recovered or resolved with sequelae; recovered or resolved; death related to adverse event; unknown

• Actions Taken – none; temporarily discontinued; permanently discontinued; other

# 13.2.1. Causality Assessment

**Causality Assessment** – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely
- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge

# 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities

#### 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begins when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs. He/she will complete the Adverse Event /eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom)
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.)
- Date the clinical site was notified
- Date and time of onset
- Date and time of resolution
- Adverse event classification, severity, and relationship to test articles, as applicable
- Treatment regimen instituted, including concomitant medications prescribed, in accordance with applicable licensing requirements
- Any referral to another health care provider if needed
- Outcome, ocular damage (if any)
- Likely etiology
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator.

Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

# 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.

# 13.4.1. Reporting Adverse Events to Sponsor

# Serious/Significant Adverse Events

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail, fax, or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations

# **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

# 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

# 13.4.3. Event of Special Interest

None

# 13.5. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes. At the Investigator's discretion, the study participant may be followed by the Investigator through delivery. However, this data will not be collected as part of the clinical study database. Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

#### 14. STATISTICAL METHODS

#### 14.1. General Considerations

All data summaries and statistical analyses will be performed using the Statistical Analysis System (SAS) software Version 9.4 (SAS Institute, Cary, NC). Throughout the analysis of data, the results for each subject/eye will be used when available for summarization and statistical analysis. Unscheduled visits will be summarized separately and will be excluded from the statistical analysis.

Summary tables (Descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation [SD], median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

Summaries will be presented by study lens type and will be performed separately by completion status (Safety Population or Per-Protocol Population). All analyses will be conducted on per-protocol population (see Section 14.3).

# 14.2. Sample Size Justification

A total of approximately 50 eligible subjects will be enrolled into the study at this site. At least 40 subjects will complete this study. There have been no prior historical dispensing studies in presbyopes with the Test article to determine sample size. This is a pilot study and the sample size calculation was not based on any power analysis. The collected data will be used to design future trials.

Using the POWER procedure in SAS 9.4, below is the summary of sample size required based on the different assumptions of the true difference. Each study hypothesis is tested with at least 90% of statistical power and 2-sided type I error of 0.05.

### • lens centration and lens movement

| | Actual Odds Ratio | Control Lens Proportion | # of eyes needed | Power |
|---|-------------------|-------------------------|------------------|-------|
| | 1.0 | 0.75 | 571 | 0.8 |
| ı | 1.5 | 0.75 | 164 | 0.8 |
| ı | 2.0 | 0.75 | 100 | 0.8 |

# 14.3. Analysis Populations

#### **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

### **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock (Per-Protocol Population). Justification of excluding subjects with protocol deviations in the Per-Protocol Population set will be documented in a memo to file.

#### **Intent-to-Treat (ITT) Population:**

All subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

#### 14.4. Level of Statistical Significance

All planned analysis for this study will be conducted with an overall type I error rate of 5%.

# 14.5. Primary Analysis

Primary efficacy analysis:

The lens centration and lens movement outcomes will be converted to a binary response where 1= lens is centered or have optimal lens movement, and 0=otherwise.

The proportion of response ("1") will be analyzed using a generalized linear mixed model with a binary distribution and logit link function for all questions. Each model will include the experimental design factors: lens, period and lens by period interaction as fixed effects; and site and subject nested in site as random effects. Other baseline characteristics known to be important such as subject group (myope/hyperope), age, gender, and/or add power will be included as fixed covariates when appropriate. The covariance between residual errors from two eyes from the same subject at the same lens wearing period will be selected based on the finite-sample corrected Akaike's Information Criterion. Covariance structures considered may include: Homogenous compound symmetry (CS) and Unstructured covariance structure (UN). The structure that returns the lowest Akaike Information Criteria Corrected (AICC) will be selected as the structure that best fit the data.

Comparisons between the study lenses will be carried out using two-sided 95% confidence intervals of odds ratios (odds ratio calculated as Test / Control) for each individual question. Non-inferiority will be concluded if the lower limit is above 0.67. Superiority will be concluded if the lower limit is above 1.0.

# 14.6. Secondary Analysis

Secondary efficacy analysis:

CLUE handling scores will be analyzed using a linear mixed model adjusting for baseline values as fixed covariates. The model will include the experimental design factors: lens, period and lens by period interaction as fixed effects. Other baseline characteristics known to be important such as subject group (myope/hyperope), age, gender, and/or add power will be included as fixed covariates when appropriate. The covariance between residual errors from the same subject across lens wearing periods will be selected based on the finite-sample corrected Akaike's Information Criterion. Covariance structures considered may include: Homogenous compound symmetry (CS) and Unstructured covariance structure (UN). The structure that returns the lowest Akaike Information Criteria Corrected (AICC) will be selected as the structure that best fit the data.

Comparisons between the Test lens and Control lens will be carried out using 95% confidence intervals constructed of least-square means (LSM) differences (Test minus Control) from the linear mixed model. The non-inferiority of the Test lens relative to the Control will be concluded if the lower confidence limit of LSM difference is above the non-inferiority margin -5. The superiority will be established if the lower confidence limit is above 0.

In all models, the Kenward and Roger method<sup>6</sup> will be used for the calculation of the denominator of degrees of freedom.

# 14.7. Other Exploratory Analyses

Not Applicable

# 14.8. Interim Analysis

Not Applicable

# 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of missing values will be included in the summary tables and listings.

Subject dropout is expected to be one of the main reasons of missing data in this clinical trial. Past clinical trials don't provide the evidence that subject dropout is systematic or not-at-random. To evaluate the impact of missing data, sensitivity analysis will be conducted using multiple imputation methods if the proportion of subject dropout is greater than the 15%. The SAS/STAT procedures PROC MI and PROC MIANALYZE will be utilized with a parametric regression method used to make at least 5 imputations.

# 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

# 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using an EDC system (Bioclinica). An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJV database manager and sent to JJV for analysis.

External Date Sources for this study include: Not Applicable

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011.<sup>1</sup>

# 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

### 16. DATA MANAGEMENT

# 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

# 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

# 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

#### 17. MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent amendments, and regulatory requirements are maintained
- Ensuring the rights and wellbeing of subjects are protected
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel
- Ensuring that protocol deviations are documented with corrective action plans, as applicable
- Ensuring that the clinical site has sufficient test article and supplies
- Clarifying questions regarding the study
- Resolving study issues or problems that may arise

• Reviewing of study records and source documentation verification in accordance with the monitoring plan

### 18. ETHICAL AND REGULATORY ASPECTS

# 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

# 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, Section 4 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>3</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with Section 8 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements.

# 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol and, if applicable, amendments
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information) and amendments
- Sponsor-approved subject recruitment materials
- Information on compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB)
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects
- Any other documents that the IEC/IRB requests to fulfill its obligation
This study will be undertaken only after IEC/IRB has given full approval of the final protocol, amendments (if any), the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol amendments
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure amendments or new edition(s)
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol amendments that increase subject risk, the amendment and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

## 18.4. Informed Consent

Each subject must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH<sup>2</sup> and ISO 14155<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

# 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States<sup>5</sup> and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their investigation related activities that, as part of the investigation will have access to the CRFs and subject records

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations. The Sponsor ensures that the personal data will be:

- processed fairly and lawfully
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes
- adequate, relevant, and not excessive in relation to said purposes
- accurate and, where necessary, kept current

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ICH/GCP guidelines,<sup>2</sup> the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH/GCP<sup>2</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

## 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study
- Scheduling a study visit outside the subject's acceptable visit range

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution
- Case Report Form signature
- Completion of any follow-up action items

## 21. PUBLICATION

This study will be registered on ClinicalTrials.gov by the Sponsor.

#### 22. REFERENCES

- 1. ISO 14155:2011: Clinical Investigation of Medical Devices for Human Subjects Good Clinical Practice. Available at: https://www.iso.org/standard/45557.html
- 2. International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP). Available at: http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. Available at: https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- 4. United States (US) Code of Federal Regulations (CFR). Available at: https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR
- 5. Health Information Portability and Accountability Act (HIPAA). Available at: https://www.hhs.gov/hipaa/for-professionals/privacy/index.html
- Keselman HJ, Algina J, Kowalchuk RK, Wolfinger RD. A Comparison of Two Approaches for Selecting Covariance Structures in the Analysis of Repeated Measures. Communications in Statistics—Simulation and Computation. 1998;27:591-604.
- 7. Kenward MG, Roger JH. Small Sample Inference for Fixed Effects from Restricted Maximum Likelihood. *Biometrics*. 1997;53:983–997.

# APPENDIX A: PATIENT REPORTED OUTCOMES (STUDY QUESTIONNAIRES)







PRO SPECIFICATIO 1 Final 2019-05-28 

5

PRO SPECIFICATIO







10


Confidential




Confidential











| 28 |
|----|
|----|





# APPENDIX B: PATIENT INSTRUCTION GUIDE

The Patient Instruction Guide will be provided separately.

# APPENDIX C: PACKAGE INSERT (APPROVED PRODUCT)

Dailies Total 1® Multifocal Contact Lenses



# DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) Soft

Contact Lenses for Daily Disposable Wear

IMPORTANT: This package insert is effective as of March 2016 and applicable to the deleficon A contact lenses described below. Please read carefully and keep this information for future use. This package insert is intended for the eye care professional, but should be made available to patients upon request. The eye care professional should provide the patient with appropriate instructions that pertain to the patient's prescribed lenses. Copies of this package insert are available without charge from Alcon by calling Customer Service at 1-800-241-5999 or download from our website at www.alcon.com. In addition, a Patient Instruction Booklet is available which is recommended to be given to patients.



CAUTION: Federal law (United States) restricts this device to sale by or on the order of a licensed eye care professional.

#### PRODUCT DESCRIPTION

DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) soft contact lenses are made from a lens material that is 33% water and 67% (dele ilcon A) polymer, a silicone containing hydrogel with added phosphatidylcholine. The core lens material containing 33% water transitions through a water gradient to a hydrogel surface layer that exceeds 80% water. Lenses contain the color additive copper phthalocyanine, a light blue tint, which makes them easier to see when handling.

#### **Lens Properties**

Refractive Index hydrated: 1.42

Light Transmittance: 93% (@ 610 nm, -1.00D)
 Oxygen Permeability (Dk): 140 x 10<sup>-11</sup> (cm²/sec)(ml

O<sub>2</sub>/ml x mm Hg), measured at 35° C (intrinsic Dk-Coulometric

method)

Water Content: 33% by weight in normal

saline

Surface Water Content: ≥ 80%

#### **Lens Parameters**

Diameter Range
 Spherical Power Range
 Base Curve Range
 8.0 to 9.2 mm

#### Lens Parameters Available<sup>1</sup>

#### DAILIES TOTAL1\* (delefilcon A) spherical

Chord Diameter: 14.1 mm

Center Thickness: 0.09 mm @ -3.00D (varies)

with power)

Base Curve:
 8.5 mm

Powers: -0.50 to -6.00D (0.25D

steps); -6.50 to -12.00D (0.50D steps) +0.50 to +6.00D (0.25D steps)

#### DAILIES TOTAL1\* Multifocal (delefilcon A)

Chord Diameter: 14.1 mm

Center Thickness: 0.09 mm @ -3.00D (varies)

with power)

Base Curve:
 8.5 mm

Powers: +6.00D to -10.00D (0.25D steps) ADD: LO, MED, HI

NOTE: Hereafter, DAILIES TOTAL1\* spherical lenses and DAILIES TOTAL1\* Multifocal contact lenses will simply be referred to as deleficon A contact lenses unless product distinction is necessary.

#### ACTIONS

When hydrated and placed on the cornea, delefilcon A contact lenses act as a refracting medium to focus light rays on the retina.

# INDICATIONS (USES)

DAILIES TOTAL1\* (delefilcon A) spherical soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes with up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual acuity.

DAILIES TOTAL1\* Multifocal (delefilcon A) soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) and/or presbyopia in phakic or aphakic persons with non-diseased eyes who may require a reading addition of +3.00 (D) or less and who may have up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual acuity.

The lenses are to be prescribed for single use, daily disposable wear. The lenses are not intended to be cleaned or disinfected and should be discarded after a single use.

# CONTRAINDICATIONS (REASONS NOT TO USE)

DO NOT use delefilcon A contact lenses when any of the following exists:

Inflammation or infection of the anterior chamber of the eye

- Active disease, injury or abnormality affecting the cornea, conjunctiva, or eyelids
- Microbial infection of the eye
- Insufficiency of lacrimal secretion (dry eye) that interferes with contact lens wear
- · Comeal hypoesthesia (reduced comeal sensitivity)
- Use of any medication that is contraindicated or interferes with contact lens wear, including eye medications
- Any systemic disease which may be exacerbated by or interferes with contact lens wear
- Allergic reactions or ocular irritation of the ocular surfaces or adnexa that may be caused by or exaggerated by the wearing of contact lenses
- Patient history of recurring eye or eyelid infections, adverse effects associated with contact lens wear, intolerance or abnormal ocular response to contact lens wear
- . If eyes become red or irritated

#### WARNINGS

Advise patients of the following warnings pertaining to contact lens wear:

- Problems with contact lenses and lens care products could result in serious injury to the eye. t is essential that patients follow their eye care professional's directions and all labeling instructions for proper use of lenses and lens care products.
   Serious eye problems, including corneal ulcers, can develop rapidly and lead to loss of vision.
- Daily wear lenses are not indicated for overnight wear, and patients should be instructed not to wear lenses while sleeping. Clinical study results have shown that the risk of serious adverse reactions is increased when contact lenses are worn overnight?
- Studies<sup>2</sup> have shown that contact lens wearers who are smokers have a higher incidence of adverse reactions than nonsmokers.
- If a patient experiences eye discomfort, foreign body sensation, excessive tearing, vision changes, or redness of the eye, the patient should be instructed to immediately remove lenses and promptly contact his or her eye care professional. It is recommended that contact lens wearers see their eye care professional regularly as directed.

#### PRECAUTIONS

To prevent damage to the eyes or to the contact lenses, the following precautions should be taken:

Special Precautions for the Eye Care Professional:
Due to the small number of patients enrolled in the clinical investigation of lenses, all refractive powers, design configurations, or lens parameters available in the lens material are not evaluated in significant numbers. Consequently when selecting an appropriate lens design and parameters, the eye care professional should consider all characteristics of the lens that can affect lens performance and ocular health, including oxygen permeability, central and peripheral thickness and optic zone diameter. The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction; therefore the continuing ocular health of the patient and lens performance on the eye should be carefully evaluated on initial dispensing and monitored on an ongoing basis by the prescribing eye care professional.

- Fluorescein, a yellow dye, should not be used while the lenses are on the patient's eyes. The lenses absorb this dye and become discolored. Whenever fluorescein is used, the eyes should be flushed thoroughly with sterile saline solution that is recommended for in eye use prior to inserting lenses. Avoid dispensing saline from an aerosol can directly into the eye.
- Patients who wear contact lenses to correct presbyopia may not achieve the best possible corrected visual acuity for either far or near vision. Visual requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.
- Before leaving the eye care professional's office, the patient should be able to promptly remove their lenses or should have someone else available who can remove their lenses for them.
- Eye care professionals should instruct the patient to remove the lenses immediately if the eye becomes red or irritated.
- Routine eye examinations are necessary to help assure the continued health of the patient's eyes. Eye care professionals should make arrangements with the patient for appropriate

follow-up visits. Alcon recommends that patients see their eye care professional once each year, or more often, as recommended by the eye care professional.

W900038292

- Diabetics may have reduced corneal sensitivity and thus are more prone to corneal injury and do not heal as quickly or completely as non-diabetics.
- Visual changes or changes in lens tolerance may occur during pregnancy or use of oral contraceptives. Caution patients accordingly.

#### Eye Care Professionals should carefully instruct patients about the following safety precautions: Handling Precautions:

- Be sure that before leaving the eye care professional's office the patient is able to promptly remove lenses or have someone else available to remove them.
- Good hygiene habits help promote safe and comfortable lens wear. Always wash, rinse and thoroughly dry hands with a lint-free towel before handling lenses.
- REMOVE A LENS IMMEDIATELY if an eye becomes red or irritated
- Always handle lenses carefully. Never use tweezers or other sharp objects such as fingernails to remove lenses from the lens container unless specifically indicated for that use.
- Do not use if blister package is damaged or not sealed completely. This may result in product contamination which can lead to a serious eye infection.
- Ensure that the correct lens for each eye is available. Shake
  the blister pack gently prior to opening. Remove the lens from
  the blister pack by carefully pouring the lens onto the palm of
  your clean hand. Ensure the lens is right side out. Inspect
  lenses prior to insertion. Do not insert damaged lenses.
- To insert lenses:
  - Wash and rinse hands thoroughly and dry completely with a clean, lint free towel before handling lenses.
  - Place a lens on the tip of your clean and dry right or left index finger, place the middle finger of the same hand close to lower eyelashes and pull down the lower eyelid.
  - Use the fingers of the other hand to lift the upper eyelid.
  - Place the lens directly on the eye (cornea) and gently roll finger away from the lens.
  - Look down and slowly remove the hand, releasing the lower lid.
  - Look straight ahead and slowly remove the other hand, releasing the upper lid.
  - Blink gently.
- To remove lenses:
  - Wash and rinse hands thoroughly and dry completely with a clean, lint free towel before handling lenses.
     Make sure hands are clean and completely dry.
  - Blink fully several times.
  - While looking up, slide the lens down onto the white part of the eye.
  - Remove the lens by pinching gently between the thumb and forefinger. Do not pinch the eye tissue.
  - If the lens is difficult to grasp, dry fingers once more and try again. Do not use rewetting drops in this instance.
- If a lens decenters on the eye, it may be possible to recenter it by:
  - Closing the eye and massaging the lens into place, or
  - Looking in the direction of the lens and blinking gently, or
     Gently pushing the off-centered lens onto the comea with light finger pressure on the edge of the upper or lower
- eyelid.

  If a lens tears in the eye it will feel uncomfortable. Advise wearers it is impossible to lose a contact lens or part of a contact lens behind the eye and to remain calm. Lens pieces

contact lens benind the eye and to remain calm. Lens pieces may be removed by pinching them as for normal lens removal, carefully avoiding pinching the eye tissue. If the lens pieces do not seem to remove easily, rinsing with saline is recommended. If this does not help, the wearer should contact an eye care professional for assistance.

# Lens Wearing Precautions:

- Patients should never exceed the prescribed wearing schedule regardless of how comfortable the lenses feel. Doing so may increase the risk of adverse effects.
- The lens should move freely on the eye at all times. If the lens sticks (stops moving) on the eye, follow the recommended directions in the Care for a Sticking Lens section. If non-movement of the lens continues, the patient should be instructed to consult their eye care professional immediately.

- The eye care professional should be consulted about wearing lenses during water sports and water related activities.
   Exposure to water or other non-sterile liquids while wearing contact lenses in activities such as swimming, water skiing, and hot tubs may increase the risk of ocular infection, including but not limited to Acanthamoeba keratitis.
- Never allow contact lenses to come into contact wi h non-sterile liquids (including tap water and saliva) as microbial contamination can occur, which may lead to permanent eye damage.
- Eye irritation, infection, or lens damage may result if cosmetics, lotion, soap, cream, hair spray, deodorant, aerosol products or foreign particles come in contact with lenses.
- Environmental fumes, smoke, and vapors should be avoided in order to reduce the chance of lens contamination or physical trauma to the cornea.
- Lenses should be disposed of each day upon removal from the eve
- Discard any lens which has become dehydrated or damaged.
   Replace with a sterile, fresh, new lens.
- Note the correct lens power for each eye to prevent getting them mixed up
- Always carry spare lenses with you or have back-up spectacles available.
- Do not share lenses with anyone as this may spread micro-organisms which could result in serious eye health problems.
- Do not use lenses beyond their expiration date.

#### Other Topics to Discuss with Patients:

- Periodic eye examinations are extremely important for contact lens wearers. Schedule and conduct appropriate follow-up examinations to determine ocular response. Alcon recommends that patients see their eye care professional once each year or as recommended by the eye care professional.
- Certain medications may cause dryness of the eye, increased lens awareness, lens intolerance, and blurred vision or visual changes. These include, but are not limited to, antihistamines, decongestants, diuretics, muscle relaxants, tranquilizers, and those for motion sickness. Caution patients using such medications accordingly and prescribe proper remedial measures.
- Visual changes or changes in lens tolerance may occur during pregnancy or use of oral contraceptives. Caution patients accordingly.

# Who Should Know that the Patient is Wearing Contact Lenses:

- Patients should inform their health care practitioners that they are wearing contact lenses.
- Patients should inform their employers that they are wearing contact lenses. Some jobs may require the use of eye protection equipment or may require that contact lenses not be worn

It is strongly recommended that patients be provided with a copy of the DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal Contact Lenses (delefilcon A) Patient Instruction Booklet available from Alcon and understand its contents prior to dispensing the lenses.

#### ADVERSE EFFECTS

Patients should be instructed to check eyes regularly to make sure they look well, feel comfortable and vision is clear. Potentially serious complications are usually accompanied by one or more of the following signs or symptoms:

- Moderate to severe eye pain not relieved by removing the lens
- Foreign body sensation
- Excessive watering or other eye secretions including mucopurulent discharge
- · Redness of the eyes
- Photophobia (light sensitivity)
- Burning, stinging or itching or other pain associated with the eyes
- Comfort is less compared to when the lens was first placed on eye
- Poor visual acuity (reduced sharpness of vision)
- · Blurred vision, rainbows or halos around objects
- Feeling of dryness

#### WHAT TO DO IF A PROBLEM OCCURS

Patients should be instructed that if any of the above signs or symptoms are noticed, he or she should:

- IMMEDIATELY REMOVE THE LENSES.
- If the discomfort or problem stops, discard the lens and replace it with a new one.
- If the discomfort or problem continues after removing lens(es) or upon insertion of a new lens, IMMEDIATELY remove the lens(es) and contact the eye care professional for identification of the problem and prompt treatment to avoid serious eye damage.
- The patient should be informed that a serious condition such as corneal ulcer, infection, corneal vascularization, or

- iritis may be present, and may progress rapidly. Less serious reactions such as abrasions, infiltrates, and bacterial conjunctivitis must be managed and treated carefully to avoid more serious complications.
- Additionally, contact lens wear may be associated with ocular changes that require consideration of discontinuation or restriction of wear. These include but are not limited to local or generalized comeal edema, epithelial microcysts, epithelial staining, in iltrates, neovascularization, endothelial polymegathism, tarsal papillary changes, conjunctival injection or iritis

#### ADVERSE EFFECT REPORTING

If a patient experiences any serious adverse effects associated with the use of **DAILIES TOTAL1\*** brand (delefilcon A) contact lenses, please notify: Alcon Medical Safety in the USA at 1-800-757-9780.

#### FITTING GUIDE AND PATIENT BOOKLET

Conventional methods of fitting contact lenses apply to delefilcon A contact lenses. For a detailed description of the fitting techniques, refer to the DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal Contact Lenses (delefilcon A) Professional Fitting and Information Guide. Both the professional fitting guide and a patient instruction booklet are available free of charge from:

Alcon Laboratories, Inc. 6201 South Freeway Fort Worth, TX, USA 76134-2099 1-800-241-5999

#### LENS WEAR & REPLACEMENT SCHEDULES

DAILY WEAR (less than 24 hours, while awake):

- To avoid tendency of the daily wear patient to overwear the lenses initially, stress the importance of adhering to a proper, initial wearing schedule. Normal daily wear of lenses assumes a minimum of 6 hours of non lens wear per 24 hour period.
- It may be advisable for patients who have never worn contact lenses previously to be given a wearing schedule that gradually increases wearing time over a few days. This allows more gradual adaptation of the ocular tissues to contact lens wear.
  - The maximum daily wearing time should be determined by the eye care professional based upon the patient's physiological eye condition because individual responses to contact lenses vary. There may be a tendency for patients to overwear the lenses initially. The eye care professional should stress the importance of adhering to the initial maximum wearing schedule. Studies have not been conducted to show that delefilcon A contact lenses are safe to wear during sleep, therefore patients should be advised to remove their lenses while sleeping. Normal daily wear of lenses assumes a minimum of 6 hours of non-lens wear per 24 hour period. Optimum individual wearing schedule will vary.
- Delefilcon A contact lensés are intended to be worn once (daily disposable wear) and then discarded at the end of each wearing period. The patient should be instructed to start the next wearing period with a fresh new lens.

## **EMERGENCY LENS CARE**

Cleaning and disinfection of daily disposable lenses is not recommended. The patient should be reminded to have replacement lenses or back-up spectacles available at all times.

#### CARE FOR A STICKING LENS

If the lens sticks (stops moving) or begins to dry on the eye, instruct the patient to apply several drops of a recommended lubricating solution (used in accordance with package labeling). The patient should wait until the lens begins to move freely on the eye before attempting to remove it. t is important that the patient wash and dry their hands thoroughly before removing the lens. If the lens continues to stick, the patient should IMMEDIATELY consult the eye care professional.

# IN OFFICE USE OF TRIAL LENSES

Eye care professionals should educate contact lens technicians concerning proper use of trial lenses.

Each contact lens is shipped sterile in a blister pack containing phosphate buffered saline solution. Hands should be thoroughly washed and rinsed and dried with a lint-free towel prior to handling a lens. In order to ensure sterility, the blister pack should not be opened until immediately prior to use. For itting and diagnostic purposes lenses should be disposed of after a single use and not be re-used from patient to patient.

#### EMERGENCIES

The patient should be informed that if chemicals of any kind (household products, gardening solutions, laboratory chemicals, etc.) are splashed into the eyes, the patient should:

etc) are splashed into the eyes, the patient should:

Flush eyes immediately with tap water or fresh saline
solution and immediately contact the eye care professional
or visit a hospital emergency room without delay.

#### HOW SUPPLIED

Each lens is packaged in a foil-sealed plastic container containing phosphate buffered saline solution with approximately 0.3% of polymeric wetting agents consisting of copolymers of polyamidoamine and poly(acrylamide-acrylic) acid and is steam sterilized THERLY. The package is marked with the base curve, diameter, dioptric power and ADD power (multifocal lenses), manufacturing lot number and expiration date.

The following may appear on the labels or cartons:

| Symbols/Signs/<br>Abbreviations | Description |
|---|---|
| 1 Zente | CAUTION: Federal law (United States) restricts this device to sale by or or<br>the order of a licensed eye care professional. |
| SMESSELE L | Steam sterilized |
| EXP | Use by date (Expiry date) |
| LOT | Batch code |
| -2 | Do not reuse |
| 98 | Do not use if blister package is damaged |
| en | Example of two letter language code (English) |
| DIA | Diameter |
| BC | Base curve |
| PWR | Power |
| D | Diopter (lens power) |
| ADD | Addition power |
| CE | European conformity sign |
| =1 | Caution |
| 13 | See product instructions |
| ION ION | Authorized Representative European Community |
| and I | Manufacturer |
| (%) | Packaging waste license sign |

\* a trademark of Novartis © 2016 Novartis

Manufacturer: Alcon Laboratories, Inc. 6201 South Freeway Fort Worth, TX, USA 76134-2099 www.alcon.com 1-800-241-5999

March 2016 W9 00 0 3 8 2 9 2 - 0 3 1 6

1 Check for actual product availability as additional parameters may be introduced over time

Schein, OD, Glynn RJ, Poggio EC, Seddon JM, Kenyon KR. The Relative Risk of Ulcerative Keratitis Among Users of Daily Wear and Extended Wear Soft Contact lenses. N Eng J Med. 1989; 32321 (12):773-783





Air Optix<sup>®</sup> Multifocal Contact Lenses Plus HydraGlyde<sup>®</sup>

# Alcon

Package Insert for: AIR OPTIX® AQUA, AIR OPTIX® plus HydraGlyde®, AIR OPTIX® for Astigmatism, AIR OPTIX® plus HydraGlyde® for Astigmatism, AIR OPTIX® AQUA Multifocal, AIR OPTIX® plus HydraGlyde® Multifocal, O₂OPTIX® (lotrafilcon B) Soft Contact Lenses

W900148888

IMPORTANT: This package insert is effective as of December 2018 and applicable to the lotrafilcon B contact lenses described below. Please read carefully and keep this information for future use. This package insert is intended for the eye care professional, but should be made available to patients upon request. The eye care professional should provide the patient with appropriate instructions that pertain to the patient's prescribed lenses. Copies of this package insert are available without charge from Alcon by calling Customer Service at 1-800-241-5999 or download from our website at www.alcon.com. Alcon also makes available a Patient Instruction Booklet, which is recommended to be given to patients.



CAUTION: Federal law (United States) restricts this device to sale by or on the order of a licensed eye care profes

# PRODUCT DESCRIPTION

PRODUCT DESCRIPTION
AIR OPTIX® AQUA, AIR OPTIX® plus HydraGlyde®, AIR OPTIX® for Astigmatism,
AIR OPTIX® plus HydraGlyde® for Astigmatism, AIR OPTIX® AQUA Multifocal,
AIR OPTIX® plus HydraGlyde® Multifocal and G<sub>v</sub>OPTIX® (obraficon B) soft contact
lenses are made of a lens material that is approximately 33% water and 67%
lotrafilcon B, a fluoro-silicone containing hydrogel which is surface treated. Lenses
contain the color additive copper phthalocyanine, a light blue handling tint, to make them easier to see when handling

#### · Lens Properties:

- Lens Properties:

  O Refractive Index (hydrated): 1.42

  Light Transmittance: ≥ 96% (@ 610 nm, -1.00D)

  Oxygen Permeabilly (Dk): 110 x 10<sup>-1</sup> (cm²sec) (ml O₂/ml x mm Hg), measured at 35 °C (infinisc Dk-Coulometric method)

  Water Content: 33% by weight in normal saline
- Lens Parameters
- Diameter Range: 13.0 to 15.0 mm
   Power Range: -20.00 to +20.00D
   Base Curve Range: 8.0 to 9.2 mm
- Lens Parameters Available<sup>1</sup>

#### AIR OPTIX® AQUA and O2OPTIX® contact lenses (spherical):

- Chord Diameter: Center Thickness:
- 14.2 mm 0.08 mm @ -3.00D (varies with power)
- Base Curve: 8 6 mm
  - Minus Powers: -0.25 to -8.00D (0.25D steps); -8.50D to -10.00D (0.50D steps)
     Plus Powers: +0.25 to +6.00D (0.25D steps)

- AIR OPTIX® plus HydraGlyde® contact lenses (spherical):
  O Chord Diameter: 14.2 mm
  O Center Thickness: 0.08 mm @ -3.00D (varies with power)
- Base Curve: 8.6 mm
- - Minus Powers: -0.25 to -8.00D in 0.25D steps; -8.50 to -12.00D in 0.50D steps
  - Plus Powers: +0.25 to +6.00D (0.25D steps): +6.50 to +8.00D

#### AIR OPTIX® for Astigmatism2 and AIR OPTIX® plus HydraGlyde® for Astigmatism contact lenses (toric):

- Chord Diameter: 14.5 mm @ -3.00D (varies with power)
  Base Curve: 8.7 mm
- - rs: Minus Powers: plano (0.00D) to -6.00D (0.25D steps); -6.50 to -10.00D (0.50D steps) Plus Powers: +0.25 to +6.00D (0.25D steps) Cylinder: -0.75D, -1.25D, -1.75D, -2.25D Axis: Full circle, 10° steps

# AIR OPTIX® AQUA Multifocal and AIR OPTIX® plus HydraGlyde® Multifocal

- Act let less.

  Chord Diameter: 14.2 mm

  Center Thickness: 0.08 mm @ -3.00D (varies with power)

  Base Curve: 8.6 mm
- - - Minus Powers: plano (0.00D) to -10.00D (0.25D steps) Plus Powers: +0.25 to +6.00D (0.25D steps) Add Powers: LO, MED, HI ADD

When hydrated and placed on the cornea, ALCON lotrafilcon B soft contact lenses act as a refracting medium to focus light rays on the retina.

INDICATIONS (Uses)
AIR OPTIX AQUA®, AIR OPTIX® plus HydraGlyde®, and O<sub>2</sub>OPTIX® (lotrafilcon B) spherical soft contact lenses are indicated for the optical correction of refractive spherical soft contact refuses are multicated for in explorations of optical correction of refractive americopia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes with up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual acuity.

AIR OPTIX® for Astigmatism and AIR OPTIX® plus HydraGlyde® for Astigmatism (lotraficon B) loric soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes with up to 6.00 diopters (0) of astigmatism.

AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde® Multifocal (lotraflicon B) soft contact lenses are indicated for the optical correction of presbyopia, with or without refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes who may require a reading addition of +3.00 diopters (D) or less and who may have up to approximately 1.50 d opters (D) of astigmatism that does not interfere with visual acuity.

The lenses may be prescribed for daily wear or extended wear for up to 6 nights of continuous wear with removal for disposal, or cleaning and disinfection (chemical, not heat) prior to reinsertion, as recommended by the eye care professional.

- CONTRAINDICATIONS (Reasons Not to Use)
  DO NOT use lotrafilcon B contact lerses when any of the following exists:

  Inflammation or infection of the anterior chamber of the eye
  Any active disease, injury or abnormality affecting the comea, conjunctiva, or

- Any active usease, injury or anothinally alrectaing the conteat, conjunctival, of eyelids that may be exaggerated by contact lens wear Microbial infection of the eye inadequate tear film (dry eye) that interferes with contact lens wear Corneal hypoesthesia (reduced corneal sensitivity). Use of any medication that is contraindicated or interferes with contact lens wear, including eye medications. Any systemic disease that may be exacerbated by or interferes with safe contact lens wear for the executions and/or executions.
- lens wear, handling, and/or care
  Allergic reactions or ocular irritation of the ocular surfaces or adnexa that may be
  caused by or exaggerated by the wearing of contact lenses
  Allergy to an ingredient in a solution which must be used to care for the contact
- lenses
  Patient history of recurring eye or eyelid infections, adverse effects associated with contact lens wear, intolerance or abnormal ocular response to contact lens

Wear
 If eyes become red or irritated

Advise patients of the following warnings pertaining to contact lens wear.

- Serious eye injury, scarring of the comea, and loss of vision may result from problems associated with wearing contact lenses and using contact lens care products. To reduce these risks, emphasize to the patient the need for strict compliance with the lens care regimen including hand washing, proper lens disinfection, deaning of the lens case, wearing restrictions, wearing schedules, and follow-up visit schedules.
- Eye problems, including comeal ulcers, can develop rapidly and lead to loss of vision. Instruct patients at the dispensing visit and subsequent visits to immediately remove their lenses and promptly contact their eye care professional if they should experience eye discomfort, foreign body sensation, excessive tearing, vision changes, redness of the eye or other problems with their eyes.
- Non-compliance with the manufacturer's labeled lens care instructions may put the patient at significant risk of developing a serious eye infection.
- Non-sterile liquids (i.e., tap water, distilled water, homemade saline solution, or saliva) should NOT be used as a substitute for any component in the lens care process. The use of tap and distilled water has been associated with Acarthamoeba keraitits, a comeal infection that is resistant to treatment and
- Smoking increases the risk of comeal ulcers for contact lens users, especially when lenses are worn overnight or while sleeping.
- The risk of microbial keratitis (a serious eye infection) has been shown to be greater among users of extended wear lenses than among users of daily wear lenses. The risk increases with the number of consecutive days that the lenses are worn between removals even with the first overnight use

To prevent damage to the eyes or to the contact lenses, the following precautions should be taken:

Special Precautions for the Eye Care Professional:

Due to the small number of patients enrolled in the clinical investigation of lenses, all refractive powers, design configurations, or lens parameters available in the lens material are not evaluated in significant numbers. Consequently when selecting an appropriate lens design and parameters, the eye care professional should consider all characteristics of the lens that can affect lens performance and coular health, including overpon promobility, contrait and engineer and cotic representations. including oxygen permeability, central and peripheral thickness and optic zone

The potential impact of these factors on the patient's ocular health should be carefully weighed against the patient's need for refractive correction; therefore the continuing ocular health of the patient and lens performance on the eye should be carefully evaluated on initial dispensing and monitored on an ongoing basis by the prescribing eye care professional.

- The following patients may not be suitable candidates and/or may experience a higher rate of adverse effects associated with contact lens wear.

  Patients with a history of non-compliance with contact lens care and disinfection regimen, wearing restrictions, wearing schedule or follow-up
- visit schedule.

  Patients who are unable or unwilling to understand or comply with any directions, warnings, precautions, or restrictions. Contributing factors may include but are not limited to age, infirmity, other mental or physical conditions, and adverse working or living conditions.

  Fluorescein, a yellow dye, should not be used while the lenses are on the patient's eyes. The lenses absorb this dye and become discolored. Whenever fluorescein is used, the eyes should be flushed thoroughly with sterile saline solution that is repromended for in eyes prior to insection lenses. Aunid
- solution that is recommended for in eye use prior to inserting lenses. Avoid dispensing saline from an aerosol can directly into the eye. Before leaving the eye care professional's office, patients should be able to promptly remove their lenses or should have someone else available who can remove their lenses for them.

- remove their lenses for them.

  Eye care professionals should instruct the patient to remove the lenses immediately if the eye becomes red or imitated.

  Routine eye examinations are necessary to help assure the continued health of the patients eyes. Eye care professionals should make arrangements with the patient for appropriate follow-up visits.

  Diabetics may have reduced comeal sensitivity and thus are more prone to corneal injury and do not heal as quickly or competely as non-diabetics.

  Visual changes or changes in lens tolerance may occur during pregnancy or use of oral contraceptives. Caution patients accordingly.

  Patients who wear contact lenses to correct presbyopia may not achieve the best correct visual aculy for either far or near vision. Vision requirements vary with the individual and should be considered when selecting the most appropriate type of lens for each patient.

Eye Care Professionals should carefully instruct patients about the following care regimen and safety precautions:

# Handling Precautions:

type of lens for each patient

- andling Precautions:

  Be sure that before leaving the eye care professional's office the patient is able to promptly remove lenses or have someone else available to remove them. Good hygiene habits help promote safe and comfortable lens wear. Always wash and rinse hands before handling lenses.

  REMOVE A LENS IMMEDIATELY if an eye becomes red or irritated.

  Carefully follow the handling, insertion, removal, deaning, disinfecting, storing and wearing instructions in the Patient Instruction Booklet for the lotrafilcon B soft contact lenses prescribed.
- Soft contact lenses prescribed.

  Always handle lenses carefully. If a lens is dropped small particles or fibers may adhere to the lens surface which can irritate the eye. Lenses should be cleaned and disinfected prior to insertion or replaced with a sterile, fresh new lens.
- Never use tweezers or other sharp objects such as fingernaits to remove lenses from the lens container. Pour the lens onto the hand.

#### Lens Wearing Precautions:

- Patients should never exceed the prescribed wearing schedule, regardless of how comfortable the lenses feel. Doing so may increase the risk of adverse
- effects.

  The lens should move freely on the eye at all times. If the lens sticks (stops moving) on the eye, follow the recommended directions in the CARE FOR A STICKING LENS section. If non-movement of the lens continues, the patient should be instructed to consult their eye care professional immediately.

  The eye care professional should be consulted about wearing lenses during

water sports and water related activities. Exposure to water while wearing contact lenses in activities such as swimming, water skiing, and hot tubs may increase the risk of ocular infection, including but not limited to Acanthamoeba

- Eye irritation, infection, or lens damage may result if cosmetics, lotion, soap, cream, hairspray, deodorant, aerosol products or foreign particles come in contact with lens
- Never allow contact lenses to come into contact with non-sterile liquids (including tap water and saliva) as microbial contamination can occur, which may
- Inducing alp water and saliva) as incloud contamination can occur, which me lead to permanent eye damage.

  Do not share lenses with anyone as this may spread micro-organisms which could result in serious eye health problems.

  Environmental fumes, smoke, and vapors should be avoided in order to reduce the chance of lens contamination or physical trauma to the comea.
- Lenses should be disposed of and replaced according to the eye care
- professional's recommendations.

  Note the correct lens power for each eye to prevent getting them mixed up.

  Always keep a supply of replacement lenses on hand or have back-up spectacles
- Do not use lenses beyond the expiration date.

#### Solution Precautions:

- Figure 1 Precadulors.

  Eye injury due to irritation or infection may result from lens contamination. To reduce the risk of contamination, review the appropriate manufacturer's labeled lens care instructions with the patient (see the LENS CARE DIRECTIONS section). Only use fresh, unexpired lens care solutions recommended for use with soft contact lenses and follow directions in the product package inserts. If a lens is exposed to air while of the eye it may become dry, brittle, and permanently damaged. If this should occur, the lens should be discarded and englaced with a new one to awaid nossible intribation or injury to the exe. Always permanently damageur. In this should occur, the lens solicin de strated and replaced with a new one to avoid possible imitation or injury to the eye. Always keep the lenses completely immersed in the recommended storage solution when lenses are not being worn.

  Do not use thermal (heat) disinfection and do not heat lens care products.

  Saliva or anything other than the recommended solution for lubricating or wetting lenses should not be used with the lenses.

Contact lens cases can be a source of bacterial growth and require proper use, cleaning and replacement at regular intervals as recommended by the lens case manufacturer or eye care professional.

# Other Topics to Discuss with Patients

- ther Topics to Discuss with Patients

  Periodic eye examinations are extremely important for contact lens wearers.

  Schedule and conduct appropriate follow-up examinations to determine ocular response. Alcon recommends that patients see their eye care professional at least once each year or as recommended by the eye care professional. Certain medications may cause dyness of the eye, increased lens awareness, lens intolerance, blurred vision, or visional changes. These include, but are not limited to antihistamines, decongestants, duretics, muscle relaxants, tranquilizers and those for motion sickness. Caution patients using medications accordingly and prescribe proper remedial measures.

  Visual changes or changes in lens tolerance may occur during pregnancy or use of oral contraceptives. Caution patients accordingly

- Who Should Know That the Patient is Wearing Contact Lenses
   Patients should inform their health care professional that they are wearing
- Patient should inform their readir care professional trial trieg are wearing contact lenses.

  Patient should inform their employers that they are wearing contact lenses. Some jobs may require the use of eye protection equipment or may require that contact. enses not be worn

It is strongly recommended that patients be provided with a copy of the AIR OPTIX® AQUA, AIR OPTIX® plus HydraGlyde®, AIR OPTIX® for Astigmatism, AIR OPTIX® plus HydraGlyde® for Astigmatism, AIR OPTIX® AQUA Multiflocal and AIR OPTIX® plus HydraGlyde® full tiflocal soft contact lens Patient Instruction Booklet available from Alcon and understand its contents prior to dispensing the

# ADVERSE FEFFCTS (Possible Problems)

ADVENCE EFFECTS (POSSIDE PRODURINS)
Patients should be instructed to check eyes regularly to make sure they look well, feel comfortable and vision is clear. Potentially serious complications are usually accompanied by one or more of the following signs and symptoms:

Moderate to severe eye pain not relieved by removing the lens
Feeling of something in the eye (foreign body sensation)

Excessive watering or other eye secretions including mucopurulent discharge

- Excessive watering or order eye secretions including mucopuratem. Redness of the eyes Sensitivity to light (photophobia) Burning, stinging, or itching or other pain associated with the eyes Comfort is less compared to when the lens was first placed on eye Poor visual acuity (reduced sharpness of vision) Blurred vision, rainbows or halos around objects Section of drivings. Feeling of dryness
  These symptoms, if ignored, may lead to more serious complications.

WHAT TO DO IF A PROBLEM OCCURS Patients should be instructed that if any of the above signs or symptoms occur, he or she should:

- If the discomfort or problem stops, then look closely at the lenses.

  If the discomfort or problem stops, then look closely at the lenses.

  If a lens is in any way damaged, DO NOT put it back on the eye. Replace with a new lens and consult the eye care professional.

  If a lens has dirt, an eyelash, or foreign body on it, or the problem stops and the lens appears undamaged, thoroughly clean, rinse and disinfect the lens before reinsertion.
- If the above symptoms continue after removal or upon reinsertion of the lens, remove the lens immediately, then promptly contact an eye care professional The patient should be informed that a serious condition such as comeal ulcer (ulcerative keratitis), infection, comeal vascularization or initis may be present. These conditions may progress rapidly and may lead to permanent loss of vision Less serious reactions such as abrasions, infiltrates and bacterial conjunctivitis.
- Less serious reactions such as advastors, initiates and bacterial compilitations, must be managed and treated properly to avoid more senious complications. Additionally contact lens wear may be associated with ocular changes that require consideration of discontinuation or restriction of wear. These include, but are not limited to, local or generalized comeal edema, epithelial microcysts, epithelial staining, infiltrates, neovascularization, endothelial polymegethism,
- constant saming, immunes, incommune and incommune payment at rataral papilitary changes, conjunctival injection or iritis.

  Occasional dyness may be relieved by blinking fully several times or by the use of contact lens rewetting drops that are approved for use with soft contact lenses. If dyness persists, consult your eye care professional.
- If a lens sticks (stops moving), apply several drops of a contact lens rewetting

solution and wait until the lens begins to move freely on the eye. If this problem persists, consult your eye care professional. If a lens decenters on the eye, it may be possible to recenter it by:

- Closing your eyelids and gently massaging the lens into place, or Looking in the direction of the lens and blinking gently, or Gently pushing the off-centered lens onto the comea with light finger
- pressure on the edge of the upper or lower eyelid.
  If a lens tears in your eye, remove the pieces carefully by pinching them as you would for normal lens removal. If the lens pieces do not seem to remove easily, do not pinch the eye tissue. Rinse with saline. If this does not help, contact the eve care professional for assistance.

#### **EMERGENCIES**

The patient should be informed that if chemicals of any kind (household products,

- gardening solutions, laboratory chemicals, etc.) are splashed into the eyes:

   Flush eyes immediately with fresh saline solution or tap water.

  Remove and discard lenses and immediately contact the eye care professional or visit a hospital emergency room without delay.

#### ADVERSE EFFECTS REPORTING

If a patient experiences any serious adverse effects associated with the use of lotrafilcon B contact lenses, please not fy: Alcon Medical Safety, in the USA at

#### FITTING GUIDE AND PATIENT BOOKLET

FITTING GUIDE AND PATIENT BOUNCE!

Conventional methods of fitting contact lenses apply to lotrafilcon B contact lenses.

For a detailed descript on of the fitting techniques, refer to the
AIR OPTIX\* AQUA, AIR OPTIX\* pius HydraGlyde\*, AIR OPTIX\* for Astigmatism,
AIR OPTIX\* Pus HydraGlyde\* for Astigmatism, AIR OPTIX\* AQUA Multifocal and
AIR OPTIX\* pius HydraGlyde\* Multifocal (lotraficon B) contact lens Professional

Fitting and Information Guide. Both the fitting guide and a Patient Instruction Booklet

rea evailable free of charge from: are available free of charge from:

Alcon Laboratories, Inc.

6201 South Freeway Fort Worth, TX 76134-2099 USA

or by calling Alcon Customer Service in the USA at 1-800-241-5999.

#### LENS WEAR AND REPLACEMENT SCHEDULES

LEMS WEAR AND REPLACEMENT SCHEDULES.

The wearing and replacement schedule should be determined by an eye care professional based on the patients individual needs and physiological conditions. The eye care professional may recommend daily wear only or extended wear periods up to 6 nights. Not everyone can reach the maximum wear time of 6 continuous

- Daily Wear (less than 24 hours, while awake)

  To avoid tendency of the daily wear patient to over wear the lenses initially, stress the importance of adhering to a proper, initial wearing schedule. Normal daily wear of lenses assumes a minimum of 6 hours of non-lens wear per 24 hour period.

  It may be advisable for patients who have never wom contact lenses previously to be given a wearing schedule that gradually increases wearing time over a wed with the strength of the coular tissues to contact lens wear.

#### Extended Wear (greater than 24 hours, including while asleep):

- The eye care professional should establish an extended wear period up to 6 continuous nights that is appropriate for each patient. Once the lens is removed, the patient's eyes should have a rest period with no lens wear of overnight or longer, as recommended by the eye care professional. It is suggested that new contact lens wearers first be evaluated on a daily
- It is suggested unliew contact term weards in its be evaluated in a dia-wear schedule. If the patient is judged to be an acceptable extended wer candidate, the eye care professional may determine an extended wear schedule based upon the response of the patient.
- See WARNINGS section for information about the relationship between wearing schedule and comeal complications.

#### Lens Replacement

The replacement schedule is determined by the eye care professional based on the patients individual needs and physiological conditions. Lenses should be discarded and replaced with a new pair each month, or more often, if recommended by the eye care professional.

## LENS HANDLING INSTRUCTIONS

- Always wash and rinse hands thoroughly and dry completely with a clean, lint-free towel before handling contact lenses. Do not use if hister package is damaged or not sealed completely. This may result in product contamination which can lead to a serious eye infection.

- Shake the bilster pack (containing a fresh new lens) gently prior to opening. Remove the lens from the blister pack (or lens storage case for previously worn lenses) by carefully pouring it onto the palm of the hand. Ensure the lens is right side out and that you have the correct lens for each eye. Inspect the lenses prior to insertion.
- Do not insert damaged or unclean lenses.

#### Lens Insertion Instructions

- Wash and rinse hands thoroughly and dry completely with a clean, lint-free towel. Place a lens on the tip of your clean and dry right or left index finger. Place the middle finger of the same hand close to lower eyelashes and pull down the lower
- Use the fingers of the other hand to lift the upper eyelid.
  Place the lens directly on the eye (comea) and gently roll finger away from the
- Look down and slowly release the lower lid.
- Look straight ahead and slowly release the upper lid. Blink gently.

#### Lens Removal Instructions

- Wash and rinse hands thoroughly, and dry completely with a clean, lint-free
- Blink fully several times.
- While looking up, use the tip of the finger to slide the lens down onto the white part of the eye.

  Remove the lens by pinching gently between thumb and forefinger. Do not pinch
- the eye tissue.
  If the lens is difficult to remove, instill a lubricating and rewetting drop and try
- again after several minutes.

  Never use tweezers, suction cups, sharp objects or finger nails to remove lenses

from the lens container or your eyes.

## WATER ACTIVITIES

Do not expose contact lenses to water while wearing them. Warning:

Water can harbor microorganisms that can lead to severe infection, vision loss or blindness. If lenses have been submersed in water when showering or swimming, discard them and replace with a new pair. Ask the eye care professional for recommendations about wearing lenses during any activity

#### LENS CARE DIRECTIONS

Patients must adhere to a recommended lens care regimen. Lenses must be cleaned, mised and disinfected after removal and prior to reinsertion on the eye according to the instructions in the package inserts provided with the lens care products recommended by the eye care professional. Failure to follow the complete regimen in accordance with the manufacturer's instructions in the package inserts may contribute to problems (see the ADVERSE EFFECTS section) and/or result in the development of serious ocular complications and discussed in the WARNINGS

sposable Wear: No lens care is indicated, as lenses are discarded upon removal from the eye. Lenses should only be cleaned, rinsed and disinfected on an emergency basis when replacement lenses are not available.

#### Replacement Wear:

When removed between replacement periods lenses must be cleaned and disinfected prior to reinsertion or be discarded and replaced with a fresh lens.

#### Basic Instructions for Lens Cleaning and Disinfection:

When lenses are dispensed, the eye care professional should recommend an appropriate system of lens care and provide the patient with instructions according to the package labeling.

The eye care professional should review the following instructions with the patient:

Each time lenses are removed from the eye they must be properly cleaned, rinsed, and disinfected before reuse. If removed while the patient is away from lens care products, the lenses may not be reinserted, but should be stored until they can be cleaned, rinsed and disinfected.

Cleaning is necessary to remove mucus, film and contamination from the lens surface. Rinsing removes all traces of the cleaner and loosened debris. Disinfecting is necessary to destroy remaining microorganisms. Lenses must be deaned, rinsed, disinfected and stored in accordance with the

- package labeling of the lens care products recommended by the eye care professional. Typical instructions for lens care products include the steps presented below. IMPORTANT: Hydrogen Peroxide disinfecting solutions, such as CLEAR CARE® PLUS Cleaning & Disinfecting Solution, are not multi-purpose solutions. For hydrogen peroxide disinfecting solutions follow the manufacturer's
- Solutions. For hydrogen percondents interesting solutions follow the maintacturins instructions.

  Soaking and Storing Your Lenses:

  O Use only fresh contact lens care solution each time you soak (store) your lenses

Warning:

Do not reuse or "top off" old solution left in your lens case since solution

The land disinfection and could lead to super infection. reuse reduces effective lens disinfection and could lead to severe infection, vision loss or blindness. To "top-off" means to add fresh solution to solution that has been stitting in your lens case.

- Rub and Rinse Time:

- Some lens care products require a rub and rinse step. If so, follow the lens care manufacturer's instructions for solution quantity and rub and rinse time to reduce the risk of serious eye infections.

  The amount of time you can store lenses before cleaning, rinsing, and
- disinfection steps need to be repeated will vary depending on the lens care product used
- va*ming:* Rub and rinse lenses for the recommended amount of time to help prevent serious eve infections.
- Never use water, saline solution, or rewetting drops to disinfect your lenses. These solutions will not disinfect your lenses. Not using the recommended disinfecting solution can lead to severe infection, vision loss or blindness.
- Discard Date for Lens Cleaning and Disinfecting Solutions
   After opening, discard any remaining solution after the period recommended by the lens care manufacturer. If using the lens care products listed below, discard remaining solution as follows:

   CLEAR CARE® PLUS Cleaning & Disinfecting Solution 3 months after

  - opening.
     OPTI-FREE® PureMoist® Multi-Purpose Disinfecting Solution 6 months after opening.

Using your lens care solution beyond the discard date could result in contamination of the solution and can lead to severe infection, vision loss or

- The above instructions are typical for a lens cleaning product, however you must always consult the instructions for the specific lens care product used.

  Alcon recommends a chemical (not heat) method of disinfection such as CLEAR CARE® PLUS Cleaning & Disinfecting Solution or OPTI-FREE® PureMoist® Multi-purpose Disinfecting Solution.

  Use of an enzymatic cleaner is optional and may be recommended by the eye care professional if warranted.
- Lens compatibility with an abrasive type deaner such as OPTI-CLEAN® II Daily Cleaner has not been tested and is not recommended.
- Heat disinfection has not been tested and is not recommended.

#### Basic Instructions for the Lens Case

Basic instructions for the Lefts case

Contact lens care solutions and contact lens cases vary and have different purposes
and instructions for use. Some cases are intended exclusively for storing contact
lenses (sometimes referred to as a lens flat pack or lens storage case), while others
are specially designed to contain a neutralizing disc for use with hydrogen peroade
deaning and disinfecting systems. If not being worn on a daily disposable basis,
lenses that have been cleaned and disinfected can be stored in the unopened case
for a period of time that varies depending on the contact lens solution and lens case
seed Always follow the instructions provided by the manifecturer for the lane care. used. Always follow the instructions provided by the manufacturer for the lens care products used.

- The eye care professional should instruct the patient on how to use the recommended lens care solution(s) and lens case.
- recommended lens care solution(s) and lens case.

  Contact lens cases can be a source of bacterial growth and require proper deaning, dyring and replacement to avoid contamination or damage to lenses:

  Clean contact lens cases with an appropriate contact lens solution and dry according to lens case instructions. Drying instructions, such as air-drying or wiping with lint-free towel, may vary depending on the lens case used.

  Replace contact lens cases at least once every 3 months, or as recommended by the lens case manufacturer.

  Replace specially designed lens cases containing a neutralizing disc according to manufacture directions.
- according to manufacturer directions, or sooner if cleaned and disinfected es cause burning and stinging.

Do not store your lenses or rinse your lens case with water or any non-sterile solution. Only use fresh disinfecting solution in order to avoid contamination of your lenses or lens case. Use of non-sterile solution can lead to severe infection, vision loss or blindness.

# To help avoid serious eye injury from contamination, the eye care professional should review the following instructions with the patient: Always wash, rinse and dry hands before handling the lenses: Use only fresh sterile solutions recommended for use with soft (hydrophilic)

- use drily fresh stellie solutions recommended to use with soft (rydrophilic) contact lenses. When opened, sterile non-preserved solutions must be discarded after the time specified in the label directions. Do not use saliva, lap water, homemade saline solution, distilled water, or anything other than a recommended sterile solution indicated for the care of soft lenses.

- Do not reuse solutions.
   Use only fresh solutions for each lens care step. Never add fresh solution to old solution in the lens case.
   Follow the manufacturer's instructions for care of the lens case.

- Replace the lens case at regular intervals to help prevent case contamination by microorganisms that can cause eye infection.
   Never use a hard (rigid) lens solution unless it is also indicated for use with
- soft contact lenses. Comeal injury may result if hard (rigid) lens solutions not indicated for use with soft lenses are used in the soft lens care regimen.

  Always keep the lenses completely immersed in the recommended storage
- solution when the lenses are not being worn to avoid lens dehydration.

  Unless specifically indicated in the labeling, do not alternate, change, or mix lens care systems or solutions for any one pair of lenses. If n doubt as to solution suitability, consult the eye care professional.

#### CARE FOR A STICKING LENS

CARE-PORA STICKING LENS

If the lens sticks (stops mowing) or begins to dry on the eye, instruct the patient to apply several drops of a recommended lubricating solution (used in accordance with package labeling). The patient should wait until the lens begins to move freely on the eye before attempting to remove: it if the lens continues to stick, the patient should IMMEDIATELY consult the eye care professional.

#### IN OFFICE USE OF TRIAL LENSES

Eye care professionals should educate contact lens technicians concerning proper

Life date photosomation among administration containing account and use of third lienses. Each contact lens is shipped sterile in a bitster pack containing phosphale buffered saline solution with or without additives. Hands should be thoroughly washed, rinsed and dried with a lint-free towel prior to handling a lens. In order to ensure sterility, the blister pack should not be opened until immediately prior to use. For fitting and diagnostic purposes, the lenses should be disposed of after a single use and not be re-used from patient to patient.

#### DISPOSAL AND RECYCLING

Dispose of contact lenses and the blister pack lidding in the waste bin, not down the sink or toilet. The carton packaging and the polypropylene (PP) plastic shell of the blister pack should be placed in the waste bin or recycled according to local waste management guidance

#### HOW SUPPLIED

Each lens is provided in a foil-sealed plastic container containing buffered saline solution and is steam sterilized .The packaging saline may contain additives, as

- AIR OPTIX® for Astigmatism and O2OPTIX® contact lenses: Phosphate Buffered
- AIR OPTIX® AQUA and AIR OPTIX® AQUA Multifocal contact lenses: PBS with
- AIR OP IX\* AQUA aim ain United Stock Market Market Stock Market

The blister package is marked with the base curve, diameter, dioptric power, cylinder and axis (where applicable), ADD power (where applicable), manufacturing lot number, and expiration date.

The package labeling may also contain a product code, as follows: LFB110 [spherical lotraficon B in phosphate buffered saline (FBS)]; LFB110c [spherical lotraficon B in PBS + Copolymer 845 (e.g., VP/DMAEMA)]; LFB110e [spherical lotraficon B in PBS + Copolymer (e.g., VP/DMAEMA) +

LEBTIOE (Spriencal localizon B in PSS + Copolymer (e.g., VP/DMAEMA) + HydraClyde;
LEBTIOT (toric lotraficon B in PBS);
LEBTIOT (toric lotraficon B in PBS + Copolymer (e.g., VP/DMAEMA));
LEBTIOTE (toric lotraficon B in PBS + Copolymer (e.g., VP/DMAEMA) + HydraClyde);
LEBTIOMFe (multifocal lotraficon B in PBS + Copolymer (e.g., VP/DMAEMA) + HydraClyde);
HydraClyde);

Lenses are supplied in cartons containing up to 12 individually sealed contact

The following may appear on the labels or cartons

| Symbol/<br>Abbreviation | Definition |
|---|---|
| <b>⊕</b> =#/ | CAUTION: Federal law (United States) restricts this device to sale by<br>or on the order of a licensed eye care professional. |
| STERILE | Sterilized using steam |
| 2 | Use-by date |
| EXP | Expirat on date |
| LOY | Batch code |
| θЛ | Two letter code for the language (Example shown: Engish) |
| 杨 | Do not use if blister package is damaged |
| C€ | European conformity mark |
| (3) | Consult instructions for use |
| A | Caution |
| 10 50 | Authorized Represen ative in the European Community |
| | Manufacturer |
| c4 | Date of manufacture |
| 6 | Packaging waste license sign |
| MI | Medical device |
| DIA | Diameter |
| BC | Base curve |
| PWR | Power |
| CYL | Cylinder power |
| D | Diopter (lens power) |
| ADD | Addition power |
| MAX ADD | Maximum effective addition power |
| LO | Low |
| MED | Medium |
| Hi | High |
| L. | Left |
| R | Right |
| VP/DMAEMA | Vinylpyrrolidone/Dimethylaminoethylmethacrylate |

Alcon

Alcon Laboratories Inc. 6201 South Freeway Fort Worth, TX 76134-2099 USA U.S. Pat.: www.alconpatents.com Date of preparation: December 2018 W900148888-1218

<sup>1</sup>Check for actual product availability, which may change over time. Manufacture of O₂OPTIX® lenses discontinued 2014

"May also be labeled as CoPTIX' for Astigmatism
"Cutter GR, Chalmers RL, Roseman M. The Clinical Presentation, Prevalence, and
Risk Factors of Focal Comeal Infiltrates in Soft Contact Lens Wearers. The CLAO Journal: Jan 1996; 22 (1):30-37.

Schein OD, Glynn RJ, Poggio EC, Seddon JM, Kenyon KR. The Relative Risk of Ulcerative Keratitis Among Users of Daily-Wear and Extended-Wear Soft Contact Lenses. N Eng J Med. 1969; 321(12):773-83.

CR-6344, vl.0 LIVC 

# APPENDIX D: BINOCULAR OVER REFRACTION

# Binocular Over-refraction Technique

- 1. Place trial frame on subject
- 2. Add +1.00 D sphere to OS
- 3. Add + 0.50DS OD and check VA
  - if VA remained unchanged or improved, repeat step 3
  - if VA decreased, add minus until best VA first achieved \*note: add minus for 0.5 seconds to avoid reflex accommodation.
- 4. Record VA
- 5. Change +1.00 D sphere to OD
- 6. Repeat steps 3 and 4

# APPENDIX E: PRESBYOPIC SYMPTOMS QUESTIONNAIRE

# **Presbyopic Symptoms Questionnaire**

- 1. Do you notice that you often have to hold things farther away so that you can read them?
- 2. Do you notice that you often have difficulty focusing on near objects (i.e., experiencing blurry vision when looking at things close-up)?
- 3. Do you often have headaches or eyestrain, or feel fatigued, when reading or conducting other near activities?
- 4. Do you often have difficulty reading small or fine prints, such as phone books, medicine bottles or package labels, etc.?
- 5. Do you often have difficulty reading under dim or low light?

# OCULAR DOMNANCE TEST

# +1.00 D LENS TEST

- Step 1 Place the subjects best sphero-cylindrical distance refraction in a trial frame.
- Step 2 Have the subject view a BVA line of letters.
- Step 3 With both eyes open alternate a +1.00 D trial lens between the right and left eye and ask the subject to indicate over which eye does the lens cause the line of letters to appear more blurred. The eye that the greatest blur is reported is the distance dominant eye. If the subject indicates that the amount of blur is about the same between the two eyes then record as neither eye dominant.

# SIGHTING OCULAR DOMINANCE

- Step 1 Ask the subject to extend both arms out and use his/her hands to form a triangle. The subject will be asked to keep both eyes open and look through the triangle at a small object on the wall (e.g., a light switch or doorknob).
- Step 2 Occlude the subject's left eye, then right eye. While alternating the occluder from the subject's eyes, ask the subject when they see the object.

If the subject sees the object when the left eye is covered, the subject is *right eye* dominant.

If the subject sees the object when the right eye is covered, the subject is *left eye* dominant.

If the subject sees the object with both eyes, the opening between the hands may be too large. Therefore, ask the subject to make a smaller opening and repeat the procedure.

# APPENDIX G: ALCON DAILIES TOTAL 1 MULTIFOCAL CONTACT LENS FITTING GUIDE

# Professional Fitting and Information Guide

DAILIES TOTAL1\*
and
DAILIES TOTAL1\* Multifocal
(delefilcon A) Soft Contact Lenses
For Single-Use, Daily Disposable Wear

Water Gradient One-Day Contact Lenses



CAUTION: Federal law (United States) restricts this device to sale by or on the order of a licensed eye care professional.



This page

left blank

# Table of Contents

| Introduction | 5 |
|-----------------------------------------------------------|----|
| Product Description | 5 |
| Lens Properties | |
| Available Lens Parameters | 6 |
| Actions | |
| Indications (Uses) | 6 |
| Contraindications, Warnings, Precautions, Adverse Effects | 7 |
| Adverse Effect Reporting | 7 |
| Fitting Guidelines (Spherical Lenses) | |
| Patient Selection | 8 |
| Pre-fitting Examination | 8 |
| Trial Lens Evaluation | 8 |
| Lens Base Curve Selection | 8 |
| Initial Lens Power Selection | 8 |
| Lens Fit Assessment | 9 |
| Final Lens Power Determination | 10 |
| Fitting Guidelines (Multifocal Lenses) | 11 |
| Pre-Fitting Examination | 11 |
| Patient Selection | 11 |
| Initial Lens Selection | 13 |
| Initial Lens Fitting Evaluation | 14 |
| Initial Lens Visual Evaluation | |
| Fitting Procedures | 16 |
| Fitting Guidelines (Monovision) | 18 |
| Patient Selection | 18 |
| Eye Selection | |
| Special Fitting Considerations | |
| Near Add Determination | |
| Trial Lens Fitting | 20 |
| Adaptation | |
| Other Suggestions | |
| Dispensing Visit | |
| Follow-Up Examinations | |
| Follow-up Examination Procedures | |
| Lens Handling Hints | |
| Lens Insertion | |
| Lens Removal | |
| Care for a Sticking Lens | |
| In Office Care of Trial Lenses | |
| Additional Information | |
| Vertex Distance Conversion Chart | |
| Product Pockago Incort | 20 |

This page

left blank

#### Introduction

Thank you for prescribing DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) daily disposable soft contact lenses. The benefits of a high oxygen transmissible and wettable lens material with a state of the art manufacturing process are combined to make DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) lenses. This guide contains important information regarding fitting procedures and aftercare of the DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) contact lens patient.

## **Daily Disposability:**

By eliminating the need for lens care, daily disposable lenses offer your patients a major advancement in wearing convenience. The next time you prescribe lenses consider the health and comfort benefits of beginning each wearing period with a new pair of fresh, sterile lenses that are worn once and then discarded.

## LightStream\* Lens Technology:

DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses are made from a proprietary silicone hydrogel material with a water content of approximately 33% water. The use of process automation, precision glass and quartz molds and photolithographic edge forming help ensure every lens has the same crisp optics, smooth surface finish and consistent edge quality from lens to lens. Delefilcon A contact lenses are produced under strictly controlled process conditions and inspected to exacting quality tolerances. As a result, you can be confident your patients will experience consistent vision, comfort, and ease of handling every day.

#### PRODUCT DESCRIPTION

DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal soft contact lenses are made a silicone containing hydrogel that is approximately 33% water and 67% delefilcon A polymer with added phosphatidylcholine. The core lens material containing 33% water transitions through a water gradient to a hydrogel surface layer that exceeds 80% water. This structure enables a silicone hydrogel lens with a water gradient that has:

- Over 80% water at the surface of the lens to mimic the water content of the cornea
- High level of oxygen transmissibility through the lens.
- · Excellent overall comfort.

The lenses contain and release phosphatidylcholine (DMPC), a phospholipid found naturally in the tears. In addition, lenses contain the color additive copper phthalocyanine, a light blue tint which makes them easier to see when handling. The lenses are packaged in strips of 5 individual blisters containing buffered saline with approximately 0.3% of polymeric wetting agents consisting of copolymers of polyamidoamine and poly(acrylamide-acrylic acid).

# **Lens Properties**

Refractive Index (hydrated): 1.42

Light Transmittance: ≥ 93% (@610 nm, -1.00D)
 Oxygen Permeability (Dk): 140 x 10<sup>-11</sup> (cm²/sec)

(ml O<sub>2</sub>/ml x mm Hg), measured at 35°C, (intrinsic Dk - Coulometric method)

Water Content 33% by weight in normal saline

Surface Water Content ≥ 80%

#### Available Lens Parameters<sup>1</sup>

**DAILIES TOTAL1\*** (delefilcon A) Spherical contact lenses

• Chord Diameter Available: 14.1 mm

• Center Thickness: 0.09 mm @ -3.00D (varies with power)

Base Curve: 8.5 mm

Powers Available: -0.50 to -6.00D (0.25D steps); -6.50 to

-12.00D (0.50D steps)

+0.50 to +6.00D (0.25D steps)

## DAILIES TOTAL1\* Multifocal (delefilcon A)

Chord Diameter: 14.1 mm

• Center Thickness: 0.09 mm @ -3.00D (varies with power)

Base Curve: 8.5 mm

• Powers: -0.25 to -10.00D (0.25D steps); plano to

+6.00D (0.25D steps) ADD: LO, MED, HI

<sup>1</sup>Check for actual product availability as additional parameters may be introduced over time.

#### **Actions**

When hydrated and placed on the cornea delefilcon A soft contact lenses act as a refracting medium to focus light rays on the retina.

## **INDICATIONS (USES)**

**DAILIES TOTAL1\*** (delefilcon A) spherical soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes with up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual acuity.

**DAILIES TOTAL1\* Multifocal** (delefilcon A) soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) and/or presbyopia in phakic or aphakic persons with non-diseased eyes who may require a reading addition of +3.00 (D) or less and who may have up to approximately 1.50 diopters (D) of astigmatism that does not interfere with visual acuity.

The lenses are to be prescribed for single use, daily disposable wear. The lenses are not intended to be cleaned or disinfected and should be discarded after a single use.

See WARNINGS for information about the relationship between wearing schedule and corneal complications.

# CONTRAINDICATIONS, WARNINGS, PRECAUTIONS AND ADVERSE EFFECTS

For additional important prescribing and safety information, refer to the Package Insert that is printed in the back of this guide.

#### ADVERSE EFFECT REPORTING

If a patient experiences any serious adverse effects associated with the use of DAILIES TOTAL1\* or DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses, in the USA please **contact Alcon Medical Safety at** 1-800-757-9780.

#### **FITTING GUIDELINES**

Please see the appropriate sections of this booklet that contain guidelines for spherical, multifocal and monovision fitting techniques.

7

# FITTING GUIDELINES (Spherical Lenses)

#### 1. Patient Selection

The patient characteristics necessary to achieve success with DAILIES TOTAL1\* (delefilcon A) spherical lenses are similar to those for other spherical soft contact lenses. A thorough pre-fitting examination should be conducted to ensure the patient is a suitable candidate for soft contact lens wear.

The following procedures should be followed when fitting DAILIES TOTAL1\* (delefilcon A) spherical lenses. For additional tips on fitting the monovision patient refer to the section *Monovision Fitting Guidelines*.

# 2. Pre-fitting Examination

## A pre-fitting examination is necessary to:

- assess the patient's motivation, physical state and willingness to comply with instructions regarding hygiene and wear schedule
- make ocular measurements for initial contact lens parameter selection
- collect baseline clinical information to which post-fitting examination results can be compared

### A pre-fitting examination should include:

- a thorough case history
- · a spherocylindrical refraction
- keratometry
- tear film assessment
- biomicroscopy

#### 3. Trial Lens Evaluation

#### A. Lens Base Curve Selection

A well-fitted lens provides good movement, centration and comfort. An optimal fit can be achieved for the vast majority of patients with the single 8.5 mm base curve.

#### B. Initial Lens Power Selection

The initial power selection should be as close as possible to the patient's prescription after taking into account spherical equivalent and vertex calculations, if necessary.

## **Spherical Equivalent Calculation**

To determine initial lens power, convert the spherocylindrical spectacle Rx to its spherical equivalent as follows:

Spherical Equivalent = Sphere power + 1/2 (Cylinder Power)
Example: Spectacle Rx: -4.50D -1.00 x 180

Spherical equivalent: -4.50D + (-0.50D) = -5.00D

# Vertex Distance Conversion

If the spherical equivalent is greater than  $\pm$  4.00D, a vertex distance correction is necessary (see *Vertex Distance Conversion Chart*) to determine the lens power required at the corneal plane.

Example: Spectacle Rx: -4.50D -1.00 x 180

Spherical equivalent: -4.50D + (-0.50D) = -5.00D Vertex compensation: -4.75 (initial lens power)

#### C. Lens Fit Assessment

Allow the lenses to settle on the eyes for approximately 10 minutes. This allows time for the patient to adapt to the lenses and time for the lens to equilibrate.

Evaluate the fit and movement of the lenses on the eye in primary and up gaze positions. The **Push-up Test**, as described below, is an additional test of the lens evaluation. The following guidelines will be helpful in fit evaluation:

#### Characteristics of a Well-fitted Lens

A well-fitted DAILIES TOTAL1\* (delefilcon A) spherical contact lens satisfies the following criteria:

- 1. Good centration and full corneal coverage in all fields of gaze.
- 2. **Sufficient lens movement to allow tear exchange** under the lens during a blink in primary or upward gaze.
- 3. Satisfactory Push-up Test
  - This test is a reliable indicator of a good fit. With the patient looking straight ahead, place your index finger on the patient's lower lid and nudge the edge of the lens upward while observing lens movement. Then pull the lid back down and observe the return of the lens.
  - A well fitted lens will move freely upward, stopping shortly after passing the limbus and then return freely to its original position.
- Good comfort and stable visual response (with over refraction).

### Characteristics of a Tight (Steep) Lens Fit

A tight or steep lens fit would display some or all of the following characteristics:

- Insufficient or no lens movement during a blink in primary or upward gaze.
- 2. Unsatisfactory Push-up Test
  - A tight fitting lens will resist movement. If successfully nudged upward, the lens may remain decentered or return slowly to its original position.
- 3. Good centration.
- 4. Good comfort.
- Fluctuating vision between blinks.

## Characteristics of a Loose (Flat) Lens Fit

A loose lens fit would display some or all of the following characteristics:

- 1. Reduced comfort, usually accompanied by lower lid sensation.
- Poor centration with limbal exposure on exaggerated eye movement.
- 3. Lens edge standoff.
- Excessive lens movement during the blink in primary or upward gaze.
- 5. Unsatisfactory Push-up Test
  - A loose fitting lens will move easily but may remain decentered or slip under the upper lid.
- 6. Vision may be blurred after the blink.

An inverted lens may mimic the characteristics of a loose lens. If any of

the above signs occur remove the lens and check to make sure it is not inverted.

# **General Fitting Tips**

- Trial fitting of the individual eye is recommended.
- A well fitting lens will show movement of 0.1 to 0.5 mm.

# D. Final Lens Power Determination

After the characteristics of a well fitted lens have been satisfied, conduct a **spherical over-refraction** to determine the proper lens power to be dispensed.

Example: Diagnostic lens: -4.50

Over-refraction: -0.25 Final lens power: -4.75

10

#### **FITTING GUIDELINES (Multifocal)**

The **DAILIES TOTAL1\* Multifocal** (delefilcon A) soft contact lens is a progressive aspheric simultaneous vision soft contact lens, intended to correct presbyopia with or without additional ammetropia, available in three ADD powers; low (LO), medium (MED) and high (HI). For each lens the near and intermediate powers are concentrated primarily in the central portion of the optical zone while the distance power is contained in the surrounding portion. The continuous changes in power across the surface of the lens allow patients requiring a reading addition of up to + 3.00D to see clearly at far, intermediate, and near distances.

Achieving high success with DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses is dependent on several factors, including the patient's motivation, expectations and visual wearing environment, as well as your skill in optimizing the lens powers to balance binocular performance at distance and near. The information in this guide is designed to provide you with the tools to manage your presbyopic patients through each stage of the process from the initial case history to post-fitting follow-up.

# 1. Pre-fitting Examination

# A pre-fitting examination is necessary to:

- determine whether a patient is a suitable candidate for DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses
- make ocular measurements and assessments for initial contact lens parameter selection
- collect baseline clinical information to which post-fitting examination results can be compared

#### A pre-fitting examination should include:

- a thorough case history
- detailed assessment of patient's individual visual demands
- understanding of patient's objectives for lens wear and expectations
- a distance spherocylindrical refraction, near add determination and measurement of pupil diameter
- keratometry
- tear assessment
- biomicroscopy

Note: The importance of a thorough case history should not be underestimated. The information gained through careful listening and probing will help greatly in satisfying each patient's unique needs.

#### 2. Patient Selection

The eye care professional should weigh several factors when considering patient selection for a DAILIES TOTAL1\* Multifocal (delefilcon A) soft contact lens fitting. When fitting a lens intended to correct for presbyopia, it is especially important to evaluate the particular visual needs, objectives, lifestyle and expectations of the individual patient. Prospective candidates may include current contact lens wearers, former wearers, and persons with no previous wear history. For former wearers it is important to determine the cause for discontinuation.

There are two general categories of candidates based on anticipated usage: those who seek to wear their lenses as their principal means

of vision correction, and those who wish to integrate the use of their contact lenses with spectacles. The integrative user often seeks to wear their lenses for sports or other occasional activities while reverting to spectacles under poor lighting or otherwise demanding vision conditions. In general, even the part-time user does not require more than a few moments re-adaptation time following an interval of no lens wear.

While candidates with greater than 1.00 diopter of refractive error have often been thought of as better candidates than those with low error or emmetropia, this is a generalization that often does not hold true for a given individual. Success is influenced by many factors and the eye care professional is encouraged to offer DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses to all interested presbyopic patients who satisfy the standard requirements for soft contact lens wear.

To summarize patient selection, the characteristics of "ideal candidates" and those that will be more difficult to fit" are listed below:

#### Ideal Candidates

- Refractive cylinder < 1.00D.</li>
- Attainable visual demands that do not depend upon resolving very fine (smaller than 20/20 letters) details at *both* distance and near for extended periods while wearing DAILIES TOTAL1\* Multifocal contact lenses.
- Emphasis on tasks where it is advantageous to have objects simultaneously in focus over a large range of viewing distances.
- Expectations consistent with actual everyday visual demands.
- Motivated to wear lenses and understands that vision may not always be as sharp as with spectacles for some distances or lighting conditions.
- Unable to adapt to monovision correction.

#### Less than Ideal Candidates

- Critical or very fine visual demands at both distance and near.
- Refractive cylinder ≥ 1.00D (any axis) in one or both eyes or against-the-rule refractive cylinder > 1.00D in one or both eyes.
- Monocular distance acuities poorer than 20/20 with spherical equivalent refractive correction.
- Myopic anisometropia where the refractive error for one of the two eyes is low (≤1.50D) and has not been habitually corrected.
- Pupil size larger (> 4 mm) or smaller (<3 mm) than norm for presbyopic population under natural illumination conditions.
- Abnormal binocular sensory function (e.g., amblyopia or strabismus).
- Expectation to discard and never use spectacles again, including reading glasses, even for special tasks or viewing conditions.
- Highly satisfied monovision wearers.
- Any other contraindications to successful contact lens wear such as tear abnormality or lid margin disease.

#### 3. Initial Lens Selection

#### A. Initial Base Curve Selection

DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses are available in a single 8.5 mm base curve.

#### **B. Initial Lens Power Selection**

Note: A careful maximum plus spherocylindrical refraction and nearpoint add determination should be conducted prior to selecting a DAILIES TOTAL1\* Multifocal (delefilcon A) trial lens. Autorefraction findings should be refined manually to rule out effects of instrument myopia and ensure proper control of residual accommodation.

The DAILIES TOTAL1\* Multifocal lens design makes selecting the initial lens power easy. You need only manipulate the distance power. The optimum starting point is with a power that is equal to or *more plus or less minus* than the vertex corrected spherical equivalent spectacle refraction.

#### C. Initial ADD Selection

Note: A careful nearpoint ADD determination should be conducted prior to selecting a DAILIES TOTAL1\* Multifocal (delefilcon A) trial lens

The DAILIES TOTAL1\* Multifocal (delefilcon A) 3 ADD SYSTEM allows personalized fitting for presbyopic patients. The table below makes initial ADD selection easy.

#### DAILIES TOTAL1\* MULTIFOCAL ADD SELECTION

| SPECTACLE ADD | BOTH EYES |
|----------------|-----------|
| Up to +1.25 | 0 |
| +1.50 to +2.00 | MED |
| +2.25 to +2.50 | 0 |

| Example 1: | OD | | os |
|-------------------------------------|------------------|--------|----------|
| Spherical Rx: | -4.50 -0.75 x 90 | | -4.00D |
| Spherical equivalent (least minus); | -4.75D | | -4.00D |
| Vertex corrected power: | -4.50D | | -4.00D |
| Spectacle Add: | | +0.75D | |
| Eye Dominance: | | OD | |
| Initial Trial Lens: | -4.50 LO | | -4.00 LO |

| Example 2: | OD | | os |
|---|---|---|---|
| Spherical Rx: | +4.25 -0.25 x 180 | | +4.00 D<br>-0.50 x 180 |
| Spherical equivalent (least minus): | +4.25D | | +3.75D |
| Vertex corrected power: | +4.50D | | +3.75D |
| Spectacle Add: | | +2.00D | |
| Eye Dominance: | | os | |
| Initial Trial Lens: | +4.50 MED | | +3.75 MED |

# 4. Initial Lens Fitting Evaluation

- a) Insert the lenses selected in Section 3 (above). If the exact power is not available, choose the next closest least minus/most plus lens power in your trial set.
- b) Allow the lenses to settle on the eyes for approximately 10 minutes. This allows time for the patient to adapt to the lenses and time for the lens to equilibrate with the patient's tears.
- c) Evaluate the fit of the lenses on the eye. The **Push-up Test** as described below is an important part of the lens evaluation. The following guidelines will be helpful in evaluating the physical fit of the lens:

#### **Characteristics of a Well-fitted Lens**

A well-fitted DAILIES TOTAL1\* Multifocal (delefilcon A) contact lens satisfies the following criteria:

- Full corneal coverage and good centration (no limbal exposure).
   A lens that is decentered > 1 mm, particularly temporal, is less likely to give adequate vision.
- Lens movement of 0.1 to 0.5 mm should be present to allow tear exchange under the lens during a blink in primary gaze or upward gaze and to avoid variable vision.

# Push-up Test:

- This test is a reliable indicator of a good fit. With the patient looking straight ahead, place your index finger on the patient's lower lid and nudge the edge of the lens upward while observing lens movement. Then pull the lid back down and observe the return of the lens.
- A well fitted lens will move freely upward, stopping shortly after passing the limbus and then return freely to its original position.
- 3. Good comfort.
- 4. Acceptable visual acuity with over-refraction.

# Characteristics of a Tight (Steep) Lens Fit

A tight or steep fit should not be dispensed. If a lens fit is judged to be too steep a flatter lens (larger base curve), if available, should be evaluated. A tight or steep lens fit would display some or all of the following characteristics:

- Good centration.
- Insufficient or no lens movement during a blink in primary gaze or upward gaze.
- Excessive conjunctival drag (visible movement of the conjunctival vessels when the lens moves during a blink or during the push-up test). Note: presbyopes often have loose conjunctiva, some conjunctival movement is occasionally seen and may not be a sign of a tight fit. See Push-up Test below.

#### **Push-up Test:**

- A tight fitting lens will resist movement. If successfully nudged upward, the lens may remain decentered or return slowly to its original position.
- Good comfort.
- Blurred vision between blinks.

#### Characteristics of a Loose (Flat) Lens Fit

If a lens fit is judged to be too flat a steeper lens (smaller base curve), if available, should be evaluated. A loose lens fit would display some or all of the following characteristics:

- 1. Decentration.
- Excessive lens movement during the blink in primary or upward gaze.

#### **Push-up Test:**

- A loose fitting lens will move very easily, well beyond the limbus and possibly encroaching upon or going beyond the pupil. It will then return very quickly to its original position and often times return lower than its original position.
- 3. Reduced comfort.
- 4. Lens edge standoff.
- 5. Blurred vision immediately after the blink.

#### 5. Initial Lens Visual Evaluation

While lenses are settling, it is helpful to take the patient from the exam room to a "real-world" setting such as a room with an outside view. Once an acceptable fit has been achieved, the visual performance of the lenses may be evaluated. Visual acuity is tested at distance. If necessary, a spherical over-refraction should be performed using a trial frame or hand held lenses rather than a phoropter. This technique is essential when fitting multifocal lenses because it allows the patient to maintain the head posture and direction of gaze (relationship between eye and head) that he or she would naturally use during everyday tasks. This ensures that the visual performance of the lens is being assessed under conditions where the on-eye positioning matches that which will occur when the lens is being used, for example, for near work activities. In addition, pupil size will not be artificially increased

15

by the reduction in light associated with looking through the aperture of the phoropter cells, or decreased by proximal cues associated with the nearness of the instrument.

### 6. Fitting Procedures

Step 1. After the trial lenses have settled for approximately 10 minutes, measure distance acuity while the patient is viewing the chart binocularly (i.e., simultaneously with both eyes). Next, evaluate the patient's subjective impression of the near vision when trying to read typical everyday material (e.g., a newspaper, magazine, and cell phone). Lighting and reading distance should be what is normal for the patient.

Step 2. If distance or near vision is unsatisfactory, perform a binocular distance over-refraction, as follows. Use hand-held trial lenses and encourage plus. For example, if a Plano and +0.25D over-refraction yields the same results, use the +0.25D endpoint. Re-check visual acuity and visual quality as described in Step 1 above. If over-refraction is other than plano, go immediately to new trial lenses, keeping ADD the same.

<u>Step 3</u>. If distance and near vision are satisfactory, dispense lenses and remind patient to use good light when reading fine print or use additional reading glasses if needed. It is helpful to let the patient experience the lenses in their natural environment before further procedures for enhancing vision are performed.

Step 4. Enhanced Near Vision. If near vision is unsatisfactory, determine the dominant eye by the following method. Determine the eye with greatest plus acceptance by placing +1.50 handheld trial lens over each eye alternately while patient views in the distance with both eyes open. Consider the eye for which binocular vision blurs *least* with the +1.50 to be the non-dominant eye. Other methods to determine the dominant eye are appropriate.

<u>Step 4A:</u> Check the patient's binocular acuity with +0.50 over the non-dominant eye to determine if near vision is improved and distance vision is still acceptable. If so, place a new trial lens with the same ADD on the non-dominant eye, adjusting the distance power by +0.50.

| Enhanced near vision, Step A | | |
|---|---|---|
| SPECTACLE ADD | DOMINANT EYE | NON-DOMINANT EYE<br>(PLUS ACCEPTED) |
| Up to +1.25 | (9) | with additional +0.50 |
| +1.50 to +2.00 | MED | with additional +0.50 |
| +2.25 to +2.50 | 9 | with additional +0.50 |

Next, re-check visual acuity and visual quality as described in Step 1 above. If satisfactory, dispense new distance lens power for the non-dominant eye. If near vision is still unsatisfactory, proceed to Step B:

Step4B: If near vision is still unsatisfactory, adjust ADD as shown below.

| Enhanced near vision, Step B | | |
|---|---|---|
| SPECTACLE ADD | DOMINANT EYE | NON-DOMINANT EYE<br>(PLUS ACCEPTED) |
| Up to +1.25 | MED | MED |
| +1.50 to +2.00 | (IED) | 0 |
| +2.25 to +2.50 | 0 | MED |

Note: It is common to question the rather non-intuitive step we suggest for enhancing vision at near in the HI ADD range, where the suggestion is to "back off" to a MED ADD for the non-dominant eye, the same suggestion we make for enhancing distance vision (below). The reason for this is that after establishing (in Step A) that increasing plus is not helpful, the next most common reason for blur at near (or distance) is unacceptable ghosting that degrades the image quality. Backing down to the MED ADD in one eye can often relieve that and actually improve vision at near.

<u>Step 5</u>: Enhanced Distance Vision. If distance over-refraction did not improve visual acuity, adjust ADD according to the chart below.

| SPECTACLE ADD | DOMINANT EYE | NON-DOMINANT EYE (PLUS ACCEPTED) |
|----------------|--------------|-----------------------------------|
| +1.50 to +2.00 | (6) | (m) |
| +2.25 to +2.50 | 0 | |

17

# FITTING GUIDELINES (Monovision)

#### Patient Selection

#### A. Monovision Needs Assessment

For a good prognosis, the patient should have adequately corrected distance and near visual acuity in each eye. Patients with reduced visual acuity, such as the amblyopic patient, may not be a good candidate for monovision.

Occupational and environmental visual demands should be considered. If the patient requires critical vision (visual acuity and stereopsis), it must be determined by trial whether this patient can function adequately with monovision. Monovision contact lens wear may not be optimal for such activities as:

- visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities: and
- driving automobiles (e.g., driving at night). Patients who cannot pass requirements for a driver's license with monovision correction should not drive with this correction. An additional over-correction can be prescribed to improve vision.

# B. Patient Education

All patients do not function equally well with monovision correction. Patients may not perform as well for certain tasks with this correction as they have with bifocal reading glasses. Each patient must understand that monovision, as well as other presbyopic contact lenses, or other alternatives, can create a vision compromise that may reduce visual acuity and depth perception for distance and near tasks. During the fitting process, it is necessary for the patient to realize the disadvantages as well as the advantages of clear near vision in straight-ahead and upward gaze that monovision contact lenses provide compared to spectacle bifocals.

#### **Eye Selection**

Generally, the non-dominant eye is corrected for near vision. The following test for eye dominance can be used:

# A). Ocular Preference Determination Methods

- Method 1 Determine which eye is the "sight eye". Have the
  patient point to an object at the far end of the room. Cover
  one eye. If the patient is still pointing directly at the object,
  the eye being used is the dominant (sighting) eye.
- Method 2 Determine which eye will accept the added power for near with the least reduction in distance vision. Place a trial spectacle near ADD lens in front of one eye and then the other while the distance refractive error correction is in place for both eyes. Determine whether the patient functions best with the near ADD lens over the right or left eye.

# B). Refractive Error Method

 For anisometropic corrections, it is generally best to fit the more hyperopic (less myopic) eye for distance and the more myopic (less hyperopic) eye for near.

## C). Visual Demands Method

 Consider the patient's occupation during the eye selection process to determine the critical vision requirements. If a patient's gaze for near tasks is usually in one direction, correct the eye on that side for near.

#### Example:

A person who places copy to the left side of the desk will usually function best with the near lens on the left eye.

## **Special Fitting Considerations**

#### **Unilateral Lens Correction**

There are circumstances where only one contact lens is required. As an example, an emmetropic patient would only require a near lens while a bilateral myope may require only a distance lens.

- · Examples:
- Emmetrope: A presbyopic emmetropic patient who requires a +1.75 diopter ADD would have a +1.75 lens on the near eye and the other eye left without a lens.
- Bilateral myope: A presbyopic patient requiring a +1.50 diopter ADD who is -2.50 diopters myopic in the right eye and -1.50 diopters myopic in the left eye may have the right eye corrected for distance and the left uncorrected for near.
- · Unilateral astigmat:
  - a) Emmetropic in one eye, astigmatic in the other

| Spectacle Rx | Potential Monovision Rx |
|---------------------|----------------------------|
| O.D. Plano | Uncorrected for distance |
| O.S1.00 -1.00 x 090 | +0.50 -1.00 x 090 for near |
| Add: +1.50 | |

Myopic in one eye, astigmatic in the other

| Spectacle Rx | Potential Monovision Rx |
|---------------------|--------------------------------|
| O.D1.50 | Uncorrected for near |
| O.S2.00 -1.75 x 090 | -2.00 -1.75 x 090 for distance |

## **Amblyopia**

The amblyopic patient may not be a good candidate for monovision.

# Astigmatism

Patients with less than 1.50 diopters of astigmatism might be successfully fit in DAILIES TOTAL1\* (delefilcon A) spherical lenses.

- Determine which eye to use for the near prescription (see Eye Selection, A-C, above)
- Add the appropriate near add power to the spherical component of the astigmatic prescription for that eye.

19

Example: Spectacle Rx Potential Monovision Rx

O.S.: -3.00 -1.75 x 165 -2.00 -1.75 x 165 for near

Add: +1.00 Dominant eye: O.D.

#### **Near Add Determination**

Always prescribe the lens power for the near eye that provides optimal near acuity at the midpoint of the patient's habitual reading distance. However, when more than one power provides optimal reading performance, prescribe the least plus (most minus) of the powers.

## **Trial Lens Fitting**

A trial lens fitting is performed in the office to allow the patient to experience monovision correction. Lenses are fit according to the directions in the *General Fitting Guidelines and Base Curve Selection* described earlier in the guide.

Case history and standard clinical evaluation procedures should be used to determine the suitability of monovision. Determine which eye is to be corrected for distance and which eye is to be corrected for near. Next determine the near ADD. With trial lenses of the proper power in place, observe the reaction to this mode of correction.

Immediately after the correct power lenses are in place, walk across the room and have the patient look at you. Assess the patient's reaction to distance vision under these circumstances. Then have the patient look at familiar near objects such as a watch face or fingernails. Again assess the reaction. As the patient continues to look around the room at both near and distance objects, observe the reactions. Only after these vision tasks are completed, should the patient be asked to read print. Evaluate the patient's reaction to large print (e.g., typewritten copy) at first and then graduate to news print and finally smaller type sizes.

After evaluating the patient's performance under the above conditions, tests of visual acuity and reading ability under conditions of moderately dim illumination should be attempted.

An initial unfavorable response in the office, while indicative of a less favorable prognosis, should not immediately rule out a more extensive trial under the usual conditions in which a patient functions.

# Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches, and feeling of slight imbalance. You should explain the adaptational symptoms to the patient. These symptoms may last for a few minutes or for several weeks. The longer these symptoms persist, the poorer the chance for successful adaptation. To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable, familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it is recommended that patients be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several

20

weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive under optimal driving conditions. After adaptation, and success with these activities, the patient should be able to drive under other conditions with caution.

### **Other Suggestions**

The success of the monovision technique may be further improved by having your patient follow the suggestions below:

- Have a third contact lens (distance power) to use when critical distance viewing is needed.
- Have a third contact lens (near power) to use when critical near viewing is needed.
- Have supplemental spectacles to wear over the monovision contact lenses for specific visual tasks. This is particularly applicable for those patients who cannot meet driver's licensing requirements with a monovision correction.
- Make use of proper illumination when carrying out visual tasks.

Success in fitting monovision can be improved by the following suggestions:

- Reverse the distance and near eyes if a patient is having trouble adapting.
- Refine the lens powers if there is trouble with adaptation. Accurate lens power is critical for presbyopic patients.
- Emphasize the benefits of the clear near vision in straight ahead and upward gaze with monovision.

The decision to fit a patient with a monovision correction is most appropriately left to the eye care professional in conjunction with the patient after carefully considering the patient's needs. All patients should be supplied with a copy of the **Patient Instruction Booklet**, which contains important instructions for the monovision wearer. You can obtain copies of the instruction book by calling customer service **in the USA at (800) 241-5999.** 

#### **DISPENSING VISIT**

To help ensure patient success the following steps should be conducted with each patient, even if they have previously worn contact lenses. Even experienced wearers are prone to develop bad habits over time.

DAILIES TOTAL1\* brand (delefilcon A) lenses are supplied sterile in foil sealed blister pack containers. Open the foil pack by peeling back the foil lidding material and gently slide the lens out of the container with your finger, or pour the lens onto the palm of your clean hand.

Conduct the following steps with each patient, even if they have previously worn contact lenses:

# A. Verification of Lens Fit

Evaluate lens fit and visual response with the lens on the eye. The criteria of a well-fitted lens should be met and the patient's visual acuity should be acceptable. If not, the patient should be refitted with a more appropriate lens

#### B. Hygiene and Lens Handling Instructions

Good hygiene and proper lens handling are important factors in achieving safe, comfortable lens wear. Instruct the patient on hygiene and handling of lenses. Patients who are unable to place and remove lenses should not be provided with them.

## C. Lens Wear and Replacement Schedules (see Package Insert)

Prescribe and explain the daily disposable wear schedule. Explain that lenses are to be discarded after each daily wearing period. Determine the maximum suggested daily wearing period based on the patient's physiological eye condition. There may be a tendency for the patient to overwear their lenses initially. For some patients who have never worn contact lenses consider a wearing schedule that allows for a gradual increase in wearing time.

# D. Lens Care Directions (see Package Insert)

The lenses are not intended to be cleaned or disinfected and should be discarded after a single use. The eye care professional may recommend lens rewetting drops, as needed.

### E. Specific Instructions for Presbyopic Patients

Specific instructions, explanations and demonstrations are important for optimizing patient success with multifocal contact lenses. The following information and instructions have proven useful in advising patients who wear DAILIES TOTAL1\* Multifocal (delefilcon A) soft contact lenses.

- A contact lens that contains different powers for distance and near involves greater technological and optical complexity than does a bifocal or multifocal spectacle lens. This is because the contact lens moves with the eye, rather than having the eye move up and down while the lens remains suspended in a frame. While the contact lens therefore gives an unobstructed field of view and greater freedom regarding where to look, these advantages may mean that the sharpness of vision may not always be exactly the same as what would be experienced with spectacles.
- Although many individuals use DAILIES TOTAL1\* Multifocal (delefilcon A) contact lenses for full-time wear, it is not unusual to find that there may be some activities where one prefers to wear spectacles, or where the disadvantages associated with spectacles are outweighed by other issues. This is an entirely normal and natural response to the challenges presented by presbyopia.
- Situations where vision with multifocal contact lenses may be less sharp or otherwise "different" than what is experienced with spectacles often involve low illumination (e.g., a semi-dark room), reduced visibility (e.g., outdoor conditions of fog or heavy rain), or isolated sources of very bright light (e.g., headlights of an oncoming vehicle on a narrow country road). Patients should be instructed to make use of good light when reading fine print.
- Patients should be aware that it might be advisable to refrain from wearing their lenses while driving, flying an airplane or operating heavy machinery while wearing their lenses until they gain some experience with the lenses in a similar visual environment.
- Small changes in lens power can often make a significant difference in the quality of the vision experienced with multifocal contact lenses. Such changes can be best tailored to

individual needs and environmental conditions that the patient will personally encounter on a day-to-day basis. Confidence and assurance that such refinements, if needed, can be achieved are important for patient motivation during the initial period of lens wear.

# F. Additional Instructions

#### Review the Package Insert

Provide the patient with all relevant information and precautions on the proper use of the lenses that are prescribed.

Provide the Patient Instruction Booklet for DAILIES TOTAL1\*
and DAILIES TOTAL1\* Multifocal (delefilcon A) Contact Lenses.
Give the patient a copy of the Patient Instruction Booklet for DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal (delefilcon A) soft contact lenses. Review the contents so the patient clearly understands the prescribed lens wear, care, and replacement schedule. In the USA you can obtain copies of the instruction book by calling Alcon customer service at (800) 241-5999.

## **Follow-Up Examinations**

Follow-up care is extremely important for continued successful contact lens wear. Follow-up care should include:

- Case history, including questions to identify any problems related to contact lens wear
- · Management of specific problems, if any, and
- A review with the patient of the lens wearing schedule, replacement schedule and handling procedures.

# **Follow-up Examination Procedures**

- Patients should be instructed to wear lenses prior to a follow-up examination.
- Record patient's symptoms, if any.
- Measure visual acuity monocularly and binocularly with the contact lenses in place.
- · Perform an over-refraction to check for residual refractive error.
- · With a biomicroscope, evaluate lens fitting.
- Remove the lenses and conduct a thorough biomicroscopic examination with fluorescein. Rinse eyes with saline before re-inserting lenses.
- Evert upper lids to determine condition of tarsal conjunctiva.
- Periodically perform keratometry and spectacle refractions. These results should be recorded to compare to the initial measurements.
- If any observations are abnormal, use professional judgment to manage the problem and restore the eye to optimal conditions. If visual requirements are not satisfied during any follow-up examination, the patient should be re-fitted with a more appropriate lens.

# **LENS HANDLING HINTS**

# **Lens Insertion**

 When about to place the lens on the eye, make sure the lens sits up on the placement finger. The finger should be dry so surface tension does not cause the lens to adhere to the finger.

 Check to see that the lens is right side out. A lens that is placed on the eye inside out may not feel comfortable or provide good vision.

One way to do this is to perform the 'taco test' by placing the lens between your thumb and index finger and squeeze the edges together gently.

- If the edges come together, the lens is right side out.
- If the edges turn outward, the lens is wrong side out. Carefully reverse it with your fingers.



Another way is to place the lens on the tip of your index finger and check its shape.

- If the edge appears bowl-shaped, it is right side out.
- If the edge has a lip or flares outward, it is wrong side out and must be reversed.
- Place the lens directly onto the cornea (placing it on the lower sclera can lead to the lens folding after a blink). While continuing to hold both lids in place, the patient should look down to seat the lens. The lids may then be released.



#### Lens Removal

- Wash hands thoroughly with soap that does not have any oils, lotions or perfumes.
- Carefully dry hands with a clean, lint-free towel.

It is important to remind patients to **dry their hands thoroughly** prior to removing their lenses. The surface of DAILIES TOTAL1\* brand lenses is designed to stay very wet and lubricious, or slippery while on the eye. If their fingertips are wet they are likely to slip across the surface of the lens making removal more difficult.

- Slide the lens off the cornea (down or to the side) onto the sclera. This
  produces a fold in the lens, which assists in removal. With the index finger
  and thumb, gently pinch the lens off the eye.
- Discard lenses.

# Care for a Sticking Lens

In the unlikely event that the lens sticks (stops moving) or begins to dry on the eye, instruct the patient to apply several drops of a recommended lubricating solution (used in accordance with package labeling). The patient should wait until the lens begins to move freely on the eye before attempting to remove it. If the lens continues to stick, the patient should immediately consult the eye care professional.

#### IN OFFICE CARE OF TRIAL LENSES

Eye care professionals should understand and educate contact lens technicians concerning proper use of trial lenses.

- Each contact lens is shipped sterile in a sealed blister pack containing phosphate buffered saline with additives. Hands should be thoroughly washed and rinsed and dried with a lint-free towel prior to handling a lens. In order to insure sterility, the blister pack should not be opened until immediately prior to use.
- Delefilcon A lenses are for daily disposable wear only and should be discarded after a single use. The lenses should be disposed of after a single use and not be re-used from patient to patient.

#### ADDITIONAL INFORMATION

For assistance with fitting or clinical questions regarding DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal contact lenses eye care professionals having questions or problems should contact Medical Information Systems in the USA at (800) 241-7468. To order DAILIES TOTAL1\* and DAILIES TOTAL1\* Multifocal contact lenses contact your Alcon sales representative or call Customer Service, in the USA at (800) 241-5999.
#### VERTEX DISTANCE CONVERSION CHART

For minus lenses, read left to right; for plus lenses, read right to left. (12 mm Vertex Distance)

| - | + | - | + | - | + | - | + |
|------|------|-------|-------|-------|-------|-------|-------|
| 4.00 | 3.87 | 7.50 | 6.87 | 12.00 | 10.37 | 19.00 | 15.50 |
| 4.25 | 4.00 | 7.62 | 7.00 | 12.50 | 10.75 | 19.25 | 15.62 |
| 4.50 | 4.25 | 7.75 | 7.12 | 12.75 | 11.00 | 19.25 | 15.75 |
| 4.75 | 4.50 | 7.87 | 7.25 | 13.00 | 11.25 | 19.75 | 16.00 |
| 5.00 | 4.75 | 8.00 | 7.37 | 13.50 | 11.50 | 20.00 | 16.12 |
| 5.12 | 4.87 | 8.12 | 7.50 | 13.75 | 11.75 | 20.25 | 16.25 |
| 5.37 | 5.00 | 8.25 | 7.62 | 14.00 | 12.00 | 20.50 | 16.50 |
| 5.50 | 5.12 | 8.50 | 7.75 | 14.25 | 12.25 | 20.75 | 16.62 |
| 5.62 | 5.25 | 8.75 | 8.00 | 14.75 | 12.50 | 21.00 | 16.75 |
| 5.75 | 5.37 | 9.00 | 8.25 | 15.00 | 12.75 | 21.25 | 17.00 |
| 5.87 | 5.50 | 9.25 | 8.37 | 15.50 | 12.75 | 21.75 | 17.25 |
| 6.00 | 5.62 | 9.50 | 8.62 | 15.75 | 13.25 | 22.25 | 17.50 |
| 6.12 | 5.75 | 9.75 | 8.75 | 16.25 | 13.50 | 22.50 | 17.75 |
| 6.37 | 5.87 | 10.00 | 9.00 | 16.75 | 13.75 | 23.00 | 18.00 |
| 6.50 | 6.00 | 10.25 | 9.12 | 17.00 | 14.00 | 23.50 | 18.25 |
| 6.62 | 6.12 | 10.50 | 9.25 | 17.25 | 14.25 | 23.75 | 18.50 |
| 6.75 | 6.25 | 10.75 | 9.37 | 17.62 | 14.37 | 24.25 | 18.75 |
| 6.87 | 6.37 | 11.00 | 9.62 | 18.00 | 14.50 | 24.75 | 19.00 |
| 7.00 | 6.50 | 11.25 | 9.75 | 18.12 | 14.75 | 25.00 | 19.25 |
| 7.12 | 6.62 | 11.50 | 10.00 | 18.50 | 15.00 | 25.50 | 19.50 |
| 7.37 | 6.75 | 11.75 | 10.25 | 18.75 | 15.25 | 26.00 | 19.75 |

This page

left blank



- ..-.!MQmlinllra ..-.!MQmlinllra

Th dearo!!| |>fb.||"loihi|\_..\_lhil prinoor.!lme! | |-fb.||"loihi|\_..\_lhil prinoor.!lme!! | |-fi.|| | |-fi.

| Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent | Independent |

• · li)'o,-lilrurtl:lt-..tollollio-.....1hiljiil>lll'll: 0j1111Llliol--tlilo!lyii...:l

-!R!I'Irliotw|<|ii !R!dry!<i111111bb' .m.s-..|!|'|!na--.!wd&||-. - PB:oan""1hi|1|pd)'|U'dirMA!|i|dryrQii"|i||t

d.
-iJt11wigw¥.:<1fii!"hiMt111fii!tii4'iJiifiji}¥ikL
-filalibii!Mditidi-j!411hii | ji|>(:!Yiii)ii)a Idiifi;!yroli
IJQii!'"firomilitit!V.
-ImI<-m:|III<!!My-t1•-.-II\11hii

-lmi< -A!III-.....ihiI--

..-.01hII-lil <sup>\*</sup>

-R!Imiiwihillirlllirt ll'Itr-Ihiltillilli: ll'III--Do|>III:plndItio!I)'O--ril'IfI!m!!!(IIIkdItn W¥ --iIi>:I yl:iM.Dini'IMII!TiviiIIVJ !=IIIItni:& IfIllildilo::olmlf11)111halli't,tIllijliilo tl-

I-ft91r.jlia1hilmll!dla11rGor<ll!hl Il'IllrJII'llokwitlo•!. .IUfii JII



### 

Elido...-n atoipps||j-|n\*-Pid|"""\*\*|rol| W'Iwdulll'Ilid1 bi.lliRtdIllih!Ktlliil Willid ==das Ilid1 MUILIER tri IMUM privit hidd II akw.llillidirull'Ilill.R 1 habilillidir (inid1b) ojuriio!-niim11:ilillidir ...-F!!rfilrQiiiHI--

Thii IIUJIIIboii'IITinII:IIiiIIN\_ol... Ilind U>IImIdd:1 ;oidI!-q IIIIi:IrmII!IIJ it;m>HwildiiIII;malliiiJ Arliiii IIII | III WII IIIII|-III!NulliiiIIII 1 !! M riilon M !!!iriIIIr hmr; 0 | 0



This page

left blank

This page

left blank



a Novartis company

Manufacturer: Alcon Laboratories, Inc. 6201 South Freeway Fort Worth, TX 76134-2099, USA

© 2016 Novartis
\*a trademark of Novartis

March 2016

www.alcon.com W900087400-0316

## APPENDIX H: ALCON AIR OPTIX MULTIFOCAL CONTACT LENS PLUS HYDRAGLYDE FITTING GUIDE

# Professional Fitting and Information Guide

AIR OPTIX\* AQUA, AIR OPTIX\* plus HydraGlyde\*,
AIR OPTIX\* for Astigmatism,
AIR OPTIX\* plus HydraGlyde\* for Astigmatism,
AIR OPTIX\* AQUA Multifocal,
AIR OPTIX\* plus HydraGlyde\* Multifocal (lotrafilcon B)
Soft Contact Lenses

For Daily Wear and Extended Wear up to 6 Nights



CAUTION: FEDERAL LAW (UNITED STATES)
RESTRICTS THIS DEVICE TO SALE BY OR
ON THE ORDER OF A LICENSED EYE CARE
PROFESSIONAL



This page

left blank

#### **Table of Contents**

| INTRODUCTION | |
|-----------------------------------------------------------|----|
| PRODUCT DESCRIPTION | 5 |
| Lens Properties | 5 |
| Available Lens Parameters | 5 |
| Actions | 6 |
| INDICATIONS (Uses) | |
| CONTRAINDICATIONS, WARNINGS, PRECAUTIONS & ADVERSE EFFECT | |
| ADVERSE EFFECT REPORTING | |
| LENS CARE DIRECTIONS | |
| FITTING GUIDELINES (Spherical Lenses) | |
| Patient Selection | |
| Pre-fitting Examination | |
| Trial Lens Evaluation | |
| Lens Base Curve Selection | |
| Initial Lens Power Selection | |
| Lens Fit Assessment | |
| Final Lens Power Determination | |
| FITTING GUIDELINES (Toric Lenses) | |
| FITTING GUIDELINES (Multifical Lenses) | |
| FITTING GUIDELINES (Monovision) | |
| DISPENSING VISIT | 30 |
| FOLLOW-UP EXAMINATIONS | |
| FOLLOW-UP EXAMINATION PROCEDURES | |
| LENS HANDLING HINTS | |
| Lens Insertion | |
| Lens Removal | |
| Care for a Sticking Lens | |
| IN OFFICE CARE OF TRIAL LENSES | |
| ADDITIONAL INFORMATION | |
| VERTEX DISTANCE CONVERSION CHART | |
| PRODUCT PACKAGE INSERT | |
| LENS CARE PRODUCT CHART FOR SOFT CONTACT LENSES. | 38 |

This page

left blank

#### INTRODUCTION

Thank you for prescribing Alcon AIR OPTIX\* AQUA, AIR OPTIX\* plus HydraGlyde\*, AIR OPTIX\* for Astigmatism, AIR OPTIX\* plus HydraGlyde\* for Astigmatism, AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal (lotrafilcon B) soft contact lenses. The lenses may be worn for daily wear and extended wear for up to six continuous nights with removal for disposal, or cleaning and disinfection (chemical, not heat) prior to reinsertion, and frequent replacement with a fresh new lens.

However, you will determine the replacement schedule as well as the length of time the patient's lenses are to be worn each day before removal for cleaning, rinsing, and disinfection. Based on these schedules, you will also determine the number of lenses each patient requires. This guide contains important information regarding fitting procedures and aftercare of the AIR OPTIX\* AQUA, AIR OPTIX\* plus HydraGlyde\*, AIR OPTIX\* for Astigmatism, AIR OPTIX\* plus HydraGlyde\* for Astigmatism, AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal (lotrafilcon B) contact lens patient.

#### PRODUCT DESCRIPTION

Alcon AIR OPTIX\* AQUA, AIR OPTIX\* plus HydraGlyde\*, AIR OPTIX\* for Astigmatism, AIR OPTIX\* plus HydraGlyde\* for Astigmatism, AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal (lotrafilcon B) contact lenses are available in spherical, toric, and multifocal lens designs. The lens material is approximately 33% water and 67% lotrafilcon B, a fluoro-silicone containing hydrogel that is surface treated. Lenses contain the color additive copper phthalocyanine, a light blue handling tint which makes them easier to see when handling. This breakthrough lens material provides a high level of oxygen to the eyes and has been surface treated to wet with the tears.

#### **Lens Properties**

Refractive Index (hydrated): 1.42
 Light Transmittance: ≥ 96%

Oxygen Permeability (Dk):
 110 x 10 -11 (cm<sup>2</sup>/sec)(ml O<sub>2</sub>/ml x mm Hg),

measured at 35° C (intrinsic Dk -

Coulometric method)

Water Content
 33% by weight in normal saline

## Available Lens Parameters<sup>1</sup> AIR OPTIX\* AQUA contact lenses

• Chord Diameter: 14.2 mm

• Center Thickness: 0.08 mm @ -3.00D (varies with power)

• Base Curve: 8.6 mm

Powers: -0.25 to -8.00D (0.25D steps);

-8.50 to -10.00D (0.50D steps)

Plus Powers: +0.25 to +6.00D (0.25D steps)

#### AIR OPTIX\* plus HydraGlyde\* contact lenses

• Chord Diameter: 14.2 mm

• Center Thickness: Varies with power (0.08 mm @ -3.00D)

Base Curve: 8.6 mm

Powers: -0.25 to -8.00D (0.25D steps);

-8.50 to -12.00D (0.50D steps)

Plus Powers: +0.25 to +6.00D (0.25D steps);

+6.50 to +8.00D (0.50D steps)

<sup>&</sup>lt;sup>1</sup> Check for actual product availability as additional parameters may be introduced over time.

## AIR OPTIX\* for Astigmatism<sup>2</sup> and AIR OPTIX\* plus HydraGlyde\* for Astigmatism contact lenses

• Chord Diameter: 14.5 mm

• Center Thickness: 0.102 mm @ -3.00D (varies with power)

• Base Curve: 8.7 mm

• Powers: Minus Powers: plano to -6.00D (0.25D steps):

-6.50 to -10.00D (0.50D steps)

Plus Powers: +0.25 to +6.00D (0.25D steps) Cylinder power: -0.75, -1.25, -1.75, -2.25

Axis: full circle (10° steps)

## AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal contact lenses

• Chord Diameter: 14.2 mm

• Center Thickness: 0.08 mm @ -3.00D (varies with power)

• Base Curve: 8.6 mm

Powers: Minus Powers: plano to -10.00D (0.25D steps)

Plus Powers: +0.25 to +6.00D (0.25D steps)

ADD: LO, MED, HI

NOTE: Hereafter, lotrafilcon B spherical, toric, and multifocal lenses may be referred to as lotrafilcon B contact lenses unless product distinction is necessary.

#### Actions

When hydrated and placed on the cornea, lotrafilcon B contact lenses act as a refracting medium to focus light rays on the retina.

#### INDICATIONS (Uses)

AIR OPTIX\* AQUA and AIR OPTIX\* plus HydraGlyde\* (lotrafilcon B) spherical soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes and up to approximately 1.50 diopters of astigmatism that does not interfere with visual acuity.

AIR OPTIX\* for Astigmatism and AIR OPTIX\* plus HydraGlyde\* for Astigmatism (lotrafilcon B) toric soft contact lenses are indicated for the optical correction of refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes and up to 6.00 diopters (D) or less of astigmatism.

AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal (lotrafilcon B) multifocal soft contact lenses are indicated for the optical correction of presbyopia, with or without refractive ametropia (myopia and hyperopia) in phakic or aphakic persons with non-diseased eyes who may require a reading addition of +3.00 diopters (D) or less and who may have up to approximately 1.50 diopters of astigmatism.

The lenses may be prescribed for daily wear or extended wear for up to 6 nights of continuous wear with removal for disposal, or cleaning and disinfection (chemical, not heat) prior to reinsertion and frequent replacement, as recommended by the eye care professional.

See *Warnings* for information about the relationship between wearing schedule and corneal complications.

<sup>&</sup>lt;sup>2</sup> May also be labeled as O<sub>2</sub>OPTIX\* for Astigmatism

#### CONTRAINDICATIONS, WARNINGS, PRECAUTIONS & ADVERSE EFFECTS

For additional important prescribing and safety information, refer to the **Package Insert** that is printed in the back of this guide.

#### **ADVERSE EFFECT REPORTING**

If a patient experiences any serious adverse effects associated with the use of Alcon® (lotrafilcon B) contact lenses, please notify Alcon Medical Safety in the USA at 1-800-757-9780.

#### **LENS CARE DIRECTIONS**

For general information about contact lens care, refer to the **Package Insert** that is printed in the back of this guide.

#### **FITTING GUIDELINES**

Please see the appropriate sections of this booklet that contain guidelines for spherical, toric, multifocal, and monovision fitting techniques.

#### FITTING GUIDELINES (Spherical Lenses)

#### 1. Patient Selection

The patient characteristics necessary to achieve success with **AIR OPTIX\* AQUA** and **AIR OPTIX\* plus HydraGlyde\*** (lotrafilcon B) soft contact lenses are similar to those for other spherical soft contact lenses. A thorough pre-fitting examination should be conducted to ensure the patient is a suitable candidate for soft contact lens wear.

The following procedures should be followed when fitting **AIR OPTIX\* AQUA** and **AIR OPTIX\* plus HydraGlyde\*** (lotrafilcon B) contact lenses. For additional tips on fitting the monovision patient refer to the section *Fitting guidelines* (*Monovision*).

#### 2. Pre-fitting Examination

#### A pre-fitting examination is necessary to:

- assess the patient's motivation, physical state and willingness to comply with instructions regarding hygiene and wear schedule
- make ocular measurements for initial contact lens parameter selection
- collect baseline clinical information to which post-fitting examination results can be compared

#### A pre-fitting examination should include:

- · a thorough case history
- · a spherocylindrical refraction
- keratometry
- · tear assessment
- biomicroscopy

#### 3. Trial Lens Evaluation

#### A. Lens Base Curve Selection:

A well-fitted lens provides good movement, centration and comfort. This can be achieved for the majority of patients with the 8.6 mm base curve.

#### B. Initial Lens Power Selection

The initial power selection should be as close as possible to the patient's prescription after taking into account spherical equivalent and vertex calculations, if necessary.

#### **Spherical Equivalent Calculation**

To determine initial lens power, convert the spherocylindrical spectacle Rx to its spherical equivalent as follows:

Spherical Equivalent = Sphere power +  $\frac{1}{2}$  (Cylinder Power)

Example: Spectacle Rx: -4.50D -1.00 x 180

Spherical equivalent: -4.50D + (-0.50D) = -5.00D

#### **Vertex Distance Conversion**

If the spherical equivalent is greater than ± 4.00D, a vertex distance correction is necessary (see *Vertex Distance Conversion Chart*) to determine the lens power required at the corneal plane.

Example: Spectacle Rx: -4.50D -1.00 x 180

Spherical equivalent: -4.50D + (-0.50D) = -5.00D Vertex compensation: -4.75 (initial lens power)

#### C. Lens Fit Assessment

Allow the lenses to settle on the eyes for approximately **5 to 10 minutes**. This allows time for the patient to adapt to the lenses and time for the lens to equilibrate.

Evaluate the fit and movement of the lenses on the eye. The **Push-up Test**, as described below, is an important part of the lens evaluation. The following guidelines will be helpful in fit evaluation:

#### Characteristics of a Well-fitted Lens

A well-fitted **AIR OPTIX\* AQUA** and **AIR OPTIX\* plus HydraGlyde\*** (lotrafilcon B) contact lens satisfies the following criteria:

- 1. Good centration and full corneal coverage in all fields of gaze.
- 2. Sufficient lens movement to allow tear exchange under the lens during a blink in primary or upward gaze.
- 3. Satisfactory Push-up Test
  - This test is a reliable indicator of a good fit. With the patient looking straight ahead, place your index finger on the patient's lower lid and nudge the edge of the lens upward while observing lens movement. Then pull the lid back down and observe the return of the lens.
  - A well-fitted lens will move freely upward, stopping shortly after passing the limbus and then return freely to its original position.
- 4. Good comfort and stable visual response (with over refraction).

#### Characteristics of a Tight (Steep) Lens Fit

A tight or steep fit should not be dispensed. If a lens fit is judged to be too steep a flatter lens (larger base curve), if available, should be evaluated. A tight or steep lens fit would display some or all of the following characteristics:

- Insufficient or no lens movement during a blink in primary or upward gaze.
- 2. Unsatisfactory Push-up Test
  - A tight fitting lens will resist movement. If successfully nudged upward, the lens may remain decentered or return slowly to its original position.
- 3. Good centration.
- 4. Good comfort.
- 5. Fluctuating vision between blinks.

#### Characteristics of a Loose (Flat) Lens Fit

If a lens fit is judged to be too flat, a steeper lens (smaller base curve), if available, should be evaluated. A loose lens fit would display some or all of the following characteristics:

- Lens edge standoff. Even minor lifting of the edge indicates a loose fitting lens.
- Reduced comfort. This finding is often the only signal of a loose fitting lens. If initial comfort doesn't improve quickly, try a steeper base curve, if available
- 3. Excessive lens movement during the blink in primary or upward gaze.
  - A loose fitting lens will move very easily, well beyond the limbus and
    possibly encroaching upon or going beyond the pupil. It will then return
    very quickly to its original position and often times return lower than its
    original position.
- 4. Poor centration with limbal exposure on exaggerated eye movement.
- 5. Vision may be blurred after the blink.

#### **General Fitting Tips**

- Trial fitting of the individual eye is strongly recommended.
- A well-fitted lens will show movement of 0.1 to 0.5 mm.
- When prescribing lotrafilcon B contact lenses for extended wear, it is important to reevaluate the lens fit for adequate movement at various times after the patient sleeps while wearing lenses. This reevaluation should include a follow-up visit as soon as possible after the patient awakens from sleeping, as well as at other times of the day. If the fit is judged to be too tight or steep, the patient must be refit into a lens that provides the criteria of a well-fitted lens.

#### D. Final Lens Power Determination

After the characteristics of a well-fitted lens have been satisfied, conduct a **spherical over-refraction** to determine the proper lens power to be dispensed.

#### Example:

Diagnostic lens: -4.50D Over-refraction: -0.25 Final lens power: -4.75D

#### FITTING GUIDELINES (Toric Lenses)

The geometry of an AIR OPTIX\* for Astigmatism and AIR OPTIX\* plus HydraGlyde\*for Astigmatism (lotrafilcon B) toric contact lens is a prism ballast design. The prism ballast design uses a toric geometry on one surface of the lens and spherical on the opposite. Stabilization is achieved by the prism at the vertical meridian on the front surface (dynamic stabilization) and with cylinder power parameters on the back surface.

To aid the fitting process, AIR OPTIX\* for Astigmatism and AIR OPTIX\* plus HydraGlyde\* for Astigmatism contact lenses feature three scribe lines on the front lens surface to enable assessment of the lens orientation. These lines are at 3, 6 and 9 o'clock positions approximately 1.0 mm in from the lens edge, with the 6 o'clock scribe line being slightly wider than the others. The lens orientation findings are then used for calculation of axis compensations.

#### 1. Patient Selection

The patient characteristics necessary to achieve success with AIR OPTIX\* for Astigmatism and AIR OPTIX\* plus HydraGlyde\* for Astigmatism contact lenses are similar to those for spherical lenses. A thorough pre-fitting examination should be conducted to ensure the patient is a suitable candidate for soft contact lens wear.

The following procedures should be followed when fitting AIR OPTIX\* for Astigmatism and AIR OPTIX\* plus HydraGlyde\* for Astigmatism lenses. For additional tips on fitting the monovision patient refer to the section *Fitting Quidelines (Monovision)*.

#### 2. Pre-fitting Examination

#### A pre-fitting examination is necessary to:

- Determine whether a patient is a suitable candidate for contact lenses in general (see the *Package Insert*, *indications* and *Contraindications* sections)
- Determine whether a patient is astigmatic to a degree requiring a toric visual correction
- Make ocular measurements for initial contact lens parameter selection
- Collect baseline clinical information to which post-fitting examination results can be compared

#### A pre-fitting examination should include:

- A thorough case history
- · A spherocylindrical refraction
- Keratometry
- Tear assessment
- Biomicroscopy

#### 3. Fitting Methods

The following method is recommended for fitting AIR OPTIX\* for Astigmatism and AIR OPTIX\* plus HydraGlyde\* for Astigmatism soft contact lenses to maximize success. This method allows for an extended trial period outside the office which will help the eye care professional to minimize chair time, reduce trial lens usage and inventories, as well as increase the accuracy of final lens orientation and the final multipack prescription.

#### **Trial Period Method**

- a) Make initial base curve selection if more than one available
- b) Determine the appropriate sphere and cylinder power
- c) Select cylinder axis based on spectacle prescription assume no rotation
- d) Place trial lens on the eye. Order trial lens if it is not in office inventory having the correct lens allows the patient to experience good vision during the trial period
- e) Evaluate fit, vision, and lens orientation
- f) Dispense lens if characteristics of a Well-fitted Lens are satisfied
- g) Reevaluate fit, vision, and lens orientation at the end of the trial period (typically a few days to a week)
- h) Order multipack after fitting adjustments, if any, are made to satisfy the characteristics of a **Well-fitted Lens**

The following alternatives are offered to describe the more traditional methods of fitting lenses. While these methods are adequate to use, they can lead to an increase in chair time, trial lens usage, and multipack purchases as the fit and vision of the lens are refined.

#### **Empirical Method**

- a) Make initial base curve selection if more than one available
- b) Determine the appropriate sphere and cylinder
- c) Select the cylinder axis assuming zero rotation
- d) Order multipack
- e) Evaluate fit, vision, and lens orientation
- f) Dispense lens if characteristics of a Well-fitted Lens are satisfied
- g) Reorder multipacks if adjustments are made

#### In Office Trial Lens Fitting Method

- a) Make base curve selection if more than one available
- b) Select diagnostic lens with similar sphere, cylinder power and axis as spectacle Rx
- c) Evaluate fit, vision, over-refraction, and lens orientation
- d) Order multipack if characteristics of a Well-fitted Lens are satisfied
- e) Reorder multipack if further adjustments are necessary

NOTE: For information on fitting the monovision wearer with toric lenses, please refer to the *Fitting guidelines (Monovision)* section.

#### 4. Initial Base Curve Selection

 A Well-fitted Lens provides good movement, centration, and comfort with the available 8.7 base curve.

#### 5. Initial Lens Power Selection

#### **Spherical Lens Power:**

- To determine the initial lens spherical power, use the spherical component of the spectacle Rx in minus cylinder form.
- If this spherical component is greater than ± 4.00D, a vertex distance correction is necessary. This will determine the spherical lens power required at the corneal plane.

#### Cylinder Lens Power:

Up to four cylinder powers may be available for AIR OPTIX\* for Astigmatism and AIR OPTIX\* plus HydraGlyde\* for Astigmatism contact lenses. When available, these four powers will normally allow correction of -0.75 to -3.00 diopters of astigmatism.

Select AIR OPTIX\* for Astigmatism contact lens cylinder power according to the chart below:

| Refraction Vertexed | AIR OPTIX* for Astigmatism and<br>AIR OPTIX* plus HydraGlyde* for<br>Astigmatism contact lens |
|---|---|
| Cylinder Power | Astiginatism contact lens |
| | Cylinder Power |
| -0.75 | -0.75 |
| -1.00 | -0.75 |
| -1.25 | -1.25 |
| -1.50 | -1.25 |
| -1.75 | -1.75 |
| -2.00 | -1.75 |
| -2.25 | -2.25 |
| -2.50 | -2.25 |
| -2.75 | -2.25 |
| -3.00 | -2.25 |

**Note:** If the combination of sphere power and cylinder power is greater than  $\pm 4.00D$ , vertex distance compensation must be performed for each power meridian.



#### Example:

Spectacle Rx: -5.00D - 1.50 x 180 (vertex distance =

12 mm)

Corneal Plane Rx: -4.75 -0.75 x 180

Toric Rx: -4.75 -0.75 x 180 (assuming no rotation)

 When the difference between the cylinder correction at the corneal plane and the selected cylinder to fit the patient differs by 0.50D or more, it is necessary to make a compensation to the spherical component using the following formula:

Corneal plane cylinder - Selected cylinder = Spherical Compensation

**Example:** 

**Spectacle Rx:** -4.50 -1.50 x 180

**Corneal Plane Rx:** -4.25 -1.25 x 180

Selected cylinder power: -0.75D

**Spherical adjustment needed** = -1.25 - (-0.75) / 2 = -0.25

**Toric Rx:** -4.50 -0.75 x 180 (assuming no rotation)

#### 6. Lens Fit Evaluation

a) Allow the lenses to settle on the eyes for approximately 5 to 10 minutes. This allows time for the patient to adapt to the lenses and time for the lens to equilibrate with the patient's tears, replacing the buffered, isotonic saline which was in the foil pack.

- b) AIR OPTIX\* for Astigmatism and AIR OPTIX\* plus HydraGlyde\* for Astigmatism (lotrafilcon B) contact lenses achieve rotational stability on the eye in just 30 seconds.
- c) Evaluate the fit of the lenses on the eye. The *Push-up Test*, as described below is an important part of the lens evaluation. The following guidelines will be helpful in fit evaluation:

#### Characteristics of a Well-fitted Lens

A well-fitted AIR OPTIX\* for Astigmatism and AIR OPTIX\* plus HydraGlyde\* for Astigmatism (lotrafilcon B) contact lens satisfies the following criteria:

- 1. Full corneal coverage and good centration (no limbal exposure)
- Sufficient lens movement to allow tear exchange under the lens during blink in primary or upward gaze

#### Push-up Test:

- This test is a reliable indicator of a good fit. With the patient looking straight ahead, place your index finger on the patient's lower lid and nudge the edge of the lens upward while observing lens movement. Then pull the lid back down and observe the return of the lens.
- A well-fitted lens will move freely upward, stopping shortly after passing the limbus and then return freely to its original position.
- 3. Good comfort
- 4. Acceptable visual acuity with over-refraction

#### Characteristics of a Tight (Steep) Lens Fit

A tight or steep fit should not be dispensed. If a lens fit is judged to be too steep a flatter lens (larger base curve), if available, should be evaluated. A tight or steep lens fit would display some or all of the following characteristics:

- 1. Good centration
- 2. Insufficient or no lens movement during a blink in primary or upward gaze

#### **Push-up Test:**

- A tight fitting lens will resist movement. If successfully nudged upward, the lens may remain decentered or return slowly to its original position.
- Good comfort
- 4. Blurred vision between blinks

#### Characteristics of a Loose (Flat) Lens Fit

If a lens fit is judged to be too flat a steeper lens (smaller base curve), if available, should be evaluated. A loose lens fit would display some or all of the following characteristics:

- 1. Decentration
- 2. Excessive lens movement during a blink in primary or upward gaze

#### **Push-up Test:**

- A loose fitting lens will move very easily, well beyond the limbus and possibly encroaching upon or going beyond the pupil. It will then return very quickly to its original position and often times return lower than its original position.
- 3. Reduced comfort
- 4. Lens edge standoff
- 5. Blurred vision immediately after the blink

#### 7. Initial Lens Orientation Evaluation

#### A. No Rotation

When the scribe lines orient vertically, the cylinder axis of the lens that is dispensed or ordered should be the same as the spectacle refractive axis - not the trial lens axis.

Contact lens cylinder axis = Spectacle refractive axis

#### B. Clockwise Rotation

When the scribe lines rotate clockwise as observed looking at the patient, (i.e., temporally for the right eye, nasally for the left eye), <u>add</u> the degree of rotation to the spectacle refractive axis - not the trial lens axis.

Spectacle refractive axis + Trial lens rotation = Axis to order

Example:

Spectacle Rx: -2.50 -0.75 x 160
Diagnostic Lens: -2.00 -0.75 x 170
Over-refraction: -0.50 sphere

**Orientation:** 10 degrees clockwise (add) (160 + 10)

**Final power to order:** -2.50 -0.75 x 170

#### C. Counterclockwise Rotation

When the scribe lines rotate counterclockwise, <u>subtract</u> the degree of rotation from the spectacle refractive axis - not the trial lens axis.

Spectacle refractive axis - Trial lens rotation = Axis to order

Example:

 Spectacle Rx:
 -2.75 -0.75 x 180

 Diagnostic Lens:
 -2.00 -0.75 x 010

 Over-refraction:
 -0.75 sphere

**Orientation:** 10 degrees counterclockwise (subtract)

(180-10)

**Final power to order:** -2.75 -0.75 x 170

 NOTE: Occasionally when a cylinder axis compensation is made for orientation, the result may fall outside the traditional range of 0 to 180 degrees. In this case, the axis in accepted notation will be the difference between the absolute value determined and 180 degrees.

Example 1:

Spectacle Rx cylinder: x 170

Orientation: 20 degrees clockwise

Axis calculation: 170 + 20 = 190

(The 190 degrees is outside the traditional axis range)

Difference: 190 - 180 = 10

Axis to order: x 010

Example 2:

Spectacle Rx cylinder: x 010

Orientation: 20 degrees counterclockwise

Axis calculation: 10 - 20 = -10

Difference: 180 - I -10 I = 170

(The -10 degrees is outside the traditional axis range)

Axis to order: x 170

 NOTE: Scribe marks on dispensed lenses must be at the same orientation as the trial lenses. Record rotation compensation as part of the final Rx.

#### D. Scribe Lines

To view the scribe lines, the following tips may be helpful:

- The first step is to narrow the slit lamp beam to approximately 0.5 mm in a horizontal orientation. Focus the beam on the lens surface at the 6 o'clock position.
- Slowly move the beam in an up and down fashion. As the beam
  passes near and through the scribe marks it will be easy to see in retro
  illumination.
- Once the scribe line is located, rotate the light beam so it is parallel to the 6 o'clock scribe mark, ensure the light beam passes through the center of the pupil, and measure the amount of lens rotation. Scribe lines are located at 3 and 9 o'clock.



#### 8. Initial Visual Evaluation

The visual result is evaluated by first performing a spherical over-refraction and then measuring visual acuity. If visual acuity is acceptable, the determination of lens power required after the over-refraction will be uncomplicated.

If the spherical over-refraction does not yield acceptable vision proceed to perform a spherocylindrical over-refraction. For the resultant lens power to order from this over-refraction call Technical Consultation in the U.S.A. at 1-800-241-7468 or visit www.virtualconsultant.alcon.com.

^Determination of final cylinder axis to order will be made after compensation for lens orientation.

#### FITTING GUIDELINES (Multifocal Lenses)

The AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal (lotrafilcon B) soft contact lens is a progressive aspheric simultaneous vision soft contact lens available in three ADD powers [low (LO), medium (MED) and high (HI)]. For each lens the near and intermediate powers are concentrated primarily in the central portion of the optical zone while distance power is contained in the surrounding portion. The continuous changes in power across the surface of the lens allow patients requiring a reading addition of up to + 3.00 D to see clearly at far, intermediate, and near distances.

Achieving high success with AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal contact lenses is dependent on several factors, including the patient's motivation, expectations and visual wearing environment, as well as your skill in optimizing the lens powers to balance binocular performance at distance and near. The information in this guide is designed to provide you with the tools to manage your presbyopic patients through each stage of the process from the initial case history to post-fitting follow-up.

#### 1. Pre-fitting Examination

#### A pre-fitting examination is necessary to:

- Determine whether a patient is a suitable candidate for AIR OPTIX\*
   AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal soft
   contact lenses
- Make ocular measurements for initial contact lens parameter selection
- Collect baseline clinical information to which post-fitting examination results can be compared

#### A pre-fitting examination should include:

- A thorough case history
- · Detailed assessment of patient's individual visual demands
- · Understanding of patient's objectives for lens wear and expectations
- A distance spherocylindrical refraction and near ADD determination
- · Eye dominance determination and measurement of pupil diameter
- Keratometry
- Tear assessment
- Biomicroscopy

Note: The importance of a thorough case history should not be underestimated. The information gained through careful listening and probing will help greatly in satisfying each patient's unique needs.

#### 2. Patient Selection

The eye care professional should weigh several factors when considering patient selection for an AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal (lotrafilcon B) soft contact lens fitting. When fitting a lens intended to correct for presbyopia, it is especially important to evaluate the particular visual needs, objectives, lifestyle and expectations of the individual patient. Prospective candidates may include current contact lens wearers, former wearers, and persons with no previous wear history. For former wearers it is important to determine the cause for discontinuation. Good success has been achieved with AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal soft contact lenses in all three wearing groups.

There are two general categories of candidates based on anticipated usage: those who seek to wear their lenses as their principal means of vision correction, and those who wish to integrate the use of their contact lenses with spectacles. The integrative user often seeks to wear their lenses for sports or other occasional activities while reverting to spectacles under poor lighting or otherwise demanding vision conditions. In general, even the part-time user does not require more than a few moments re-adaptation time following an interval of no lens wear.

While candidates with greater than 1.00 diopter of refractive error have often been thought of as better candidates than those with low error or emmetropia, this is a generalization that often does not hold true for a given individual. Success is influenced by many factors and the eye care professional is encouraged to offer AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal (lotrafilcon B) soft contact lenses to all interested presbyopic patients who satisfy the standard requirements for soft contact lens wear.

To summarize patient selection, the characteristics of "ideal candidates" and those that will be more difficult to fit are listed below:

#### **Ideal Candidates**

- Refractive cylinder ≤ 1.00 D
- Near add > +0.75 D
- Attainable visual demands that do not depend upon resolving very fine (smaller than 20/20 letters) details at both distance and near for extended periods
- Emphasis on tasks where it is advantageous to have objects simultaneously in focus over a large range of viewing distances
- Expectations consistent with actual everyday visual demands
- Motivated to wear lenses and understands that vision may not always be as sharp as with spectacles for some distances or lighting conditions
- Unable to adapt to monovision correction

#### **Less than Ideal Candidates**

- Critical or very fine visual demands at both distance and near
- Emerging presbyope with plano or very low distance powers
- Refractive cylinder ≥ 1.50 D (any axis) in one or both eyes or against-therule refractive cylinder > 1.00 D in one or both eyes
- Monocular distance acuities poorer than 20/20 with spherical equivalent refractive correction
- Myopic anisometropia where the refractive error for one of the two eyes is low (≤1.50 D) and has not been habitually corrected
- Pupil size larger (> 4 mm) or smaller (< 3 mm) than norm for presbyopic population under natural illumination conditions
- Abnormal binocular sensory function (e.g., amblyopia or strabismus)
- Expectation to discard and never use spectacles again, even for special tasks or viewing conditions
- Highly satisfied monovision wearers
- Any other contraindications to successful contact lens wear such as tear abnormality or lid margin disease

#### 3. Initial Lens Selection

#### A. Initial Base Curve Selection

AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\*
Multifocal contact lenses are available in a single 8.6 mm base curve.

#### B. Initial Lens Power Selection

Note: A careful maximum plus spherocylindrical refraction and nearpoint add determination should be conducted prior to selecting an AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal trial lens. Some practitioners have reported that adding 0.25D of plus provides a more efficient fit success. Autorefraction findings should be refined manually to rule out effects of instrument myopia and ensure proper control of residual accommodation.

The AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal soft contact lens design makes selecting the initial lens power easy. The optimum starting point is with a power that is more plus or least minus, vertex-corrected equivalent spectacle refraction.

#### C. Initial ADD Selection

The AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal contact lens 3 ADD SYSTEM allows personalized fitting for presbyopic patients. The table below makes initial ADD selection easy.

AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal ADD Selection

| SPECTACLE ADD | BOTH EYES |
|----------------|-----------|
| Up to +1.25 | Lo |
| +1.50 to +2.00 | MED |
| +2.25 to +2.50 | |

| Example 1: | | | |
|-------------------------------------|------------------|--------|----------|
| some acceptance of the second | OD | | os |
| Spherical Rx: | -4.50 -0.75 x 90 | | -4.00D |
| Spherical equivalent (least minus): | -4.75D | | -4.00D |
| Vertex corrected power: | -4.50D | | -4.00D |
| Spectacle ADD: | | +0.75D | |
| Eye Dominance: | | OD | |
| Initial Trial lens: | 4.50 LO | | -4.00 LO |

| Example 2: | | | |
|-------------------------|-------------------|--------|-------------------|
| | OD | | os |
| Spherical Rx: | +4.25 -0.25 x 180 | | +4.00 -0.50 x 180 |
| Spherical equivalent | +4.25D | | +3.75D |
| (least minus): | | | |
| Vertex corrected power: | +4.50D | | +3.75D |
| Spectacle ADD: | | +2.00D | |
| Eye Dominance: | | OS | |
| Initial Trial lens: | +4.50 MED | | +3.75 MED |

#### 4. Initial Lens Fitting Evaluation

- a) Insert the lenses selected in Step 3 above. If the exact power is not available, choose the next closest lens power in your trial set.
- b) Allow the lenses to settle on the eyes for approximately **5 to 10 minutes**. This allows time for the patient to adapt to the lenses and time for the lens to equilibrate with the patient's tears.
- c) Evaluate the fit of the lenses on the eye. The *Push-up Test* as described below is an important part of the lens evaluation. The following guidelines will be helpful in evaluating the physical fit of the lens:

#### Characteristics of a Well-fitted Lens

A well-fitted AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal (lotrafilcon B) contact lens satisfies the following criteria:

- Full corneal coverage and good centration (no limbal exposure). A lens that is decentered >1 mm, regardless of the direction, is less likely to give adequate vision.
- 2. Lens movement of 0.3 mm or less should be present to allow tear exchange under the lens during a blink in primary gaze or upward gaze.

#### Push-up Test:

- This test is a reliable indicator of a good fit. With the patient looking straight ahead, place your index finger on the patient's lower lid and nudge the edge of the lens upward while observing lens movement. Then pull the lid back down and observe the return of the lens.
- A well-fitted lens will move freely upward, stopping shortly after passing the limbus and then return freely to its original position.
- 3. Good comfort
- 4. Acceptable visual acuity with over-refraction

#### Characteristics of a Tight (Steep) Lens Fit

A tight or steep fit should not be dispensed. If a lens fit is judged to be too steep a flatter lens (larger base curve), if available, should be evaluated. A tight or steep lens fit would display some or all of the following characteristics:

- 1. Good centration
- 2. Insufficient or no lens movement during a blink in primary gaze or upward gaze

3. Excessive conjunctival drag (visible movement of the conjunctival vessels when the lens moves during a blink or during the push-up test). Note: presbyopes often have loose conjunctiva, some conjunctival movement is occasionally seen and may not be a sign of a tight fit. See *Push-up Test* below.

#### **Push-up Test:**

- A tight fitting lens will resist movement. If successfully nudged upward, the lens may remain decentered or return slowly to its original position.
- 4. Good comfort
- 5. Blurred vision between blinks

#### Characteristics of a Loose (Flat) Lens Fit

If a lens fit is judged to be too flat a steeper lens (smaller base curve), if available, should be evaluated. A loose lens fit would display some or all of the following characteristics:

- 1. Decentration
- 2. Excessive lens movement during the blink in primary or upward gaze

#### **Push-up Test:**

- A loose fitting lens will move very easily, well beyond the limbus and possibly encroaching upon or going beyond the pupil. It will then return very quickly to its original position and often times return lower than its original position.
- 3. Reduced comfort
- 4. Lens edge standoff
- 5. Blurred vision immediately after the blink

#### 5. Initial Lens Visual Evaluation

While lenses are settling, it is helpful to take the patient from the exam room to a "real-world" setting such as a room with an outside view. Once an acceptable fit has been achieved, the visual performance of the lenses may be evaluated. Visual acuity is tested at distance. If necessary, a spherical over-refraction should be performed using a trial frame or hand held lenses rather than a phoropter. This technique is essential when fitting multifocal lenses because it allows the patient to maintain the head posture and direction of gaze (relationship between eye and head) that he or she would naturally use during everyday tasks. This ensures that the visual performance of the lens is being assessed under conditions where the on-eye positioning matches that which will occur when the lens is being used, for example, for near work activities. In addition, pupil size will not be artificially increased by the reduction in light associated with looking through the aperture of the phoropter cells, or decreased by proximal cues associated with the nearness of the instrument.

#### 6. Fitting Procedures

Step 1. After the trial lenses have settled for 15 minutes, measure distance acuity while the patient is viewing the chart binocularly (i.e., simultaneously with both eyes). Next, evaluate the patient's subjective

impression of the near vision when trying to read typical everyday material (e.g., a newspaper, magazine, and cell phone). Lighting and reading distance should be what is normal for the patient.

- Step 2. If distance or near vision is unsatisfactory, perform a distance over-refraction on eye as follows. Use hand-held trial lenses and encourage plus. For example, if a plano and a +0.25D over-refraction yields the same results, use the +0.25 endpoint. Re-check visual acuity and visual quality as described in step 1 above. If over-refraction is other than plano, go immediately to new trial lenses, keeping the ADD the same.
- Step 3. If distance and near vision are satisfactory, dispense lenses and remind patient to use good light when reading fine print. It is helpful to let the patient experience the lenses in their natural environment before further procedures for enhancing vision are performed.
- Step 4. Enhanced Near Vision. If near vision is unsatisfactory, determine the dominant eye by the following method. Determine the eye with greatest plus acceptance by placing +1.50 handheld trial lens over each eye alternately while patient views the distance with both eyes open. Consider the eye for which binocular vision blurs least with the +1.50 to be the non-dominant eye.
  - Step 4A: Check the patient's binocular acuity with +0.50 over the non-dominant eye to determine if near vision is improved and distance vision is still acceptable. If so, place a new trials lens with the same ADD on the non-dominant eye, adjusting the distance power by +0.50.

| Enhanced near vision, Step A | | |
|---|---|---|
| SPECTACLE ADD | DOMINANT EYE | NON-DOMINANT EYE<br>(PLUS ACCEPTED) |
| Up to +1.25 | 0 | with additional +0.50 |
| +1 50 to +2.00 | 0 | with additional +0.50 |
| +2 25 to +2.50 | 0 | with additional +0.50 |

Next, re-check visual acuity and visual quality as described in Step 1 above. If satisfactory, dispense new distance lens power for the non-dominant eye. If near vision is still unsatisfactory, proceed to Step B:

Step 4B: If near vision is still unsatisfactory, adjust ADD as shown below.

| SPECTACLE ADD | DOMINANT EYE | NON-DOMINANT EYE<br>(PLUS ACCEPTED) |
|----------------|--------------|-------------------------------------|
| Up to +1.25 | | |
| +1.50 to +2.00 | | 0 |
| +2.25 to +2.50 | 0 | |

Note: It is common to question the rather non-intuitive step we suggest for enhancing vision at near in the HI ADD range, where the suggestion is to "back-off" to a MED ADD for the non-dominant eye, the same suggestion we make for enhancing distance vision (below). The reason for this is that after establishing (in Step A) that increasing plus is not helpful, the next most common reason for blur at near (or distance) is unacceptable ghosting that degrades the image quality. Backing down to the MED ADD in one eye can often relieve that and actually improve vision at near.

Step 5: Enhanced Distance Vision. If distance over-refraction did not improve visual acuity, adjust ADD according to the chart below.

| SPECTACLE ADD | DOMINANT EYE | NON-DOMINANT EYE<br>(PLUS ACCEPTED) |
|----------------|--------------|-------------------------------------|
| +1.50 to +2.00 | 0 | (HED) |
| +2.25 to +2 50 | 0 | MED |

#### Dispensing Visit (Multifocal lenses)

AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal (lotrafilcon B) soft contact lenses are supplied in multipack cartons with individual foil-sealed lens containers. Locate the opening flap on the multipack carton and pull up to break the seal.

The lenses are supplied in an easy-to-open foil container designed to maintain sterility of the lens and saline storage solution. To open an individual lens container peel back the lid and carefully remove the lens from its container. (Do not use tweezers or other tools to remove the lens from the package. This could damage the lens.)

Conduct the following steps with each patient, even if they have previously worn contact lenses:

#### 1. Evaluation of Lens Fit

Evaluate lens fit and visual response with the lens on the eye. The criteria of a well-fitted lens should be met and the patient's visual acuity should be acceptable. If not, the patient should be refitted with a more appropriate lens.

#### 2. Lens Placement and Removal Directions

Instruct the patient on proper lens placement and removal procedures. Patients who are unable to place and remove lenses should not be provided with them.

#### 3. Specific Instructions for Presbyopic Patients

Specific instructions, explanations and demonstrations are important for optimizing patient success with multifocal contact lenses. The following information and instructions have proven useful in advising patients who wear AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* soft contact lenses.

- a. A contact lens that contains different powers for distance and near involves greater technological and optical complexity than does a bifocal or multifocal spectacle lens. This is because the contact lens moves with the eye, rather than having the eye move up and down while the lens remains suspended in a frame. While the contact lens therefore gives an unobstructed field of view and greater freedom regarding where to look, these advantages may mean that the sharpness of vision may not always be exactly the same as what would be experienced with spectacles.
- b. Although many individuals use AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal soft contact lenses for full-time wear, it is not unusual to find that there may be some activities where one prefers to wear spectacles, or where the disadvantages associated with spectacles are outweighed by other issues. This is an entirely normal and natural response to the challenges presented by presbyopia.
- c. Situations where vision with multifocal contact lenses may be less sharp or otherwise "different" than what is experienced with spectacles often involve low illumination (e.g., a semi-dark room), reduced visibility (e.g., outdoor conditions of fog or heavy rain), or isolated sources of very bright light (e.g., headlights of an oncoming vehicle on a narrow country road). Patients should be instructed to make use of good light when reading fine print.
- d. Patients should be aware that it might be advisable to refrain from wearing their lenses while driving, flying an airplane or operating heavy machinery under these conditions until they gain some experience with the lenses in a similar visual environment.
- e. Small changes in lens power can often make an enormous difference in the quality of the vision experienced with multifocal contact lenses. Such changes can be best tailored to individual needs only after the lenses have been worn during the tasks and environmental conditions that the patient will personally encounter on a day-to-day basis. Confidence and assurance that such refinements, if needed, can be achieved is important for patient motivation during the initial period of lens wear.


#### FITTING GUIDELINES (Monovision)

#### 1. Patient Selection

#### A) Monovision Needs Assessment

For a good prognosis, the patient should have adequately corrected distance and near visual acuity in each eye. Patients with reduced visual acuity, such as the amblyopic patient, may not be a good candidate for monovision. Occupational and environmental visual demands should be considered. If the patient requires critical vision (visual acuity and stereopsis), it must be determined by trial whether this patient can function adequately with monovision. Monovision contact lens wear may not be optimal for such activities as:

- visually demanding situations such as operating potentially dangerous machinery or performing other potentially hazardous activities; and
- driving automobiles (e.g., driving at night). Patients who cannot pass requirements for a driver's license with monovision correction should not drive with this correction. An additional over-correction can be prescribed to improve vision

#### B) Patient Education

All patients do not function equally well with monovision correction. Patients may not perform as well for certain tasks with this correction as they have with bifocal reading glasses. Each patient must understand that monovision, as well as other presbyopic contact lenses, or other alternatives, can create a vision compromise that may reduce visual acuity and depth perception for distance and near tasks. During the fitting process, it is necessary for the patient to realize the disadvantages as well as the advantages of clear near vision in straight-ahead and upward gaze that monovision contact lenses provide compared to spectacle bifocals.

#### 2. Eye Selection

Generally, the non-dominant eye is corrected for near vision. The following test for eye dominance can be used:

#### A) Ocular Preference Determination Methods

- Method 1 Determine which eye is the "sight eye". Have the patient point
  to an object at the far end of the room. Cover one eye. If the patient is
  still pointing directly at the object, the eye being used is the dominant
  (sighting) eye.
- Method 2 Determine which eye will accept the added power for near with the least reduction in distance vision. Place a trial spectacle near add lens in front of one eye and then the other while the distance refractive error correction is in place for both eyes. Determine whether the patient functions best with the near add lens over the right or left eye.

#### B) Refractive Error Method

 For anisometropic corrections, it is generally best to fit the more hyperopic (less myopic) eye for distance and the more myopic (less hyperopic) eye for near.
#### C) Visual Demands Method

 Consider the patient's occupation during the eye selection process to determine the critical vision requirements. If a patient's gaze for near tasks is usually in one direction, correct the eye on that side for near.

#### Example:

A person who places copy to the left side of the desk will usually function best with the near lens on the left eye.

#### 3. Special Fitting Considerations

### **Unilateral Lens Correction**

There are circumstances where only one contact lens is required. As an example, an emmetropic patient would only require a near lens while a bilateral myope may require only a distance lens.

#### Examples:

- Emmetrope: A presbyopic emmetropic patient who requires a +1.75 diopter add would have a +1.75 lens on the near eye and the other eye left without a lens.
- **Bilateral myope**: A presbyopic patient requiring a +1.50 diopter add who is -2.50 diopters myopic in the right eye and -1.50 diopters myopic in the left eye may have the right eye corrected for distance and the left uncorrected for near.

#### Unilateral astigmat:

a) Emmetropic in one eye, astigmatic in the other

Spectacle Rx
O.D. Plano
O.S. -1.00 -1.00 x 090
Add: +1.50

Potential Monovision Rx
Uncorrected for distance
+0.50 -1.00 x 090 for near

b) Myopic in one eye, astigmatic in the other

Spectacle Rx
O.D. -1.50
O.S. -2.00 -1.75 x 090

Potential Monovision Rx
Uncorrected for near
-2.00 -1.75 x 090 for distance

#### **Amblyopia**

The amblyopic patient may not be a good candidate for monovision.

#### **Astigmatism**

Although patients with less than 1.50 diopters of astigmatism might be successfully fit in AIR OPTIX\* AQUA and AIR OPTIX\* plus HydraGlyde\* (lotrafilcon B) spherical lenses, patients with ≥ 0.75 diopters of astigmatism might be better candidates for monovision using AIR OPTIX\* for Astigmatism and AIR OPTIX\* plus HydraGlyde\* for Astigmatism (lotrafilcon B) toric soft contact lenses (check available cylinder powers).

- Determine which eye to use for the near prescription (see *Eye Selection*, A-C, above)
- Add the appropriate near add power to the spherical component of the astigmatic prescription for that eye.

| Example: | Spectacle Rx | Potential Monovision Rx |
|---|---|---|
| | O.D.: -2.50 – 0.75 x 180 | -2.50 -0.75 x 180 for distance |
| | O.S.: -3.00 - 1.75 x 165 | -2.00 -1.75 x 165 for near |
| | Add: +1.00 | |
| Domina | nt Eye: O.D. | |

#### **Near Add Determination**

Always prescribe the lens power for the near eye that provides optimal near acuity at the midpoint of the patient's habitual reading distance. However, when more than one power provides optimal reading performance, prescribe the least plus (most minus) of the powers.

#### Trial Lens Fitting

A trial lens fitting is performed in the office to allow the patient to experience monovision correction. Lenses are fit according to the directions in the *Fitting Guidelines* and *Base Curve Selection* sections described earlier in the guide.

Case history and standard clinical evaluation procedures should be used to determine the suitability of monovision. Determine which eye is to be corrected for distance and which eye is to be corrected for near. Next determine the near add. With trial lenses of the proper power in place, observe the reaction to this mode of correction.

Immediately after the correct power lenses are in place, walk across the room and have the patient look at you. Assess the patient's reaction to distance vision under these circumstances. Then have the patient look at familiar near objects such as a watch face or fingernails. Again assess the reaction. As the patient continues to look around the room at both near and distance objects, observe the reactions. Only after these vision tasks are completed, should the patient be asked to read print. Evaluate the patient's reaction to large print (e.g., typewritten copy) at first and then graduate to news print and finally smaller type sizes.

After evaluating the patient's performance under the above conditions, tests of visual acuity and reading ability under conditions of moderately dim illumination should be attempted.

An initial unfavorable response in the office, while indicative of a less favorable prognosis, should not immediately rule out a more extensive trial under the usual conditions in which a patient functions.

#### Adaptation

Visually demanding situations should be avoided during the initial wearing period. A patient may at first experience some mild blurred vision, dizziness, headaches, and feeling of slight imbalance. You should explain the adaptational

symptoms to the patient. These symptoms may last for a few minutes or for several weeks. The longer these symptoms persist, the poorer the chance for successful adaptation.

To help in the adaptation process, the patient can be advised to first use the lenses in a comfortable, familiar environment such as in the home.

Some patients feel that automobile driving performance may not be optimal during the adaptation process. This is particularly true when driving at night. Before driving a motor vehicle, it is recommended that patients be a passenger first to make sure that their vision is satisfactory for operating an automobile. During the first several weeks of wear (when adaptation is occurring), it may be advisable for the patient to only drive under optimal driving conditions. After adaptation, and success with these activities, the patient should be able to drive under other conditions with caution.

#### Other Suggestions

The success of the monovision technique may be further improved by having your patient follow the suggestions below:

- Have a third contact lens (distance power) to use when critical distance viewing is needed.
- Have a third contact lens (near power) to use when critical near viewing is needed.
- Have supplemental spectacles to wear over the monovision contact lenses for specific visual tasks. This is particularly applicable for those patients who cannot meet driver's licensing requirements with a monovision correction.
- Make use of proper illumination when carrying out visual tasks.

Success in fitting monovision can be improved by the following suggestions:

- Reverse the distance and near eyes if a patient is having trouble adapting.
- Refine the lens powers if there is trouble with adaptation. Accurate lens power is critical for presbyopic patients.
- Emphasize the benefits of the clear near vision in straight ahead and upward gaze with monovision.

The decision to fit a patient with a monovision correction is most appropriately left to the eye care professional in conjunction with the patient after carefully considering the patient's needs. All patients should be supplied with a copy of the *Patient Instruction Booklet*, which contains important instructions for the monovision wearer. You can obtain copies of the booklet by contacting an Alcon customer service representative in the USA at (800) 241-5999.

29

#### **DISPENSING VISIT**

To help ensure patient success the following steps should be conducted with each patient, even if they have previously worn contact lenses. Even experienced wearers are prone to develop bad habits over time.

AIR OPTIX\* AQUA, AIR OPTIX\* plus HydraGlyde\*, AIR OPTIX\* for Astigmatism, AIR OPTIX\* plus HydraGlyde\* for Astigmatism, AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal (lotrafilcon B) soft contact lenses are supplied sterile in foil sealed blister pack containers. Open the foil pack by peeling back the foil lidding material and gently slide the lens out of the container with your finger, or pour the lens onto the palm of your clean hand.

Conduct the following steps with each patient, even if they have previously worn contact lenses:

#### A. Verification of Lens Fit

Evaluate lens fit and visual response with the lens on the eye. The criteria of a well-fitted lens should be met and the patient's visual acuity should be acceptable. If not, the patient should be refitted with a more appropriate lens.

### **B. Hygiene and Lens Handling Instructions**

Good hygiene and proper lens handling are important factors in achieving safe, comfortable lens wear. Instruct the patient on hygiene and handling of lenses. Patients who are unable to place and remove lenses should not be provided with them.

C.Lens Wear and Replacement Schedules (see Package Insert)
Prescribe and explain the patient's wearing and replacement schedules.

### D. Lens Care Directions (see Package Insert)

Recommend an appropriate cleaning, rinsing, and disinfecting system, and provide the patient with instructions for proper lens care, including the case.

#### E. Additional Instructions

### Review the Package Insert

Provide the patient with all relevant information and precautions on the proper use of the lenses that are prescribed.

Provide the Patient Instruction Booklet for AIR OPTIX\* AQUA, AIR OPTIX\* plus HydraGlyde\*, AIR OPTIX\* for Astigmatism, AIR OPTIX\* plus HydraGlyde\* for Astigmatism AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\*Multifocal (lotrafilcon B) soft contact

Give the patient a copy of the *Patient Instruction Booklet* for the contact lenses you have prescribed. Review the contents so the patient clearly understands the prescribed lens wear, care, and replacement schedule. You can obtain copies of the instruction book by contacting Alcon customer service in the USA at (800) 241-5999.

#### **FOLLOW-UP EXAMINATIONS**

Follow-up care is extremely important for continued successful contact lens wear and for monitoring the patient's ocular response to lens wear. Follow-up care should include:

- Case history, including questions to identify any problems related to contact lens wear
- · Management of specific problems, if any, and
- A review with the patient of the lens wearing schedule, replacement schedule, and proper lens care and handling procedures.

### **Follow-up Examination Procedures**

- Prior to a follow-up examination, the contact lenses should be worn for at least four continuous hours.
- · Record patient's symptoms, if any.
- Measure visual acuity monocularly and binocularly with the contact lenses in place.
- Perform an over-refraction to check for residual refractive error.
- With a biomicroscope, evaluate lens fitting characteristics and examine the lens surface for deposits.
- Remove the lenses and conduct a thorough biomicroscopic examination with fluorescein. Rinse eyes with saline before re-inserting lenses.
- Evert upper lids to determine condition of tarsal conjunctiva.
- Periodically perform keratometry and spectacle refractions. These results should be recorded to compare to the initial measurements.
- If any observations are abnormal, use professional judgment to manage the problem and restore the eye to optimal conditions. If visual requirements are not satisfied during any follow-up examination, the patient should be re-fitted with a more appropriate lens.

#### **LENS HANDLING HINTS**

#### **Lens Insertion**

- When about to place the lens on the eye, make sure the lens sits up on the placement finger. The finger should be dry so surface tension does not cause the lens to adhere to the finger.
- Check to see that the lens is right side out. A lens that is placed on the eye inside out may not feel comfortable or provide good vision.

One way to do this is to place the lens between your thumb and index finger and squeeze the edges together gently.

- If the edges come together, the lens is right side out.
- If the edges turn outward, the lens is wrong side out. Carefully reverse it with your fingers.



Another way is to place the lens on the tip of your index finger and check its shape.

- · If the edge appears bowl-shaped, it is right side out.
- If the edge has a lip or flares outward, it is wrong side out and must be reversed.



The lens may be engraved with "CIBA". If the lens is engraved, look at the lens engraving at the edge of the lens.

- Place the lens on the tip of your index finger and hold it up against a light source.
- If the lens is right side out, you should be able to read "CIBA" at the edge of the lens. If the lens is inside out, the engravings will be reversed. Carefully turn the lens right side out with your fingers.



 Place the lens directly onto the cornea (placing it on the lower sclera can lead to the lens folding after a blink). While continuing to hold both lids in place, the patient should look down to seat the lens. The lids may then be released.

#### Lens Removal

- To remove the lens from the cornea, assure that the fingers are clean and dry.
- Slide the lens off the cornea (down or to the side) onto the sclera. This
  produces a fold in the lens, which assists in removal. With the index finger and
  thumb, gently pinch the lens off the eye.
- Remember to remove the same lens first (right or left), then the other lens.
   This helps avoid getting the lenses mixed up.
- It may be easier to remove contact lenses if you use rewetting drops (approved for use with soft lenses) recommended by the eye care professional 10 to 15 minutes before lens removal. This will also help prevent lens tearing during the removal process.

#### Care for a Sticking Lens

If the lens sticks (stops moving) or begins to dry on the eye, instruct the
patient to apply several drops of a recommended lubricating solution (used
in accordance with package labeling). The patient should wait until the lens
begins to move freely on the eye before attempting to remove it. If the lens
continues to stick, the patient should IMMEDIATELY consult the eye care
professional.

#### IN OFFICE CARE OF TRIAL LENSES

Eye care professionals should understand and educate contact lens technicians concerning proper use of trial lenses.

- Each contact lens is shipped sterile in a sealed blister pack containing phosphate buffered saline solution with or without additives. Hands should be thoroughly washed and rinsed and dried with a lint-free towel prior to handling a lens. In order to insure sterility, the blister pack should not be opened until immediately prior to use.
- For fitting and diagnostic purposes, the lenses should be disposed of after a single use and not be re-used from patient to patient.

#### ADDITIONAL INFORMATION

Alcon is pleased to assist with fitting or clinical questions regarding AIR OPTIX\* AQUA, AIR OPTIX\* plus HydraGlyde\*, AIR OPTIX\* for Astigmatism, AIR OPTIX\* plus HydraGlyde\* for Astigmatism, AIR OPTIX\* AQUA Multifocal and AIR OPTIX\* plus HydraGlyde\* Multifocal (lotrafilcon B) soft contact lenses. Eye care professionals having questions or problems should contact the Alcon Technical Consultation department, in the USA at (800) 241-7468. To order these contact lenses contact your Alcon sales representative or call Customer Service, in the USA at (800) 241-5999.

This page

left blank

# **VERTEX DISTANCE CONVERSION CHART**

For minus lenses, read left to right; for plus lenses, read right to left. (12 mm Vertex Distance)

| ` | | | , | | | | |
|------|------|-------|-------|-------|-------|-------|-------|
| - | + | - | + | - | + | - | + |
| 4.00 | 3.87 | 7.50 | 6.87 | 12.00 | 10.37 | 19.00 | 15.50 |
| 4.25 | 4.00 | 7.62 | 7.00 | 12.50 | 10.75 | 19.25 | 15.62 |
| 4.50 | 4.25 | 7.75 | 7.12 | 12.75 | 11.00 | 19.25 | 15.75 |
| 4.75 | 4.50 | 7.87 | 7.25 | 13.00 | 11.25 | 19.75 | 16.00 |
| 5.00 | 4.75 | 8.00 | 7.37 | 13.50 | 11.50 | 20.00 | 16.12 |
| 5.12 | 4.87 | 8.12 | 7.50 | 13.75 | 11.75 | 20.25 | 16.25 |
| 5.37 | 5.00 | 8.25 | 7.62 | 14.00 | 12.00 | 20.50 | 16.50 |
| 5.50 | 5.12 | 8.50 | 7.75 | 14.25 | 12.25 | 20.75 | 16.62 |
| 5.62 | 5.25 | 8.75 | 8.00 | 14.75 | 12.50 | 21.00 | 16.75 |
| 5.75 | 5.37 | 9.00 | 8.25 | 15.00 | 12.75 | 21.25 | 17.00 |
| 5.87 | 5.50 | 9.25 | 8.37 | 15.50 | 12.75 | 21.75 | 17.25 |
| 6.00 | 5.62 | 9.50 | 8.62 | 15.75 | 13.25 | 22.25 | 17.50 |
| 6.12 | 5.75 | 9.75 | 8.75 | 16.25 | 13.50 | 22.50 | 17.75 |
| 6.37 | 5.87 | 10.00 | 9.00 | 16.75 | 13.75 | 23.00 | 18.00 |
| 6.50 | 6.00 | 10.25 | 9.12 | 17.00 | 14.00 | 23.50 | 18.25 |
| 6.62 | 6.12 | 10.50 | 9.25 | 17.25 | 14.25 | 23.75 | 18.50 |
| 6.75 | 6.25 | 10.75 | 9.37 | 17.62 | 14.37 | 24.25 | 18.75 |
| 6.87 | 6.37 | 11.00 | 9.62 | 18.00 | 14.50 | 24.75 | 19.00 |
| 7.00 | 6.50 | 11.25 | 9.75 | 18.12 | 14.75 | 25.00 | 19.25 |
| 7.12 | 6.62 | 11.50 | 10.00 | 18.50 | 15.00 | 25.50 | 19.50 |
| 7.37 | 6.75 | 11.75 | 10.25 | 18.75 | 15.25 | 26.00 | 19.75 |

### Alcon

AR OPTE" AQUA, AR OPTE" pius HydraShyde", AR OPTE" for Astignastism, AR OPTE" pius HydraShyde" (AR OPTE" pius HydraShyde" Mullifocal, OPTE (Pius HydraShyde Mullifocal, OPTE (Pius HydraShyde Mullifocal, OPT

(Souly

THE CONTROL PRODUCT OF PROBLEM STATES TO THE CONTROL THAT BOTTON IN THE CONTROL OF T

THE CHARGE TERMINATION OF THE CHARGE T

- 3. Properties: Perfective 1.48 11 mm, -1.0000 (give the minute perfective 1.48 11 mm, -1.0000) (give the manufacture 2.48 5 mm, -1.0000) (give the manufacture 2.48 5 mm, -1.0000) (give the minute

t Diversion: 14.3 met or Trichrone: 8.09 men 69 - 3.000 (vertoe with power) CANN: 5.0 men

6 Care 1.

- Minus Present -0.56 to -0.000 (0.250) steps; -0.000 to -10.000 (0.250) steps; -0.000 to -10.000 (0.250) steps; -0.000 to -10.000 (0.250) steps; -0.000 to -10.000 (0.250) steps; -0.000 to -10.000 (0.250) steps; -0.000 (0.250) step

FTOT glass dipersibilitating context issues (poberced):
Int Manuster: 14.2 mm (6 -5.000 (revise with power) as Career: 8.8 mm

SEC.

Silvane Prosestor. -0.236 for -8.0000 file 5.3800 sheper. -0.400 for -12.0000 file
0.3010 sheper.

Plane Proventor. -0.955 for +8.0000 file.5500 sheper. +8.400 for +8.00000
(0.3010 sheper)

The Proventor -0.955 for +8.0000 file.5500 sheper. +8.400 for +8.00000
(0.3010 sheper)

FBC" for Antigrestians and SUB CRTEET plue bharaitedas for other context broom by the

AND ENTITY The Additional Control of the Section Control of the Sect

And the second of the second o

36

The age came prodimental discust the consideral should reventing larges early agent early update early update early update early update early update early update early updates early updates early updates, dearly early and by take a partial should be a partial or bedocker, bedocking update of any and by take Accordinated in the bedocker, bedocking update of the bedocker, bedocking updated by an all finallies.
 Figs Fartifactor, britishou, or the ordering any terms of Experience, buffer, update, early, instructions, described, amonthing traderia are frantify a particular construction in the second state of the secon

ner'n riedannerhendelikarin. Driedelikene preder for weekt syn in promott gelding finem redheld typ ga u. augstel of impiecemment laneme om benril er 'mnen lands-u.a genalikalis.

With Misself Rates That the Petitish is Medicing Contract Lances:

Private struct lighter that beetly one confession! That They are westing account that they are westing account.

The contractions have only the transportion, or desirable and of purposes and the purpose of the

JJVC Confidential

"PETTOPA ABBASE PORTING!" BASINLES!"

PETTOPA ABBASE PORTING! BASINLES!"

PETTOPA ABBASE PORTING! BASINLES!"

ABBASE PORTING PORTING! BASINLES!"

ABBASE PORTING PORTI



The contract and the contract contract and the contract c

er. Ne si kone on Bio the of year abean und stry right or lost ledae, finger. Finaer stabilis linger of Pau seems hand close to loves sychostop and pull finant

edicidist legist of transpositions them the state of the supposition of the color head in tit the uppositional of the color head in tit the uppositional of the color head in tit the uppositional of the color sample to the color head in tit the color of

Totales.

Misch skely exceed theme.

White Solvings up, use this tip of the thyger to state this time scient which the writer part of this eye.

Reminist the least by presence power access a second constitution of physical values of the second constitution and a second constitution of the second cons

The state several retributes, the state options of these helps to remove the state of the state

·<u>'</u>1:':.,'C":C:',.=r

DERIG (1992) In Ling Community or conformation of the Conformation of the

The second before the special for a large clocking particult, Transmitt you must be lower particulation on it special for a large clocking particult, Transmitt you must belower coronal The indehoculation in the interpolation product or disabled particulation and a CLEME (VIETE FALIS Concepts, is bishwinching biochemis or GMP) - FEEC \*\*
Particulation\*\* Can't a propose (Definitionally biochemis or GMP) - FEEC \*\*
Particulation\*\* Can't definition of Can't in Committee (Definitionally biochemis or GMP) - FEEC \*\*
Particulation\*\* Can't be not closes to began desired or for in concernmentable,

The confidence (Can't biochemis or Committee) and mist for incommittee (Can't biochemis or Can't biochemis or in the incommittee).

• Rect delirectation has not been taped and fit and recommendate.
Branche behavioration for the Lauro Stome
Carrian de an ears and fittes are attrained from assess very and fittes all fittes and properties of the Lauro Stome
Lauro and the second and the second and the second and the second and the second conde, with other an expectation provided to contain a read-entiring allows. The read-entire globars in the second properties are an expectation provided and provided and the second and

Others controlled they closed with the appropriate activated type solution and closed controlled they closed with the appropriate activated type solution and solve when it is a solution and the appropriate activated the solution and solve the solution and the appropriate activated the appropriate activated the largest controlled they associate all solved course enterly 2 inscribed, or see the physical appropriate price and solved course enterly 2 inscribed solved and appropriate activation and appropriate activation and physical appropriate price and solved activation, or source 8° deleveral and placetonisms delevation.

intense could summing one congrega.

Secondary

The secondary could be secondary to the could be selected as the could be

To being acceled a contract cape below from condemolarization, the oper care postulational should region by stationing absolution within the goldward of the contract contract of the provision of the contract of the contrac

All ACTION for Subspeciation, LL,DETIES CONTROL to succe Prospection Subsections Subsection Subsect

Fauses are erobyes; ja con

| žprava<br>Milovalsiku | Presstylline |
|---|---|
| <b>Short</b> | DELTER's femant lane Abdad Andrey wednis Ah<br>deuter in winder w.m. Der order of all Committings an<br>protections. |
| School | distinut originani |
| 2 | Uno-by desc |
| 207 | September sinks |
| I.RT | Bhilich sechs |
| <b>(</b> ) | tampia al lare mbar segrego-ordo piùglido |
| | Darrad son F idden persona in derrageni |
| C Same | Europus kadinsky audi avi falliei šalyusuda |
| | Dané interiero ir an |
| A | Deser |
| 19 (84) | учина под добительную устраную добител. |
| eri . | linahive |
| 8 | Pasinging remain illement algo |
| 10% | Chavales' |
| ec . | Bee sand |
| PAR | Puter |
| 3 | Libitata jane inasadi |
| Ann | म्हर्जीका कृतका |
| MAX. SERI | Ministers alleafest scielles seuter |
| Γē | ier |
| 986 | Bisins |
| - # | 睁 |
| L | let |
| ħ | Rex |
| WYDERFER. | Very protein all the protein and the state of the state o |

37

### LENS CARE PRODUCT CHART FOR SOFT CONTACT LENSES

CLEAR CARE\* Cleaning & Disinfecting Solution

3% Hydrogen peroxide based solution for cleaning, disinfecting & protein removal

CLEAR CARE\* PLUS Cleaning & Disinfecting Solution

3% Hydrogen peroxide based solution for cleaning, disinfecting & protein removal. Contains HydraGlyde\* Moisture Matrix multi-functional block copolymer that is primarily designed for wetting and lubricating silicone hydrogel lenses.

OPTI-FREE\* PureMoist\* Multi-Purpose Disinfecting Solution Multi-purpose solution for cleaning, rinsing, disinfecting, and protein removal. Contains HydraGlyde\* Moisture Matrix multi-functional block copolymer that is primarily designed for wetting and lubricating silicone hydrogel lenses.

### Other ALCON® Lens Care Products

**OPTI-FREE\* Rewetting Drops** 

Lubricating and rewetting

CLEAR CARE\* RINSE & GO\*

Rinsing Solution

Rinsing and storage

This page

left blank



Alcon Laboratories, Inc. 6201 South Freeway Fort Worth, TX 76134-2099, USA

U.S. Pat.: www.alconpatents.com

© 2014, 2016, 2018 Novartis \*a trademark of Novartis

March 2018

www.alcon.com W900127043-0318

# APPENDIX I: CLINICAL TECHNICAL PROCEDURES (CTP)

- LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS
- EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING
- DETERMINATION OF NEAR ADD
- NEAR logMAR VISUAL ACUITY MEASUREMENT PROCEDURE
- LENS FITTING CHARACTERISTICS
- SUBJECT REPORTED OCULAR SYMPTOMS
- DETERMINATION OF DISTANCE SPHEROCYLINDRICAL

### REFRACTIONS

- BIOMICROSCOPY SCALE
- KERATOMETRY
- DISTANCE AND NEAR VISUAL ACUITY EVALUATION
- ETDRS DISTANCE VISUAL ACUITY MEASURMENT PROCEDURE
- VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION

**TESTING** 

# LIMBAL & CONJUNCTIVAL (BULBAR) REDNESS

















# Attachment E



# EXPANDED SODIUM FLUORESCEIN CORNEAL STAINING










## Attachment A



# DETERMINATION OF NEAR ADD

























#### NEAR LOGMAR VISUAL ACUITY MEASUREMENT PROCEDURE







#### LENS FITTING CHARACTERISTICS












CR-6344, v1.0





### MOVEMENT Minimal, Acceptable (-1)



#### SUBJECT REPORTED OCULAR SYMPTOMS



# DETERMINATION OF DISTANCE SPHEROCYLINDRICAL REFRACTIONS



















#### BIOMICROSCOPY SCALE
















#### KERATOMETRY



#### DISTANCE AND NEAR VISUAL ACUITY EVALUATION






| Title: | Distance and Near Visual Acuity Evaluation |
|--------------|--------------------------------------------|
| ATTACHMENT A | · |

#### ETDRS DISTANCE VISUAL ACUITY MEASURMENT PROCEDURE










## VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION

















#### PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6344 Protocol Title Comparison of Two Silicone Hydrogel

Multifocal Contact Lenses

Version and Date: 1.0 19 July 2019

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155,<sup>1</sup> GCP and ICH guidelines,<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> United States (US) Code of Federal Regulations (CFR),<sup>4</sup> and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from, or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| _ | Signature | Date |
| | | - |
| | Name and Professional Position (Printed) | |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | |